# **PROTOCOL PA0009 AMENDMENT 3**

# EUdraCT Number: 2017-001003-74 IND Number: 128708 Sponsor: UCB Biopharma SRL pitchen and Allée de la Recharate de la Recharat

BELGIUM BELGIUM 1070 Brussels

| Protocol/Amendment number | Date | Type of amendment |
|-----------------------------------------|--------------|-------------------|
| Final protocol | 15 May 2017 | Not applicable |
| Protocol amendment 1 | 27 June 2017 | Not applicable |
| Protocol amendment 2 | 09 Mar 2018 | Substantial |
| Protocol amendment 2.1 (Czech Republic) | 11 Jun 2018 | Substantial |
| Protocol amendment 3 | 11 Dec 2019 | Nonsubstantial |

# **Confidential Material**

## Confidential

This document can This document is the property of UCB and may not – in full or in part – be passed on, reproduced, published, or otherwise used without the express permission of UCB.

> 

11 Dec 2019 PA0009

# STUDY CONTACT INFORMATION

# **Sponsor**

UCB BIOPHARMA SRL

Allée de la Recherche 60

1070 Brussels

**BELGIUM** 

# **Sponsor Study Physician**

| Name: | , MD | ansio |
|----------|-----------------|--------|
| Address: | UCB | O T |
| | 208 Bath Road | tag |
| | Slough, SL1 3WE | 29.0 |
| | UNITED KINGDOM | |
| Phone: | | icalil |

# **Clinical Project Manager**

| Name: | ALD italie |
|----------|----------------|
| Address: | UCB COLUMNOT |
| | 208 Bath Road |
| | Slough SL1 3WE |
| | UNITED KINGDOM |
| Phone: | |

# **Clinical Trial Biostatistician**

| Name: | |
|----------|----------------|
| Address: | UCB |
| 6/1/5 | 208 Bath Road |
| d'Ob | Slough SL1 3WE |
| allino | UNITED KINGDOM |
| Phone: | |


# **Clinical Monitoring Contract Research Organization**

| Name: | PRA Health Sciences |
|----------|----------------------------------|
| Address: | 4130 Park Lake Avenue, Suite 400 |
| | Raleigh, NC 27612 |
| | UNITED STATES |
| Phone: | +1-919-786-8200 |
| Fax: | +1-919-786-8201 |

# **SERIOUS ADVERSE EVENT REPORTING**

| | | Serious adverse event reporting (24h) |
|---|---|---|
| | Fax | |
| | | USA and Canada: +1 800 880 6949 or +1 866 890 3175 |
| | Email | Global: DS_ICT@ucb.com |
| This document of | annot be use | Europe and Rest of the World: +32 2 386 24 21 USA and Canada: +1 800 880 6949 or +1 866 890 3175 Global: DS_ICT@ucb.com Global: DS_ICT@ucb.com How support any market any mark |


# **TABLE OF CONTENTS**

| LIS | T OF A | BBREVIATIONS | | .9 |
|---|---|---|---|---|
| 1 | SUMM | MARY | | 13 |
| 2 | INTRO | DDUCTION | | 13 |
| 2.1 | <b>Psoriat</b> | tic arthritis | | 13 |
| 2. | .1.1 | Clinical studies. | | 14 |
| | .1.2 | Nonclinical studies | | 16 |
| 3 | STUD | Y OBJECTIVES | | 16 |
| 3.1 | Primar | y objective | on <sup>s</sup> | 16 |
| 3.2 | Second | dary objectives | | 17 |
| 3.3 | Other o | objectives | | 17 |
| 4 | STUD | Y VARIABLES | 1 | 17 |
| 4.1 | Primar | y variables | 1 | 17 |
| 4. | .1.1 | Primary safety variables | 1 | 17 |
| 4.2 | Second | Y OBJECTIVES y objective dary objectives objectives Y VARIABLES y variables Primary safety variables dary variables Secondary safety variable Secondary efficacy variables variables Safety variables Efficacy variables PK variable Immunological variable Y DESIGN description Rescue therapy Study duration per subject | 1 | 17 |
| 4. | .2.1 | Secondary safety variable | 1 | 17 |
| 4. | .2.2 | Secondary efficacy variables | 1 | 17 |
| 4.3 | Other v | variables | 1 | 17 |
| 4. | .3.1 | Safety variables | 1 | 17 |
| 4. | .3.2 | Efficacy variables | 1 | 18 |
| 4. | .3.3 | PK variable | 1 | 18 |
| 4. | .3.4 | Immunological variable | 1 | 18 |
| 5 | STUD | Y DESIGN | 1 | 18 |
| 5.1 | Study o | description | 1 | 18 |
| 5. | .1.1 | Rescue therapy | 1 | 19 |
| 5. | .1.2 | Study duration per subject | 1 | 19 |
| | .1.3 | Planned number of subjects and sites | 1 | 19 |
| 5. | .1.4 | Anticipated regions and countries | 1 | 19 |
| 5.2 | Schedu | ule of study assessments | | |
| 5.3 | Schem | afic diagram | 2 | 23 |
| 5.4 | Rationa | ale for study design and selection of dose | 2 | 23 |
| 6 | SELEC | CTION AND WITHDRAWAL OF SUBJECTS | 2 | 24 |
| <b>6.</b> 1 | Inclusi | on criteria | 2 | 24 |
| 6.2 | Exclus | sion criteria | 2 | 25 |
| 6.3 | Withdr | rawal criteria | 2 | 25 |
| 6. | .3.1 | Potential drug-induced liver injury investigational medicinal product discontinuation criteria | | 27 |
| 7 | CTLID | VTDEATMENT | , | 77 |

| 7.1 | Descri | ption of investigational medicinal product | 27 |
|---|---|---|---|
| 7.2 | Treatn | nent to be administered | 28 |
| 7.3 | Packag | ging | 28 |
| 7.4 | Labeli | ng | 28 |
| 7.5 | Handli | ing and storage requirements | 29 |
| 7.6 | Drug a | accountability | 29 |
| 7.7 | Proced | lures for monitoring subject compliance | 30 |
| 7.8 | Conco | mitant medications/treatments | 30 |
| 7 | .8.1 | Permitted concomitant treatments (medications and therapies) Prohibited concomitant treatments (medications and therapies) ng | .s30 |
| 7 | .8.2 | Prohibited concomitant treatments (medications and therapies) | 32 |
| 7.9 | Blindi | ng | 33 |
| 7.10 | ) Rando | mization and numbering of subjects | 33 |
| 8 | STUD | Y PROCEDURES BY VISIT | 33 |
| 8.1 | Visit 1 | | 33 |
| 8.2 | Week | 4 (Visit 2) and Week 8 (Visit 3) | 34 |
| 8.3 | Week | 12 (Visit 4), Week 24 (Visit 5), Week 36 (Visit 6), and Week 72 (Visit 9) | |
| 8.4 | Week | 16, Week 20, Week 28, Week 32, Week 40, Week 44, Week 52, Week 56, | Week |
| | 64, W | eek 68, Week 76, Week 80, Week 88, and Week 92 | 36 |
| 8.5 | Week | 48 (Visit 7) and Week 96 (Visit 11) | 36 |
| 8.6 | Week | 60 (Visit 8) and Week 84 (Visit 10) | 37 |
| 8.7 | Week | 100 (Visit 12) | 38 |
| 8.8 | | 104 (Visit 13) or Early Termination Visit | |
| 8.9 | SFU V | risit (20 weeks after the final dose of IMP) | 40 |
| 8.10 | Early [ | Termination Visit | |
| | l Unsch | eduled Visit | 40 |
| 9 | | SSMENT OF SAFETY | |
| 9.1 | Adver | se events | 41 |
| 9 | .1.1 | Definition of AE | 41 |
| 9 | .1.2 | AEs of special interest | 41 |
| 9 | .1.3 | Other safety topics of interest | 42 |
| 9 | .1.4 | Procedures for reporting and recording AEs | 42 |
| 9 | .1.5 | Description of AEs | 42 |
| 9 | .Y.6 | Follow-up of AEs | 43 |
| No 9 | .1.7 | Definition of AE AEs of special interest Other safety topics of interest Procedures for reporting and recording AEs Description of AEs Follow-up of AEs Rule for repetition of an AE | 43 |
| 9 | .1.8 | Pregnancy | 43 |
| | .1.9 | Suspected transmission of an infectious agent via a medicinal product | |
| | .1.10 | Overdose of investigational medicinal product | |
| 9 | .1.11 | Safety signal detection | 44 |

| 9.2 | Serious | s AEs | 45 |
|---|---|---|---|
| 9 | .2.1 | Definition of SAEs | 45 |
| 9 | .2.2 | Procedures for reporting serious adverse events | 46 |
| 9 | .2.3 | Follow-up of SAEs | 46 |
| 9.3 | Immed | liate reporting of AEs | 46 |
| 9.4 | Anticip | pated SAEs | 47 |
| 9.5 | Labora | tory measurements | 47 |
| 9 | .5.1 | Evaluation of PDILI | 48 |
| | 9.5.1. | Consultation with Medical Monitor and local hepatologist | 52 |
| | 9.5.1. | 2 Immediate action: determination of IMP discontinuation | 52 |
| | 9.5.1. | 3 IMP restart/rechallenge | 52 |
| | 9.5.1. | 4 Testing: identification/exclusion of alternative etiology | 52 |
| | 9.5.1. | 5 Follow-up evaluation | 54 |
| 9.6 | Other s | safety measurements | 54 |
| 9 | .6.1 | Vital signs | 54 |
| 9 | .6.2 | Body weight | 55 |
| 9 | .6.3 | Physical examination | 55 |
| 9 | .6.4 | 12-lead ECG | 55 |
| 9 | .6.5 | Evaluation of PDILI Consultation with Medical Monitor and local hepatologist Immediate action: determination of IMP discontinuation IMP restart/rechallenge Testing: identification/exclusion of alternative etiology Follow-up evaluation safety measurements Vital signs Body weight Physical examination 12-lead ECG Tuberculosis and TB risk factor assessment and management Tuberculosis assessment by IGRA | 55 |
| | 9.6.5. | The distribution of the second | |
| | 9.6.5. | 2 Tuberculosis questionnaire. | 56 |
| | 9.6.5. | | |
| 9 | .6.6 | Pregnancy testing. | 57 |
| 9 | .6.7 | Assessment of suicidal ideation and behavior | 57 |
| 10 | ASSES | SSMENT OF EFFICACY | 57 |
| | | oint evaluation for ACR response | |
| 10.2 | 2 28 join | t evaluation for determination of DAS28(CRP) | 58 |
| 10.3 | <b>Patient</b> | 's Globa PAssessment of Disease Activity | 58 |
| 10.4 | Physic: | ian's Global Assessment of Disease Activity | 58 |
| 10.5 | Patient | 's Assessment of Arthritis Pain | 58 |
| 10.6 | Health | Assessment Questionnaire-Disability Index score | 59 |
| 10.7 | 7 CRP le | evels | 59 |
| | | 0, ACR50, and ACR70 response | |
| 2.01 | BSA-P | <sup>2</sup> SO | 59 |
| 10.1 | 10.10 Psoriasis Area and Severity Index (PASI)60 | | |
| 10.1 | 10.11 MDA60 | | |
| 10.1 | 10.12 DAS28(CRP)61 | | |
| 10.1 | 3 1 | MASES | 61 |

| 10.14 LDI | |
|---|---|
| 10.15 Hospital Anxiety and Depression Scale | 61 |
| 10.16 PsAID-9 | 62 |
| 10.17 SF-36 | 62 |
| 11 ASSESSMENT OF IMMUNOGENICITY | 62 |
| 12 STUDY MANAGEMENT AND ADMINISTRATION | 62 |
| 12.1 Adherence to protocol | 62.12 |
| 12.2 Monitoring | |
| 12.2 Monitoring 12.2.1 Definition of source data 12.2.2 Source data verification 12.3 Data handling 12.3.1 Case Report form completion 12.3.2 Database entry and reconciliation | |
| 12.2.2 Source data verification | 63 |
| 12.3 Data handling | 64 |
| 12.3.1 Case Report form completion | 64 |
| 12.3.2 Database entry and reconciliation | 64 |
| 12.3.3 Subject Screening and Enrollment log/Subject Identification | 1 Code list64 |
| 12.4 Termination of the study | 65 |
| 12.5 Archiving and data retention | 65 |
| 12.6 Audit and inspection | 65 |
| 12.7 Good Clinical Practice | 66 |
| 13 STATISTICS | 66 |
| 12.3.3 Subject Screening and Enrollment log/Subject Identification 12.4 Termination of the study | 66 |
| 13.2 General statistical considerations | 66 |
| 13.3 Planned safety analyses | 66 |
| 13.3.1 Safety analyses | 66 |
| 13.4 Planned efficacy analyses | 67 |
| 13.4.1 Subgroup analysis | 67 |
| 13.5 Planned immunogenicity analyses | |
| 13.6 Other analyses | 68 |
| 13.7 Handling of protocol deviations | |
| 13.8 Handling of dropouts or missing data | |
| 13.9 Planned interim analysis and data monitoring | |
| 13.10 Determination of sample size | |
| 14 ETHICS AND REGULATORY REQUIREMENTS | |
| 143 Informed consent | |
| 14.2 Subject identification cards | |
| 14.3 Institutional Review Boards and Independent Ethics Committees | |
| 14.4 Subject privacy | |
| 14.5 Protocol amendments | |
| 15 FINANCE, INSURANCE, AND PUBLICATION | 70 |

| | 16 REFERI | ENCES | 71 |
|---|---|---|---|
| | 17 APPEN | DICES | 75 |
| | 17.1 Markedl | y abnormal laboratory values | 75 |
| | | Amendment 1 | |
| | | Amendment 2 | |
| | | Amendment 3 | |
| | 18 DECLA | RATION AND SIGNATURE OF INVESTIGATOR | 115 |
| | 19 SPONS | OR DECLARATION | (110 |
| | | LIST OF TABLES Schedule of study assessments. Prohibited or restricted medications Additional prohibited psoriasis treatments Anticipated SAEs for the population of subjects with psoriatic arthritis | , |
| | Table 5–1: | Schedule of study assessments | 20 |
| | Table 7-1: | Prohibited or restricted medications | 32 |
| | Table 7-2: | Additional prohibited psoriasis treatments | 32 |
| | Table 9–1: | Anticipated SAEs for the population of subjects with psoriatic arthritis | 47 |
| | Table 9-2: | Laudiatory incasurcincins | |
| | Table 9-3: | Required investigations and follow-up for PDILI PDILI laboratory measurements | 50 |
| | Table 9–4: | PDILI laboratory measurements | 53 |
| | Table 9–5: | PDILI information to be collected | 54 |
| | Table 10–1: | Swelling and tenderness grading | 58 |
| | Table 10–2: | Body areas for calculation of percent BSA for PASI | 60 |
| | Table 10–3: | MDA criteria in PsA | 61 |
| | Table 17-1: | Definitions of markedly abnormal hematology values | 75 |
| | Table 17–2: | Definitions of markedly abnormal biochemistry values | 75 |
| | | SUPY | |
| | | LIST OF FIGURES | |
| | Figure 5–1: | Schematic diagram | 23 |
| | , b | | |
| | anno | | |
| | CO. | | |
| -9 | ILLE, | | |
| 900 | )~ | | |
| This | | Body areas for calculation of percent BSA for PASI MDA criteria in PsA Definitions of markedly abnormal hematology values Definitions of markedly abnormal biochemistry values LIST OF FIGURES Schematic diagram | |


# LIST OF ABBREVIATIONS

**ACR** American College of Rheumatology

OP m application and any extensions or variations thereof. American College of Rheumatology 20, 50, 70% response criteria ACR20, 50, 70

AΕ adverse event

**AESI** adverse event of special interest

ALP alkaline phosphatase

**ALT** alanine aminotransferase AS ankylosing spondylitis AST aspartate aminotransferase

axSpA axial spondyloarthritis

BP blood pressure **BSA** body surface area

CDcluster of differentiation

**CDMS** clinical data management system

Chinese Hamster Ovarian **CHO** 

confidence interval CI

COX-2 cyclooxygenase-2

Clinical Project Manager **CPM** 

Contract Research Organization **CRO** 

C-reactive protein CRP

Disease Activity Score-28 joint count C-reactive protein DAS28(CRP)

disease-modifying antirheumatic drug **DMARD** 

exposure-adjusted event rate **EAER** 

Sexposure-adjusted incidence rate **EAIR** 

**ECG** electrocardiogram

**eCRF** electronic Case Report form

electronic Columbia-Suicide Severity Rating Scale

electronic data capture

**Enrolled Set** 

**Early Termination FAS** Full Analysis Set

**FDA** Food and Drug Administration

**GCP** Good Clinical Practice

| | GI | gastrointestinal |
|---|---|---|
| | GMP | Good Manufacturing Practice |
| | HADS | Hospital Anxiety and Depression Scale |
| | HADS-A | Hospital Anxiety and Depression Scale—Anxiety |
| | HADS-D | Hospital Anxiety and Depression Scale—Depression |
| | HAQ-DI | Health Assessment Questionnaire—Disability Index |
| | HRQoL | Hospital Anxiety and Depression Scale—Depression Health Assessment Questionnaire—Disability Index Health-Related Quality of Life Investigator's Brochure Inflammatory Bowel Disease International Council for Harmonisation Independent Ethics Committee Immunoglobulin G interferon-gamma release assay interleukin interleukin-17 receptor A investigational medicinal product |
| | IB | Investigator's Brochure |
| | IBD | Inflammatory Bowel Disease |
| | ICH | International Council for Harmonisation |
| | IEC | Independent Ethics Committee |
| | IgG | Immunoglobulin G |
| | IGRA | interferon-gamma release assay |
| | IL | interleukin |
| | IL-17-RA | interleukin-17 receptor A |
| | IMP | investigational medicinal product |
| | IP | investigational medicinal product interphalangeal Institutional Review Board |
| | IRB | Institutional Review Board |
| | IUD | intrauterine device |
| | IUS | intrauterine hormone-releasing system |
| | iv | intravenous |
| | IXRS | interactive web or voice response system |
| | LDI | Leeds Dactylitis Index |
| | LTB | latent tuberculosis |
| | MAb 8 | monoclonal antibody |
| | MABES MCMC | Maastricht Ankylosing Spondylitis Enthesitis Index |
| | MCMC XV | Markov Chain Monte Carlo |
| | MCP | metacarpophalangeal |
| | MDA | Minimal Disease Activity |
| 1 | MedDRA | Medical Dictionary for Regulatory Activities |
| | MI | multiple imputation |
| | NOAEL | no adverse effect level |
| | NRI | nonresponder imputation |

**NSAID** 

nonsteroidal anti-inflammatory drug

**NTMB** nontuberculous mycobacteria **OLE** 

**PASI** Psoriasis Area and Severity Index

ity extensions of variations thereof. Psoriasis Area and Severity Index 75%, 90%, 100% PASI75, PASI90,

open-label extension

PASI100

PD pharmacodynamics

**PDILI** potential drug-induced liver injury

**PFS** prefilled syringe

Patient's Global Assessment of Disease Activity **PGADA** 

Physician's Global Assessment of Disease Activity **PhGADA** 

PIP proximal interphalangeal

PK pharmacokinetics PS **Patient Safety PsA** psoriatic arthritis

Psoriatic Arthritis Impact of Disease PsAID-9

**PSO** psoriasis

Patient's Assessment of Arthritis Pain **PtAAP** psoralen plus ultraviolet A light therapy **PUVA** 

Q4W every 4 weeks (monthly) rheumatoid arthritis RA

**RCTC** Rheumatology Common Toxicity Criteria

SAE serious adverse event subcutaneous(ly) sc

Short-Form 36-item Health Survey SF-36

**SFU** Safety Follow-up SJC swollen joint count

**SOP** Standard Operating Procedure

SS Safety Set  $t_{1/\!\!/2}\,\mathcal{C}^{\!\!/}$ half-life

treatment-emergent adverse event

TP THE HOCH TP tuberculosis T helper 17

**TJC** tender joint count **TNF** tumor necrosis factor

| $TNF\alpha$ | tumor necrosis factor-alpha |
|-------------|-----------------------------|
| ULN | upper limit of normal |
| UVA | ultraviolet A |
| VAS | visual analog scale |

The document control he used to support any materials alterial and any settle for the support of

# **SUMMARY**

PA0009 is a multicenter, open-label extension (OLE) study evaluating the long-term safety, PA0008 is a multicenter, Phase 2b, randomized, double-blind, placebo-controlled, parallel-group, dose-ranging study to evaluate the efficacy and safety of bimekizumab in 200 subjects with active PsA.

In the PA0009 OLE study, bimekizumab will be administered at a diagram (Q4W) subcutaneously (sc) for all subjects regard!

Up to 200 subjects from Panager tolerability, and efficacy of bimekizumab in subjects with psoriatic arthritis (PsA). Only subjects

in PA0008.

The primary objective of PA0009 is to assess the long-term safety and tolerability of bimekizumab administered over a period of up to 100 weeks (~2 years). The primary safety variables are the incidences of treatment-emergent adverse events (TEAEs) and treatment-emergent serious adverse events (SAEs).

The secondary objective is to assess the long-term efficacy of bimekizumab over a period of up to 104 weeks (~2 years). The secondary efficacy variables include the American College of Rheumatology 20% (ACR20) response at Week 48 (with a responder defined as a subject with an improvement from PA0008 Baseline of ≥20% in the swollen and tender joint counts and at least 3 of the other 5 components of the core set of American College of Rheumatology [ACR] response measures), American College of Rheumatology 50% (ACR50) response at Week 48; American College of Rheumatology 70% (ACR70) response at Week 48, change from PA0008 Baseline in the Maastricht Ankylosing Spondylitis Enthesitis Index (MASES) at Week 48, change from PA0008 Baseline in the Leeds Dactylitis Index (LDI) at Week 48, the Psoriasis Area and Severity Index 75 (PASI75) response, and the Psoriasis Area and Severity Index 90 (PASI90) response at Week 48. The secondary safety variable is the withdrawal due to TEAEs.

Other objectives are to evaluate the impact on dactylitis, enthesitis, and patient-reported quality of life, and to assess the plasma concentrations and immunogenicity of bimekizumab.

The study duration for each subject is estimated to be up to a maximum of 120 weeks: an Open-Label Treatment Period of up to 100 weeks (~2 years), followed by a Safety Follow-up (SFU) Visit 20 weeks after the final dose of bimekizumab.

# INTRODUCTION

# **Psoriatic arthritis**

Psoriatic arthritis, a chronic inflammatory musculoskeletal disorder, occurs in approximately 6% to 41% of people affected by psoriasis (PSO) (Ogdie and Weiss, 2015). A substantial proportion of subjects have polyarthritis (McHugh et al, 2003). Disease-modifying antirheumatic drugs (DMARDs) and biological agents targeting tumor necrosis factor-alpha (TNFα), interleukin (IL)-17, and IL-12/23 are effective in PsA (Kavanaugh et al, 2012;

 Kavanaugh et al, 2009; Gottlieb et al, 2009; Gladman et al, 2007; Genovese et al, 2007; Kavanaugh et al, 2006; Antoni et al, 2005a; Antoni et al, 2005b; Mease et al, 2005; Mease et al, 2004, McInnes et al, 2015; Mease et al, 2015). However, some subjects are not

magnificated various isoforms comprising the IL-17 cytokine family in the pathophysiology of PSO and of PsA (Raychaudhuri et al, 2012; Fujishima et al, 2010; Watanabe et al, 2009; Harper et al, 2009; Johansen et al, 2009). Numbers of IL-17A positive cells are increased and localized in psoriatic skin lesions (Fujishima et al, 2010; Watanabe et al, 2009; Harper et al, 2009; Johansen et al, 2009). and II 17 overexpressed in the serum and skin lesions of and IL-17F in particular is a lesions of and IL-17F in particular is a lesions of and IL-17F. (Fujishima et al, 2010; Watanabe et al, 2009). Cluster of differentiation (CD) 4+ T helper 17 (Th17) cells, IL-17A, and IL-17 receptor A (IL-17-RA) have recently been shown to play a role in PsA (Raychaudhuri et al, 2012). Anti-IL-17 antibodies have been shown to be effective treatments for PSO (Papp et al, 2012; Leonardi et al, 2012; Hueber et al, 2010) and have also shown activity in subjects with rheumatoid arthritis (RA), PsA, and ankylosing spondylitis (AS) (McInnes et al, 2014; Mease et al, 2015; Hueber et al, 2010; Genovese et al, 2010). Taken together these data suggest that inhibition of both IL-17A and IL-17F could be therapeutically effective in subjects with PSO, PsA, and axial spondyloarthritis (axSpA).

Bimekizumab (UCB4940) is an engineered, humanized full-length monoclonal antibody (mAb) of immunoglobulin (IgG) 1 subclass of approximately 150,000 Dalton which is expressed in a genetically engineered Chinese Hamster Ovarian (CHO) cell line. Bimekizumab has high affinity for human IL-17A and human IL-17F and selectively and potently inhibits the activity of both isoforms in vitro. Therefore, it permits an evaluation of the potential for additional efficacy, which may be conferred by dual inhibition of both cytokines, in patients suffering from diseases in which both cytokines are active.

### Clinical studies 2.1.1

Four clinical studies of bimekizumab have been completed: UP0008 in 39 subjects with mild-to-moderate plaque PSO, RA0124 in 30 healthy volunteers, UP0031 in 12 healthy volunteers, and PA0007 in 53 subjects with PsA.

UP0008 was a Phase 1, single ascending dose study in adults with mild-to-moderate PSO affecting ≤5% body surface area (BSA). In this blinded study, single doses of up to 640mg (approximately 8mg/kg in an 80kg adult) were evaluated. A total of 26 subjects with PSO with <5% of body surface involvement were treated with a range of single intravenous (iv) doses from 8 to 640mg. The pharmacokinetics (PK) of bimekizumab was linear in the tested dose range. There were no clinically relevant safety findings identified at any dose and all doses were well tolerated. The prespecified exploratory assessment of disease activity showed clinically relevant and statistically significant improvements at the higher doses studied.

RA0124 was a Phase 1, open-label, parallel-group, single-dose study in healthy subjects. The primary objective of this study was to determine the absolute bioavailability of single sc doses of bimekizumab (80 and 160mg). The secondary objectives were to evaluate the dose proportionality of bimekizumab 80 and 160mg sc and to evaluate the safety and tolerability of


these sc doses and 160mg given by iv infusion. In RA0124, the absolute bioavailability was similar for the 2 doses tested (0.656 and 0.631 for the bimekizumab 80mg and 160mg sc doses, respectively). The median half-life  $(t_{1/2})$  following sc administration was similar to that following iv administration (27.81 days and 28.25 days for bimekizumab 160mg sc and bimekizumab 160mg iv, respectively).

Dinity of 2 bimekizumab formulations (a based formulation 2x80mg and an based formulation 1x160mg) administered by sc injection to healthy volunteers. Results similar geometric means for AUC between the 2 bimekizumab formulations mg=653.8day\*μg/mL; 1x160mg=628.3day\*μg/mL) and the relative izumab 1x160mg versus 2x80mg formulation on fidence interval (CD) 75 An additional Phase 1 study, UP0031, evaluated the relative bioavailability and safety and tolerability of 2 bimekizumab formulations (a show similar geometric means for AUC between the 2 bimekizumab formulations (2x80mg=653.8day\*μg/mL; 1x160mg=628.3day\*μg/mL) and the relative bioavailability for the bimekizumab 1x160mg versus 2x80mg formulations was calculated as 96.1% with a 95% confidence interval (CI): 72.7, 127.0. The wide 95% CI was expected due to the small sample size in UP0031.

Bimekizumab has also been investigated in a Phase 1b, proof-of-concept, randomized, placebo-controlled, multiple-dose study (PA0007). A total of 53 subjects have been randomized. The primary objective of PA0007 was to assess the safety and PK of multiple dose administration of iv bimekizumab in subjects with PsA. Four active doses and a placebo were tested. Drug was administered as a loading dose of bimekizumab 80, 160, 240, or 560mg at Week 1, and 2 additional doses of bimekizumab 40, 80, 160, or 320mg at Week 4 and Week 7. In each treatment group, subjects received a total of doses of bimekizumab, administered every 3 weeks. There were no unexpected clinically relevant safety findings and all doses were well tolerated. The PK was linear across the tested dose range and no change in PK was observed following multiple doses. Observed changes in inflammatory biomarkers were consistent with expectations based on the IL-17A and IL-17F mechanism of action. The exploratory analysis showed clinically relevant improvement in activity of PsA and in skin involvement in those subjects with concomitant active psoriatic lesions. Data from the top 3 bimekizumab dose groups pooled showed that, by Week 9, 80% (95% confidence interval [CI]: 62.7, 90.5) of subjects achieved an ACR20 response (vs.16.7% [95% CI: 4.7, 44.8] in the placebo group) and 100% (95% CI: 79.6, 100.0) of 26 subjects with active psoriatic lesions had achieved a PASI75 response (vs 0% [95% CI: 0.0, 43.4] in the placebo group).

Infections (mostly nasopharyngitis) were the most commonly reported events in both the active-treatment and the placebo group. None of the infections were considered serious or required treatment with antibiotics. Two subjects in the active-treatment group experienced 1 local candida infection each (oropharyngitis and vulvovaginitis) that were nonserious and resolved with topical therapy. There was a reduction in mean neutrophil count in the active-treatment group, although this drop was not clinically relevant and a clear relationship with dose or time was not evident. Some increases in liver function tests were reported, but none

In the bimekizumab clinical studies to date, the most commonly reported gastrointestinal (GI) adverse events (AEs) were abdominal distension, abdominal pain, diarrhea flatulare and vomiting. All of these events, except 1 events of intensity. The state of the state adverse events (AEs) were abdominal distension, abdominal pain, diarrhea, flatulence, nausea, intensity. T helper-17 and other IL-17-producing cell types are present in a high frequency in the physiologic, healthy state of the intestinal mucosa. Interleukin-17 is recognized as an important player in the pathophysiology of infectious and immune-mediated GI diseases and has been

shown to contribute to the gut barrier function (Ivanov et al, 2008). Clinical data with secukinumab suggest that the drug may worsen symptoms of coexisting Crohn's disease in patients with psoriasis and ankylosing spondylitis (Baeten et al., 2015).

pharmacodynamics (PD), and efficacy of multiple doses of bimekizumab administered as add-on therapy to stable certolizumab pegol (Cimzia®) therapy in subjects with moderate to severe D A to UC0011 is a Phase 2 study, which will evaluate the afficiency of the study of the severe D A to the severe D A loading dose and 2 sc maintenance doses of bimekizumab in subjects with moderate to severe active ulcerative colitis. PS0010, PS0011, PS0016, and PS0018 are Phase 2 studies, which will evaluate the PD, PK, safety, and/or efficacy of bimekizumab administered sc to subjects with PSO. AS0008 is a Phase 2, double-blind, randomized, placebo-controlled, multiple-dose study to evaluate the efficacy and safety of bimekizumab in subjects with active AS.

A Phase 2b dose-ranging study (PA0008) was designed to investigate the dose-response relationship, efficacy and safety of various bimekizumab dose regimens in subjects with active PsA. The current Phase 2b OLE study (PA0009) will allow access to bimekizumab for subjects who completed the lead-in study PA0008, while allowing the collection of further data on the long-term safety and efficacy of bimekizumab in this subject population.

Additional information on the clinical data for bimekizumab is available in the current version of the Investigator's Brochure (IB).

### 2.1.2 **Nonclinical studies**

Parallel inhibition of IL-17A and IL-17F has shown potent effects in a variety of animal models of inflammatory disease. Intravenously administered bimekizumab was well tolerated in repeat dose toxicology studies in Cynomolgus monkeys with a no adverse effect level (NOAEL) of 200mg/kg/week. The findings of note in toxicity studies were diarrhea related to infectious enteritis (observed in the single dose study) and asymptomatic mild colonic ulceration in a proportion of animals (in the repeat-dose study); this latter finding was not associated with hematology abnormalities. Data suggest that bimekizumab has induced primary lesions to the mucosa-associated lymphoid tissue via a pharmacologically related mechanism. In a second repeat-dose study, none of the minor apoptosis/necrosis findings observed in gut associated lymph nodes were seen. In animals given the highest dose of bimekizumab in the study (20mg/kg/week), a slightly higher number of protozoa (Balantidium coli) was observed in the cecum and color as compared to the control animals and low dose animals. Therefore, gut associated lymph node lesions observed in the first study are considered to be accidental and/or linked to exaggerated pharmacology and proliferation of Balantidium coli and are considered the result of a change in local mucosal immunity.

auditional inform version of the IB. Additional information on the nonclinical data for bimekizumab is available in the current

# STUDY OBJECTIVES

# **Primary objective**

The primary objective of this open-label study is to assess the long-term safety and tolerability of bimekizumab administered over a period of up to 100 weeks (~2 years).


### 3.2 Secondary objectives

The secondary objectives of the study are as follows:

To assess the long-term efficacy of bimekizumab

### 3.3 Other objectives

The other objectives are:

- To assess the impact on dactylitis and enthesitis
- To assess the impact on patient-reported quality of life
- To assess plasma concentrations of bimekizumab
- To assess the immunogenicity of bimekizumab

### 4 STUDY VARIABLES

Jextensions or variations thereof. All efficacy variables will be analyzed relative to the Baseline Visit of PA0008. Safety variables measured at the start of PA0009 will be referred to as PA0009 entry values.

### 4.1 **Primary variables**

### 4.1.1 **Primary safety variables**

The primary safety variables are the incidences of TEAEs and treatment-emergent SAEs.

### 4.2 Secondary variables

### 4.2.1 Secondary safety variable

The secondary safety variable is the withdrawal due to TEAEs.

### 4.2.2 Secondary efficacy variables

The secondary efficacy variables are:

- ACR20, ACR50, and ACR70 response at Week 48
- Change from Baseline of PA0008 in MASES at Week 48
- Change from Baseline of PA0008 in the LDI at Week 48
- PASI75 and PASI90 response at Week 48

### 4.3 Other variables

### 4.3.1 Safety variables

Other safety variables are listed below.

- Change from PA0009 Laboratory Baseline (defined as the earliest date in PA0009 at or prior to PA0009 Week 12) for clinical laboratory variables (hematology and biochemistry, excepting high-sensitivity C-reactive protein [CRP]) at each visit)
- Change from Baseline of PA0008 in vital signs (pulse, temperature, and blood pressure) and body weight

### 4.3.2 Efficacy variables

Other efficacy variables are listed below and will be evaluated at scheduled visits in accordance with the schedule of study assessments in Table 5–1.

- Change from Baseline of PA0008 in MASES

  Change from Baseline of PA0008 in MASES

  Change from Baseline of PA0008 in MASES

  Change from Baseline of PA0008 in MASES

- Change from Baseline of PA0008 in Psoriatic Arthritis Impact of Disease (PsAID)-9
- Change from Baseline of PA0008 in Short Form 36-item Health Survey (SF-36)
- Change from Baseline of PA0008 in the Hospital Anxiety and Depression Scale (HADS): HADS-Anxiety (HADS-A) and HADS-Depression (HADS-D) scores
- Depression and anxiety status "normal" as defined by HADS-D and HADS-A <8

### 4.3.3 PK variable

The PK variable is the plasma concentration of bimekizumab evaluated at scheduled visits up to 104 weeks (2 years) in accordance with the schedule of study assessments in Table 5–1.

### Immunological variable 4.3.4

The immunological variable is the anti-bimekizumab antibody detection evaluated at scheduled visits up to 104 weeks (2 years) in accordance with the schedule of study assessments in Table 5–1.

### 5 STUDY DESIGN

### Study description 5.1

PA0009 is a multicenter OLE study to assess the long-term safety, tolerability, and efficacy of bimekizumab in eligible adult subjects with PsA who completed the Phase 2b study PA0008. At Week 48 of PA0008, all eligible subjects continuing into PA0009 will undergo their final PA0008 study assessments and any nonoverlapping PA0009 entry assessments and will then receive their first open-label dose of bimekizumab.

The OLE study will assess the safety, tolerability, and efficacy of bimekizumab for a period of up to 100 weeks (~2 years). Bimekizumab will be administered at a dose of 160mg Q4W upon entry into PA0009, regardless of the dose received in PA0008.

Additionally, as described in (Section 5.1.1), other treatments may be used in addition to bimekizumab per Investigator discretion. Subjects not responding to treatment may be withdrawn from the treatment and study at the discretion of the Investigator.

A schedule of study assessments is presented in Table 5–1.

A study schematic diagram of PA0009 is presented in Figure 5–1.

### 5.1.1 Rescue therapy

The study duration for The study duration for each subject is estimated to be up to a maximum of 120 weeks:

Open-Label Treatment Period: up to 100 weeks (~2 vears)

SFU Visit: 20 --- 1

- SFU Visit: 20 weeks after the final dose of bimekizumab

The subject may remain in the study until the study ends after 120 weeks, until the Sponsor decides to close the study, or until bimekizumab development is stopped by the Sponsor, whichever comes first. The Sponsor may consider transitioning the subject into another bimekizumab study or program.

The end of the study is defined as the date of the last visit of the last subject in the study.

### 5.1.3 Planned number of subjects and sites

Up to 200 subjects from the ongoing PA0008 Phase 2b study could be enrolled into this study at any of the sites participating in PA0008

### Anticipated regions and countries 5.1.4

The regions planned for study conduct are the same as in PA0008 (Europe and North America).

### 5.2 Schedule of study assessments

rhis document cannot be used to support A schedule of study assessments is provided in Table 5–1.

Table 5–1: Schedule of study assessments

| Table 5–1: Schedul | e of s | tudy | ass | sess | mei | nts | | | | | | | | | | | | igi | Ö, | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Protocol activity | | | | | | | | Т | reatn | nent l | Perio | d | | | | | ~ `` | 101. | | SFU |
| Weeks <sup>a</sup> | EV <sup>b</sup> | 4 | 12 | 16 | 24 | 28 | 36 | 40 | 48 | 52 | 60 | 64 | 72 | 76 | 84 | 88 | 96 | 100 | W104/ | - |
| | | 8 | | 20 | | 32 | | 44 | | 56 | | 68 | | 80 | | 92 | | | ET | |
| Visit <sup>a</sup> | 1 | 2/3 | 4 | H <sup>c</sup> | 5 | H <sup>c</sup> | 6 | H <sup>c</sup> | 7 | H <sup>c</sup> | 8 | Hc | 9 | Hc | 10 | H <sup>c</sup> | 11 | 12 | 13 | |
| Informed consent | X <sup>d</sup> | | | | | | | | | | | | | 20 | 1 | | | | | |
| Inclusion/exclusion | Xe | | | | | | | | | | | | | 9.0 | | | | | | |
| Concomitant medications | Xf | X | X | | X | | X | | X | | X | *. | X. | | X | | X | X | X | X |
| Adverse events | Xf | X | X | | X | | X | | X | | X | (3) | X | | X | | X | X | X | X |
| eC-SSRS | X <sup>e,f</sup> | X | X | | X | | X | | X | 4 | X | 56// | X | | X | | X | X | X | X |
| HADS | X <sup>e,f</sup> | | X | | X | | X | | X( | ) .:((<br>() | 3X | | X | | X | | X | X | X | |
| HAQ-DI | X <sup>e,f</sup> | | X | | X | | X | _< | $\mathbf{x}$ | 130 | X | | X | | X | | X | X | X | |
| SF-36 | X <sup>e,f</sup> | | X | | X | | X | Ž) | NY. | | X | | X | | X | | X | X | X | |
| PGADA | X <sup>e,f</sup> | | X | | X | | X | | X | | X | | X | | X | | X | X | X | |
| PtAAP | X <sup>e,f</sup> | | X | | X | | X | | X | | X | | X | | X | | X | X | X | |
| PsAID-9 | X <sup>e,f</sup> | | X | | X | 2 | X | | X | | X | | X | | X | | X | X | X | |
| TB questionnaire | X <sup>e,f</sup> | | X | | X | 7 | X | | X | | X | | X | | X | | X | X | X | X |
| Vital signs (pulse,<br>temperature, BP) <sup>g</sup> | Xe | X | X | 20C | XX | | X | | X | | X | | X | | X | | X | X | X | X |
| Body weight | X <sup>e,f</sup> | | Xc | 76, | X | | X | | X | | X | | X | | X | | X | X | X | X |
| Physical examination <sup>h</sup> | X <sup>e,f</sup> | 5 | ý, | | | | | | X | | | | | | | | X | | X | X |
| TJC (78) and SJC (76) | X <sup>e,f</sup> | ree | X | | X | | X | | X | | X | | X | | X | | X | X | X | |
| BSA affected by PSO (BSA palm method) | Xed | | X | | X | | X | | X | | X | | X | | X | | X | X | X | |
| PASI <sup>i</sup> | X <sup>e,f</sup> | | X | | X | | X | | X | | X | | X | | X | | X | X | X | |
| MASES onfidential | X <sup>e,f</sup> | | X | | X | | X | | X | | | | X | | | | X | | X | |

Table 5–1: Schedule of study assessments

| Protocol activity | | | | | | | | T | reatn | nent ] | Perio | d | | | | | ď | 70 | | SFU |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Weeks <sup>a</sup> | EVb | 4 | 12 | 16 | 24 | 28 | 36 | 40 | 48 | 52 | 60 | 64 | 72 | 76 | 84 | 88 | 96 | 100 | W104/ | - |
| | | 8 | | 20 | | 32 | | 44 | | 56 | | 68 | | 80 | | 92 | | | ET | |
| Visita | 1 | 2/3 | 4 | Hc | 5 | Hc | 6 | Hc | 7 | Hc | 8 | H° | 9 | Hc | 10 | Hc | 11 | 12 | 13 | |
| LDI | X <sup>e,f</sup> | | X | | X | | X | | X | | X | | X | 20 | X | | X | X | X | |
| PhGADA | X <sup>e,f</sup> | | X | | X | | X | | X | | X | | X | 6 | X | | X | X | X | |
| ECG | X <sup>e,f</sup> | | | | | | | | X | | | | 20,0 | • | | | X | | X | |
| Hematology/biochemistry/<br>urine pregnancy <sup>j,k</sup> | X <sup>e,f</sup> | | X | | X | | X | | X | 7 | X | olica | X | | X | | X | X | X | X |
| Blood Sample for CRPk | X <sup>e,f</sup> | | X | | X | | X | | X | O <sub>S</sub> | X | ζ, | X | | X | | X | X | X | X |
| Blood sample for<br>bimekizumab plasma<br>concentrations <sup>k</sup> | $X^{e,f}$ | | X | | X | | X | S | X | 121 | 2, | | X | | | | X | | X | X |
| Blood sample for anti-<br>bimekizumab antibodies <sup>k</sup> | X <sup>e,f</sup> | | X | | X | < | X | | X | | | | X | | | | X | | X | X |
| IGRA TB test <sup>1</sup> | Xe | | | | | | Ko | | X | | | | | | | | X | | | X |
| IXRS | X | X | X | | X | 4 | X | | X | | X | | X | | X | | X | X | X | X |
| Bimekizumab administration | X | X | X | X | X | $\beta_{\rm X}$ | X | X | X | X | X | X | X | X | X | X | X | X | | |

BP=blood pressure; BSA=body surface area; CRP=C-reactive protein; eC-SSRS=electronic Columbia-Suicide Severity Rating Scale; ECG=electrogardiogram; ET=Early Termination; EV=Entry Visit; H=home; HADS=Hospital Anxiety and Depression Scale; HADD

ECG=electrocardiogram; ET=Early Termination; EV=Entry Visit; H=home; HADS=Hospital Anxiety and Depression Scale; HAQ-DI=Health Assessment Questionnaire—Disability Index; IGRA=interferon-gamma release assay; IXRS=interactive voice or web response system; LDI=Leeds Dactylitis Index; MASES= Maastricht Ankylosing Spondylitis Enthesitis Score; PASI=psoriasis area severity index; PGADA=Patient's Global Assessment of Disease Activity; PhGADA=Physician's Global Assessment of Disease Activity; PsAID=Psoriatic Arthritis Impact of Disease; PSO=psoriasis; PtAAP=Patient's Assessment of Arthritis Pain; SF-36=Short Form 36-item Health Survey; SFU=Safety Follow-Up; SJC=swollen joint count; TB=tuberculosis; TJC=tender joint count

Note: The SFU Visit will occur 20 weeks after the final dose of study medication.

<sup>&</sup>lt;sup>a</sup> Visit windows are ±7 days from the scheduled visit day (relative to the first dose) with a minimum of 21 days and a maximum of 35 days in between doses at all visits except the SFU Visit. For the SFU Visit (20 weeks after the final dose), the visit should occur no more than 3 days prior to the scheduled visit date and within 7 days after the scheduled visit date (-3 days/+7 days).

Table 5–1: Schedule of study assessments

| Protocol activity | | Treatment Period | | | | | | | | | | | SFU | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Weeks <sup>a</sup> | EV <sup>b</sup> | 4 | 12 | 16 | 24 | 28 | 36 | 40 | 48 | 52 | 60 | 64 | 72 | 76 | 84 | 88 | 96 | 100 | W104/ | - |
| | | 8 | | 20 | | 32 | | 44 | | 56 | | 68 | | 80 | | 92 | | | ET | |
| Visit <sup>a</sup> | 1 | 2/3 | 4 | H <sup>c</sup> | 5 | H <sup>c</sup> | 6 | H <sup>c</sup> | 7 | H <sup>c</sup> | 8 | Hc | 9 | Hc | 10 | H° | 11 | 12 | 13 | |

b PA0009 entry will occur at the end of the lead-study PA0008. At Week 48 of PA0008, all subjects continuing into PA0009 will undergo the final PA0008 study assessments and any nonoverlapping PA0009 entry assessments before receiving their first open-label dose of bimekizumab.

Confidentia

<sup>&</sup>lt;sup>c</sup> From the Entry Visit onwards, self-administration training will be provided to the subject/caregivers/appropriate designee by the study nurse. At Week 8 and Week 12, the subject/caregiver/appropriate designee will perform administrations under the supervision of the site staff to ensure that study medication is being properly and safely injected.

d Ensure that a separate Informed Consent form was completed by the subject for PA0009 prior to study entry.

<sup>&</sup>lt;sup>e</sup> To be performed prior to the first dose of open-label bimekizumab.

f Assessment will be performed at Week 48 of the lead-in study PA0008 and will be used as the PA0009 entry value.

g At PA0009 study entry collect pulse and BP prior to drug administration and then at 30 minutes and 1 hour after dosing. At all other visits collect pulse and BP prior to drug administration and once after dosing.

h Includes evaluation of signs and symptoms of active TB and risk for exposure to TB.

<sup>&</sup>lt;sup>1</sup> If the BSA affected by PSO was ≥3% at Baseline of PA0008, determine the PASI.

i If there has been a delay in menses, perform a urine pregnancy test.

<sup>&</sup>lt;sup>k</sup> All blood samples are to be taken prior to dosing.

<sup>&</sup>lt;sup>1</sup> It is recommended that the QuantiFERON TB Test be performed. This assessment will be performed at study entry, unless an IGRA negative result is available from less than 6 weeks prior to the first dose of open-label bimekizumab.

11 Dec 2019

PA0009

### 5.3 Schematic diagram

A study schematic diagram of PA0009 is provided in Figure 5–1.

Figure 5–1: Schematic diagram



IMP=investigational medicinal product; O4W=every 4 weeks; sc=subcutaneous; SFU=Safety Follow-up Note: Self-administration will be allowed after 3 months of treatment (from Week 16 onwards) as described in Table 5–1.

Note: Additionally, as described in (Section 5.1.1 and Section 7.8.1), other treatments may be used in addition to bimekizumab per Investigator discretion. Subjects not responding to treatment may be withdrawn from the study at the discretion of the Investigator.

<sup>a</sup> Subjects will receive their final dose of study drug on Week 100 and the SFU Visit will be conducted 20 weeks after the last dose of IMP.

### Rationale for study design and selection of dose 5.4

A dose of 160mg Q4W was selected based on the current understanding of PK/PD of bimekizumab in PsA (data from PA0007). Based on this analysis, a dose of 160mg Q4W is expected to provide an optimal response in most of the subjects. Based on the modeling outcome, UCB expects that the ACR50 response would maximize at 160mg Q4W, and hence, this dose was selected for PA0009.

A bimekizumab dose of 160mg Q4W is currently being used in ongoing Phase 2b clinical studies.

Doses greater than 160mg have been previously studied in the development of bimekizumab. In the single ascending dose study, UP0008, a single dose of bimekizumab 640mg was tested. In the multiple dose study, PA0007, a bimekizumab 560mg loading dose followed by 2 subsequent 320mg doses every 3 weeks was tested. At exposure levels achieved at these doses, the compound had no significant safety concerns. In the previous clinical studies, bimekizumab was administered av and in the current study bimekizumab will be administered sc (bioavailability of bimekizumab is 64%). Due to lower bioavailability, bimekizumab exposure is expected to be lower with sc administration compared with after iv administration, therefore, the dose regimens are expected to be

As more data for bimekizumab become available in this indication, doses and dosing regimen may be modified accordingly.

# 6 SELECTION AND WITHDRAWAL OF SUBJECTS

# 6.1 Inclusion criteria

To be eligible to participate in this study, all of the following criteria must be met:

1a. An Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written Informed Consent form is signed and dated by the subject.

Bimekizumab

- 2a. Subject is considered reliable and capable of adhering to the protocol (eg, able to understand and complete questionnaires), visit schedule, or medication intake according to the judgment of the Investigator.
- 3. In the opinion of the Investigator, the subject is expected to benefit from participation in an OLE study.
- 4. Subject completed PA0008 without meeting any withdrawal criteria.
- 5. **Female** subjects must be postmenopausal (at least 1 year), permanently sterilized (eg, tubal occlusion, hysterectomy, bilateral salpingectomy) or, if of childbearing potential (and engaged in sexual activity that could result in procreation), must be willing to use a highly effective method of contraception until 20 weeks after last administration of study medication, and have a negative pregnancy test at the last visit of PA0008. The following methods are considered highly effective when used consistently and correctly:
  - combined (estrogen and progestogen) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal)
  - progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
  - intrauterine device (IUD)
  - intrauterine hormone-releasing system (IUS)
  - bilateral tubal occlusion
  - vasectomized partner
  - sexual abstinence if it is in accordance with a subject's preferred and common lifestyle. Subjects who use abstinence as a form of birth control must agree to abstain from heterosexual intercourse until 20 weeks after the last dose of IMP. Study personnel must confirm the continued use of abstinence is still in accordance with the subject's lifestyle at regular intervals during the study.

Male subjects with a partner of childbearing potential must be willing to use a condom when sexually active, up until 20 weeks after the last administration of study medication (anticipated 5 half-lives).

### 6.2 **Exclusion criteria**

Subjects are not permitted to enroll in the study if any of the following criteria are met:

- 2. Subjects with any current sign or symptom that may indicate a medically significant active infection (except for the common cold) or has had an infection requiring systemic antibiodic within 2 weeks of study entry. The medical monitor must be a entry into PA0009 in such cases
- 3. Subjects who meet any withdrawal criteria in PA0008. For any subject with an ongoing SAE, or a history of serious infections (including hospitalizations) in the lead-in study, the Medical Monitor must be consulted prior to the subject's entry into PA0009.

### 6.3 Withdrawal criteria

Subjects are free to withdraw from the study at any time, without prejudice to their continued care.

Subjects should be withdrawn from the study and will be asked to complete the Early Termination (ET) Visit and SFU Visit (20 weeks after the last received dose) if any of the following events occur:

- 1. Subject withdraws his/her consent.
- 2. There is confirmation of a pregnancy in a female subject during the study, as evidenced by a positive pregnancy test.
- 3. The Sponsor or a regulatory agency requests withdrawal of the subject.
- 4. Subject develops an illness that in the opinion of the Investigator would interfere with his/her continued participation, if the risk of continuing participation outweighs the potential benefit.
- 5. Subject develops erythrodermic, guttate, or generalized pustular form of PSO.
- 6. Subjects considered to have either a suspected new latent tuberculosis (LTB) infection or who develops an active tuberculosis (TB) or nontuberculosis mycobacterium infection during the study (including but not limited to, conversion demonstrated by interferon-gamma release assay (IGRA) or other diagnostic means) must be immediately discontinued from study medication and an unscheduled visit must be conducted as soon as possible, but not later than the next regular visit.

The subject must be permanently withdrawn if further examinations result in a diagnosis of active TB, or if the subject is diagnosed with LTB infection with no initiation of prophylactic treatment, prematurely discontinues prophylactic treatment, or, in the opinion of the Investigator or Sponsor, is noncompliant with prophylactic TB therapy.

Confirmed active TB is an SAE and must be captured on an SAE Report form and provided to the Sponsor in accordance with SAE reporting requirements. As with all SAEs, periodic follow-up reports should be completed as per protocol requirements until such time as the TB infection resolves.

- 7. Subject is noncompliant with the study procedures or medications that may present a risk to the safety of the subject in the opinion of the Investigator.
- 8. Subject uses prohibited concomitant medications as defined in Section 7.8.2 that may present
- Subject develops laboratory abnormalities (with or without clinical symptoms) of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) as defined in Section 6.3.1; neutrophils <0.5x10<sup>9</sup>/L (neutropenia); lymphocytes <0.5x10<sup>9</sup>/L (lymphopenia). Any laboratory value or change judged to be clinically significant by the Inventor prompt consideration of whether the subject of product (IMP). For officer 9. Subject develops laboratory abnormalities (with or without clinical symptoms) of alanine Table 17-1 and Table 17-2 will be flagged to the Investigator and to the medical monitor but do not trigger mandatory withdrawal unless listed above. (Refer to Section 6.3.1 for withdrawal criteria in relation to potential drug-induced liver injury [PDILI].)
- 10. Subject has active suicidal ideation as indicated by a positive response ("Yes") to Questions 4 or 5 or to the suicidal behavior questions of the "Since Last Visit" version of the self-rated electronic Columbia-Suicide Severity Rating Scale (eC-SSRS). The subject should be referred immediately to a Mental Healthcare Professional and must be withdrawn from the study.
- 11. Subjects with a HADS-D score >15 must be withdrawn. Any subject who develops a HADS-D score of >10 during the study should be referred immediately to a Mental Healthcare Professional for further evaluation and potential withdrawal by the Investigator.
- 12. Subjects with newly diagnosed inflammatory bowel disease (IBD) or with IBD flares during the study must:
  - Be referred, as appropriate, to a health care professional treating IBD, such as a gastroenterologist
  - Discontinue IMP and be followed-up until resolution of active IBD symptoms

If IBD flares increase in severity or frequency during the study, the Investigator should use clinical judgment in deciding whether the subject should continue in the study and contact the Medical Monitor and UCB study physician to confirm the subject's suitability for continued participation in the study.

All subjects who withdraw from the study due to an AE must be followed until resolution of the event or until the event is considered stable. All subjects who withdraw from the study due to development of a laboratory abnormality must be closely monitored.

Investigators should attempt to obtain information on subjects in the case of withdrawal or discontinuation. For subjects considered lost to follow-up, the Investigator should make an effort (at least 1 phone call and 1 written message to the subject) and document his/her effort (date and summary of the phone call and copy of the written message in the source documents), to complete the final evaluation. All results of these evaluations and observations, together with a narrative description of the reason(s) for removing the subject, must be recorded in the source

Bimekizumab

documents. The electronic Case Report Form (eCRF) must document the primary reason for withdrawal or discontinuation.

Investigators should contact the Medical Monitor, whenever possible, to discuss the withdrawal of a subject in advance.

# 6.3.1 Potential drug-induced liver injury investigational medicinal product discontinuation criteria

Subjects with PDILI must be assessed to determine if IMP must be discontinued. In addition, all concomitant medications and herbal supplements that are not medically necessary should also be discontinued.

The PDILI criteria below require immediate discontinuation of IMP:

Subjects with either of the following:

- ALT or AST  $\geq$ 5x upper limit of normal (ULN)
- ALT or AST  $\ge 3xULN$  and coexisting total bilirubin  $\ge 2xULN$
- Subjects with ALT or AST ≥3xULN who exhibit temporally associated symptoms of hepatitis or hypersensitivity. Hepatitis symptoms include fatigue, nausea, vomiting, right upper quadrant pain or tenderness. Hypersensitivity symptoms include fever (without clear alternative cause), rash, or eosinophilia (ie, >5%).

The PDILI criterion below allows for subjects to continue on IMP at the discretion of the Investigator.

• Subjects with ALT or AST ≥3xULN (and ≥2x Baseline) and <5xULN, total bilirubin <2xULN, and no eosinophilia (ie, ≤5%), with no fever, rash, or symptoms of hepatitis (eg, fatigue, nausea, vomiting, right upper quadrant pain or tenderness).

Evaluation of PDILI must be initiated as described in Section 9.5.1.

If subjects are unable to comply with the applicable monitoring schedule, IMP must be discontinued immediately.

Investigators should attempt to obtain information on subjects in the case of IMP discontinuation to complete the final evaluation. Subjects with PDILI should not be withdrawn from the study until investigation and monitoring are complete. All results of these evaluations and observations, as well as the reason(s) for IMP discontinuation and subject withdrawal (if applicable), must be recorded in the source documents. The CRF must document the primary reason for IMP discontinuation.

# 7 STUDY TREATMENT

# Description of investigational medicinal product

Bimekizumab will be supplied by UCB Clinical Trial Supply Operations or designee.

The IMP will consist of the following:

• Bimekizumab will be supplied as a clear to opalescent, colorless to slightly brown, sterile, preservative–free solution in a 1mL prefilled syringe (PFS).

Further details of the IMP and specifications are provided in the Investigational Medicinal Product Handling Manual.

# 7.2 Treatment to be administered

All subjects will receive bimekizumab 160mg Q4W sc (Section 5.1).

The IMP (bimekizumab) will be administered at the visits indicated in Table 5–1. The minimum time between doses should be no less than 21 days and no more than 35 days for Q4W dosing.

The IMP is to be administered as 1 sc injection for the 160mg dose. Administration will occur at the study site for the first 3 months of PA0009.

Thereafter and in between the quarterly study visits at the site, the subjects will have the option to perform self-administration at home. From the Entry Visit onwards, self-administration training will be provided to the subject/caregivers/appropriate designee by the study nurse. At Week 8 and Week 12, the subject/caregiver/appropriate designee will perform administration under the supervision of the site staff to ensure that study medication is being properly and safely injected.

Once subjects/caregivers/appropriate designees as determined by the Investigator (or designee) have been trained, the study medication may be administered at home. The subject will receive the required number of injections at each visit needed to perform the monthly administrations at home. Subjects who are unable to or decide not to self-administer or those without a family member/friend/caregiver (or appropriate designee) who can help will not be discontinued but may continue to visit the site for only study treatment administration. If administered at home, the subject/caregiver (or appropriate designee) will document the date, body location, and time point of administration of study medication.

Suitable areas for sc injections are the lateral abdominal wall, upper outer thigh, and upper arm if the IMP is injected by a healthcare provider or a caregiver. Injection sites should be rotated and injections should not be given into areas where the skin is tender, bruised, red, or hard. It is also acceptable to inject in the upper arm if the preferred areas of the abdomen or thigh are covered in lesions, tender, or bruised.

An IMP Handling Manual will be provided to each site containing instructions regarding drug preparation and dosing.

# 7.3 Packaging

Bimekizumab will be packaged and labeled according to Good Manufacturing Practice (GMP) guidelines and applicable laws or regulations. It will be suitably packaged in such a way as to protect the product from deterioration during transport and storage. Further information regarding storage and transport conditions are provided in the IMP Handling Manual.

# 7.4 Labeling

Clinical drug supplies will be labeled in accordance with the current International Council for Harmonisation (ICH) guidelines on Good Clinical Practice (GCP) and GMP and will include any locally required statements. If necessary, labels will be translated into the local language.


# 7.5 Handling and storage requirements

Investigational Medicinal Product must be stored under refrigerated conditions (2°C to 8°C) protected from light. The IMP must not be frozen.

The investigator (or designee) is responsible for the safe and proper storage of IMP at the site. Investigational medicinal product stored by the investigator is to be kept in a secured area with limited access according to the storage conditions mentioned on the label.

Appropriate storage conditions must be ensured either by controlling the temperature (eg, room, refrigeration unit) or by completion of a temperature log in accordance with local requirements on a regular basis (eg, once a week), showing actual and minimum/maximum temperatures reached over the time interval.

In case an out-of-range temperature is noted, it must be immediately communicated to the Clinical Project Manager (CPM) (or designee) before further use of the IMP.

Investigational medicinal product will be shipped to the study sites in temperature-controlled containers. Out-of-range shipping or storage conditions must be brought to the attention of the Sponsor or designee, immediately. Authorization to use any out-of-range IMP must be documented and received prior to dispensing or administering the IMP at the study site.

The Investigator (or designee) will instruct the subject how to handle the IMP during the transport and how to store the IMP following the instruction guide. Cooler bags with freezer packs will be provided to the subjects. Specific attention will be put on the transport from site to home using cold bags; the subject will be instructed to put the IMP as quickly as possible into his/her refrigerator. In case of broken refrigerator or broken or lost syringes, the subject will inform the site immediately and new IMP will be prepared. All efforts should be made to follow the treatment schedule as per protocol.

# 7.6 Drug accountability

A Drug Accountability form will be used to record IMP dispensing and return information on a by-subject basis and will serve as source documentation during the course of the study. Details of any IMP lost, damaged (due to breakage or wastage), not used, partially used, disposed of at the study site, or returned to the sponsor or designee must also be recorded on the appropriate forms. All supplies and pharmacy documentation must be made available throughout the study for UCB (or designee) to review.

The Investigator (or designee) is responsible for retaining all used, unused, and partially used containers of IMP until returned or destroyed.

The Investigator may assign some of the Investigator's duties for drug accountability at the study site to an appropriate pharmacist/designee.

The Investigator must ensure that the IMP is used only in accordance with the protocol.

Periodically, and/or after completion of the clinical phase of the study, all used (including empty containers), partially used, unused, damaged, and/or expired IMP must be reconciled and either destroyed at the site according to local laws, regulations, and UCB Standard Operating Procedures (SOPs) or returned to UCB (or designee). Onsite destruction of used kits only may be allowed with prior approval from the Sponsor or designee after reconciliation. The

subjects/caregivers return the documentation together with any used/unused containers at the next scheduled clinic visit.

Investigational medicinal product intended for the study cannot be used for any other purpose

The IMP will be administered in the clinic during the first 3 months of treatment (Visit 1 [study entry] through Visit 4 [W12]) and compliance will be determined at the visit by study percention at home will be possible at Was 1 (4, 68, 76, 80, 88, and 92 Date 1). diary. All used PFS will be disposed of by subjects/caregivers/appropriate designee as determined by the Investigator in an acceptable disposal (sharps) container directly after the administration. The subjects/caregivers return the documentation together with any used/unused containers at the next scheduled clinic visit.

Drug accountability must be recorded on the Drug Accountability Form If a subject is noncompliant with the study procedures or medications that may present a risk to the safety of the subject in the opinion of the Investigator, then the subject should be withdrawn as described in Section 6.3.

### Concomitant medications/treatments 7.8

All concomitant medications, including over the counter products, herbal, traditional remedies, vitamin/mineral supplements, other dietary supplements, "nutraceuticals," and hormones must be recorded in the subject's source documentation (eg, clinical chart) and on the eCRF. This record should include the name of the drug, the dose, the route and date(s) of administration, and the indication for use.

The Investigator should examine the acceptability of all concomitant procedures, medications, topical preparations, and dietary supplements not explicitly prohibited in this study, and if necessary, discuss with the Medical Monitor.

In order to ensure that appropriate concomitant therapy is administered, subjects will be instructed to consult with the Investigator prior to taking any medication (either self-administered nonprescription drugs or prescription therapy prescribed by another physician).

### Permitted concomitant treatments (medications and therapies) 7.8.1

Medication changes are permitted at any time after enrollment into this extension study. Medication changes and additions are permitted with the following guidelines:

- Investigator as outlined below. Subjects may receive these add-on therapies while continuing to receive bimekizumab. Under no circumstances should subjects have a concomitant biologic agent while receiving bimekizumab.

   For subjects taking the subjects taking the subjects have a concomitant biologic agent while receiving bimekizumab.
  - made to a different NSAID/COX-2. Changes from an NSAID to a COX-2 inhibitor or from a COX-2 inhibitor to an NSAID are permitted up to the maximum approved or

11 Dec 2019

PA0009

- tolerated dose, whichever is less. Only 1 NSAID/COX-2 inhibitor may be taken at a given time.
- For subjects not taking NSAID/COX-2 inhibitors, either can be initiated, up to the maximum approved or tolerated dose, whichever is lower. Only 1 NSAID/COX-2 may be taken at a given time.
- Methotrexate may be added or increased to a maximum dose of 25mg/week, or the maximum tolerated dose, whichever is lower. The route of administration may be changed from oral to sc or from sc to oral. It is strongly recommended that subjects taking MTX should also take folic acid supplementation.
- Sulfasalazine may be given up to a maximum dose of 3g/day, or the maximum tolerated dose, whichever is lower, for peripheral arthritis symptoms.
- Leflunomide may be given at a maximum dose of 20mg/day (or an average of 20mg/day if not dosed daily), or the maximum tolerated dose, whichever is lower, for peripheral arthritis symptoms. Leflunomide should not be used concomitantly with MTX.
- Apremilast may be given at a maximum dose of 30mg twice daily, or the maximum tolerated dose, whichever is lower.
- Combination DMARDs (optimally 2) are allowed except that leflunomide and MTX may not be given together.
- No other oral DMARDs are permitted during this OLE study.
- Steroid tapers for disease activity or disease related reasons are allowed with an average daily dose of 20mg prednisone or prednisone equivalent per day for a maximum of 14 days.
- Up to 1 injection per joint for up to 3 discrete joints is permitted per 12-month period. Investigators should follow the guidance in the CRF instructions for proper scoring of the injected joints.
- Intra-articular hyaluronic acid injections are permitted into joints for which they are approved as per local labels.
- Intra-bursal corticosteroid injections are also permitted at the discretion of the Investigator.
- A decrease in dose or dosing frequency of any agent is permitted at any time.
- Subjects with persistent active disease in spite of added concomitant therapy/therapies mentioned above should be withdrawn from the study at the discretion of the Investigator.

# **Psoriasis treatments**

For freatment of PSO, subjects may continue to use topical moisturizers, emollients, salicylic acid preparations, bath oils, and oatmeal bath preparations for skin conditions during the study, as needed. Over-the-counter shampoos for the treatment of PSO of the scalp are also permitted. Mild topical steroids are permitted for use limited to the face, axillae, and/or genitalia, as needed. More potent topical steroids, topical retinoids, vitamin D analogues, and/or coal tar preparations may be used as medically required to treat a flare. Use of psoralen and ultraviolet A light (PUVA/UVA) therapy for the treatment of PSO is discouraged through the duration of the study.

# 7.8.2 Prohibited concomitant treatments (medications and therapies)

Prohibited and/or restricted medications are summarized in Table 7-1 and Table 7-2.

Table 7-1: Prohibited or restricted medications

| Drug class | Dose | Comments |
|---|---|---|
| Analgesics, including opioid analgesics (acetaminophen/paracetamol, etc) | Any dose | Any ad hoc use in the 24 hours prior to any study visit is prohibited. Stable doses of analgesics (including opioids) permitted. |
| TNF inhibitor: -infliximab -adalimumab -etanercept -golimumab -certolizumab pegol | Any dose | This applies to biosimilar versions of any TNF inhibitors. |
| Any non-TNF biologic medications | Any dose | Any exposure history is prohibited. |
| All other DMARDs | Any dose | Only permitted medications as per Section 7.8.1. |

DMARD=disease-modifying antirheumatic drug; TNF=tumor necrosis factor

Table 7-2: Additional prohibited psoriasis treatments

| Drug class | R. 11/10 |
|---|---|
| Phototherapy | ixer. |
| High potency topical s esters use except as de | teroid, vitamin D analogues, topical retinoids, keratolytics, coal tar, fumaric acid tailed in Section 7.8.1 |
| Systemic retinoids | OK |

Subjects who take prohibited medications may be withdrawn from study treatment but followed until the SFU Visit. The decision to withdraw a subject for taking prohibited medications should be made in consultation with the Medical Monitor.

# Vaccines 😞

Administration of live, attenuated vaccines is not allowed during the conduct of the study or for 20 weeks after the last dose of study drug. Administration of non-live, inactivated vaccines is allowed during the study at the discretion of the Investigator.

Live vaccinations include, but are not limited to, the following: anthrax vaccine, intranasal influenza vaccine, measles-mumps-rubella vaccine, polio live oral vaccine, smallpox vaccine, TB Bacillus Calmette-Guérin vaccine, typhoid live oral vaccine, varicella vaccine, and yellow fever vaccine.

# 7.9 Blinding

This is an open label study. All subjects' treatment assignments during the lead-in studies will remain blinded until final database lock of PA0008.

# 7.10 Randomization and numbering of subjects

This is an OLE study and no randomization will be performed. All subjects will receive bimekizumab 160mg Q4W sc.

Subjects will continue with the 5-digit subject numbers assigned by the interactive web or voice response system (IXRS) in the preceding study.

# 8 STUDY PROCEDURES BY VISIT

The schedule of study assessments (Table 5–1) provides a general overview of study assessments. A list of procedures to be completed at each visit is provided in the sections that follow.

- Visit windows of ±7 days on either side of the scheduled dosing are permitted for all visits other than the SFU Visit (see below); however, the Investigator should try to keep the subjects on the original dosing schedule. The window of ±7 days is relative to the first dose (PA0009 entry) and applicable for all subsequent visits. Changes to the dosing schedule outside of the 14-day window must be discussed with the Medical Monitor.
- The minimum time between doses should be no less than 21 days and no more than 35 days for Q4W dosing.
- For the SFU Visit (20 weeks after the last dose), the visit should occur no more than 3 days prior to the scheduled visit date and within 7 days after the scheduled visit date (-3 days/+7 days).

The Investigator should make efforts to maintain the original visit schedule. Changes to the dosing schedule outside of the allowed windows must be discussed with the Medical Monitor and may result in subject withdrawal.

# 8.1 Visit 1

The PA0009 entry assessments noted with an "\*" will be obtained at the Week 48 Visit of PA0008 and do not need to be recorded on the eCRF for this study.

The following procedures or assessments will be completed prior to administration of IMP:

- Ensure that a separate ICF is completed by the subject for PA0009 (must be done prior to any PA0009 study procedures)
- Assessment of inclusion/exclusion criteria
- Record concomitant medications\*
- Record AEs\*
- eC-SSRS\*
- HADS\*

- Administer the Health Assessment Questionnaire—Disability Index (HAQ-DI)\*
- Administer the SF-36\*
- Administer the Patient's Global Assessment of Disease Activity (PGADA)\*
- Administer the Patient's Assessment of Arthritis Pain (PtAAP)\*
- Administer the PsAID-9\*
- Administer the TB questionnaire\*
- Measure vital signs (temperature, pulse, and blood pressure [BP])\*
- Measure body weight\*
- Perform a physical examination, including an evaluation for signs and symptoms of active TB and risk for exposure to TB\*
- Perform tender joint count (TJC)/swollen joint count (SJC)\*
- Determine BSA affected by PSO using the BSA palm method\*
- If the BSA affected by PSO is ≥3% at Baseline of PA0008, determine the Psoriasis Area and Severity Index (PASI)\*
- Determine the MASES\*
- Determine the LDI\*
- Perform the Physician's Global Assessment of Disease Activity (PhGADA)\*
- Perform an electrocardiogram (ECG)\*
- Collect samples for hematology/biochemistry/urine pregnancy\*
- Collect blood sample for CRP\*
- Collect blood sample for bimekizumab plasma concentrations and anti-bimekizumab antibody detection\*
- Perform an IGRA TB test if applicable
- Record visit in the IXRS
- Bimekizumab will be administered after all of the above assessments have been completed. The following procedures or assessments will be completed following administration of IMP:
- Collect pulse and BP at 30 minutes and 1 hour after dosing

# 8.2 Week 4 (Visit 2) and Week 8 (Visit 3)

The following procedures or assessments will be completed prior to administration of IMP:

- Record concomitant medications
- Record AEs

11 Dec 2019 PA0009

- eC-SSRS
- Measure vital signs (temperature, pulse, and BP)
- Record visit in the IXRS
- 3 of Variations thereof. Bimekizumab will be administered after all of the above assessments have been completed

The following procedures or assessments will be completed following administration of IMP:

Collect pulse and BP once after dosing at any time

# Week 12 (Visit 4), Week 24 (Visit 5), Week 36 (Visit 6), and 8.3 Week 72 (Visit 9)

The following procedures or assessments will be completed prior to administration of IMP:

- Record concomitant medications
- Record AEs
- eC-SSRS
- **HADS**
- Administer the HAQ-DI
- Administer the SF-36
- Administer the PGADA
- Administer the PtAAP
- Administer the PsAID-9
- Administer the TB questionnaire
- Measure vital signs (temperature, pulse, and BP)
- Measure body weight
- Perform TJC/SJC
- Determine BSA affected by PSO using the BSA palm method
- If the BSA affected by PSO is ≥3% at Baseline of PA0008, determine the PASI
- Determine the MASES
- Determine the LDI

Perform the PhGADA

- Collect samples for hematology/biochemistry
- If there has been a delay in menses, perform a urine pregnancy test
- Collect blood sample for CRP


- Collect blood sample for bimekizumab plasma concentrations and anti bimekizumab antibody detection
- Record visit in the IXRS
- Bimekizumab will be administered after all of the above assessments have been completed

The following procedures or assessments will be completed following administration of IMP:

• Collect pulse and BP once after dosing at any time

# 8.4 Week 16, Week 20, Week 28, Week 32, Week 40, Week 44, Week 52, Week 56, Week 64, Week 68, Week 76, Week 80, Week 88, and Week 92

Subjects will be given the opportunity for self-administration of bimekizumab. Adverse events will be captured spontaneously if the subject decides to visit the site to receive the bimekizumab administration.

# 8.5 Week 48 (Visit 7) and Week 96 (Visit 11)

The following procedures or assessments will be completed prior to administration of IMP:

- Record concomitant medications
- Record AEs
- eC-SSRS
- HADS
- Administer the HAQ-DI
- Administer the SF-36
- Administer the PGADA
- Administer the PtAAP
- Administer the PsAID-9
- Administer the TB questionnaire
- Measure vital signs (temperature, pulse, and BP)
- Measure body weight
- Perform a physical examination, including an evaluation for signs and symptoms of active TB and risk for exposure to TB
- Perform TJC/SJC
- Determine BSA affected by PSO using the BSA palm method
- If the BSA affected by PSO is  $\ge 3\%$  at Baseline of PA0008, determine the PASI
- Determine the MASES
- Determine the LDI
- Perform the PhGADA
- Perform an ECG
- Collect samples for hematology/biochemistry
- If there has been a delay in menses, perform a urine pregnancy test
- Collect blood sample for CRP
- Collect blood sample for bimekizumab plasma concentrations and anti bimekizumab antibody detection
- Perform an IGRA TB test
- Record visit in the IXRS
- Bimekizumab will be administered after all of the above assessments have been completed. The following procedures or assessments will be completed following administration of IMP:
- Collect pulse and BP once after dosing at any time

# 8.6 Week 60 (Visit 8) and Week 84 (Visit 10)

The following procedures or assessments will be completed prior to administration of IMP:

- Record concomitant medications
- Record AEs
- eC-SSRS
- HADS
- Administer the HAQ-DI
- Administer the SF-36
- Administer the PGADA
- Administer the PtAAP
- Administer the PsAID-9
- Administer the TB questionnaire

Measure vital signs (temperature, pulse, and BP)

- Measure body weight
- Perform TJC/SJC
- Determine BSA affected by PSO using the BSA palm method
- If the BSA affected by PSO is ≥3% at Baseline of PA0008, determine the PASI

Determine the LDI

**UCB** 

- Perform the PhGADA
- Collect samples for hematology/biochemistry
- If there has been a delay in menses, perform a urine pregnancy test
- Collect blood sample for CRP
- Record visit in the IXRS
- Bimekizumab will be administered after all of the above assessments have been completed The following procedures or assessments will be completed following administration of IMP:

Collect pulse and BP once after dosing at any time
8.7 Week 100 (Visit 12)
The following procedures or assessments will be completed prior to administration of IMP:

- Record concomitant medications

- Administer the HAQ-DI
- Administer the SF-36
- Administer the PGADA
- Administer the PtAAP
- Administer the PsAID-9
- Administer the TB questionnaire
- Measure vital signs (temperature, pulse, and BP)
- Measure body weight
- Perform TJC/SJC
- Determine BSA affected by PSO using the BSA palm method
- If the BSA affected by PSO is ≥3% at Baseline of PA0008, determine the PASI
- Determine the LDI
- Perform the PhGADA
- Collect samples for hematology/biochemistry
- If there has been a delay in menses, perform a urine pregnancy test

- Collect blood sample for CRP
- Record visit in the IXRS

The following procedures or assessments will be completed following administration of IMP:

# 8.8

The following procedures or assessments will be completed:

- A IMP:

  A IMP:
  A IMP:
  A IMPRICATION
  A IMPRICATIO

- Determine the MASES
- Determine the LDI

Perform the PhGADA

- Perform an ECG
- Collect samples for hematology/biochemistry
- If there has been a delay in menses, perform a urine pregnancy test
- Collect blood sample for CRP

- Collect blood sample for bimekizumab plasma concentrations and anti bimekizumab antibody detection
- Record visit in the IXRS

# 8.9 SFU Visit (20 weeks after the final dose of IMP)

The following procedures or assessments will be completed:

- Record concomitant medications
- Record AEs
- eC-SSRS
- Administer the TB questionnaire
- Measure vital signs (temperature, pulse, and BP)
- Measure body weight
- Perform a physical examination, including an evaluation for signs and symptoms of active TB and risk for exposure to TB
- Collect samples for hematology/biochemistry
- If there has been a delay in menses, perform a urine pregnancy test
- Collect blood sample for CRP
- Collect blood sample for bimekizumab plasma concentrations and anti bimekizumab antibody detection
- Perform an IGRA TB test
- Record visit in the IXRS

# 8.10 Early Termination Visit

Subjects withdrawing early from the study (see Section 6.3) will undergo the same assessments as the Week 104 Visit (see Section 8.8) and will enter the SFU Period.

# 8.11 Unscheduled Visit

At the Investigator's discretion, an Unscheduled Visit may be completed at any time during the study but prior to the SFU Visit, if deemed necessary for the subject's safety and well-being.

If an Unscheduled Visit is conducted due to safety or efficacy reasons, an eC-SSRS assessment will be performed with the subject during the visit. If an Unscheduled Visit is conducted for reasons other than safety or efficacy concerns (eg, replacement of lost medication, repeated collection of a laboratory specimen due to collection or analysis issues) an eC-SSRS will not be required at these visits.

11 Dec 2019 PA0009

At this visit, any of the following assessments may be performed, depending on the reason for the visit:

- , pulse, and BP)
  ...auon
  record 12-lead ECG
  If medically indicated, obtain blood sample(s) for standard safety laboratory tests (hematology, serum chemistry)
  Obtain urine sample for standard safety laboratory tests (including women of childbearing potential).

  ASSESSMENT

### 9

#### 9.1 Adverse events

#### 9.1.1 **Definition of AE**

An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

In order to ensure complete safety data collection, all AEs occurring during the study (ie, after the signing of the ICF), including any pretreatment and posttreatment periods required by the protocol, must be reported in the eCRF even if no IMP was taken but specific study procedures were conducted. This includes all AEs not present prior to the initial visit and all AEs that recurred or worsened after the initial visit.

Signs or symptoms of the condition/disease for which the IMP is being studied should be recorded as AEs only if their nature changes considerably or their frequency or intensity increases in a chinically significant manner as compared to the clinical profile known to the investigator from the subject's history or study entry.

Adverse events that occurred during the PA0008 lead-in study and are still deemed ongoing at the time of enrolment (signed ICF) will be captured in the database and followed up, as described in Section 9.1.6.

### 9.1.2 **AEs of special interest**

An AE of special interest (AESI) is any AE that a regulatory authority has mandated be reported on an expedited basis, regardless of the seriousness, expectedness, or relatedness of the AE to the administration of a UCB product/compound.

Potential Hy's Law, defined as ≥3xULN ALT or AST with coexisting ≥2xULN total bilirubin in the absence of  $\geq 2xULN$  alkaline phosphatase (ALP), with no alternative explanation for the biochemical abnormality, must ALWAYS be reported to UCB as an AESI (ie, without waiting for any additional etiologic investigations to have been concluded). Follow-up information should then be reported if an alternative etiology is identified during investigation and monitoring of the subject.

### 9.1.3 Other safety topics of interest

Pre-specified safety topics of interest for the study are: infections (serious, opportunistic, fungal and TB), neutropenia, hypersensitivity, suicidal ideation and behavior, depression, major cardiovascular events, liver function test changes/enzyme elevations, malignancies, and inflammatory bowel diseases (with gastroenterology referral, as appropriate). This is based on findings from the IMP clinical program to date, potential risks generally associated with biologic immunomodulators, or findings from other medicines with a related mechanism of action. There are no specific AE reporting requirements for these topics, however special monitoring, additional data collection activities, and/or enhanced signal detection activities (within UCB) are in place.

### Procedures for reporting and recording AEs 9.1.4

The subject will be given the opportunity to report AEs spontaneously. A general prompt will also be given at each study visit to detect AEs. For example:

"Did you notice anything unusual about your health (since your last visit)?"

In addition, the Investigator should review any self-assessment procedures (eg, diary cards) employed in the study.

9.1.5 **Description of AEs**When recording an AE, the Investigator should use the overall diagnosis or syndrome using standard medical terminology, rather than recording individual symptoms or signs. The eCRF and source documents should be consistent. Any discrepancies between the subject's own words on his/her own records (eg. diary card) and the corresponding medical terminology should be clarified in the source documentation.

When recording the intensity of an AE in the CRF (ie, mild, moderate, or severe), the Investigator should use the following criteria:

- Mild: the subject is aware of the sign or symptom (syndrome), but it does not interfere with his/her usual activities and/or is of no clinical consequence
- Moderate: the AE interferes with the usual activities of the subject or it is of some clinical consequence

Severe: the subject is unable to work normally or to carry out his/her usual activities, or the AE is of definite clinical consequence

Details for completion of the AE eCRF (including judgment of intensity and relationship to IMP) are described in the eCRF Completion Guidelines.

### 9.1.6 Follow-up of AEs

An AE should be followed until it has resolved, has a stable sequelae, the Investigator If an AE is ongoing at the end of the study for a subject, follow-up should be provided until resolution/stable level of sequelae is achieved, or until the Investigator no longer deems the clinically significant, or until the subject is lost to follow-up. If no follow-up should be provided until Investigator must provide a justification. The follow-up. If no follow-up should be provided until Investigator must provide a justification. The follow-up. If no follow-up should be provided until Investigator must provide a justification. The follow-up should be provided until Investigator must provide a justification. determines that it is no longer clinically significant, or the subject is lost to follow-up. This

### 9.1.7 Rule for repetition of an AE

An increase in the intensity of an AE should lead to the repetition of the AE being reported with:

- The outcome date of the first AE that is not related to the natural course of the disease being the same as the start date of the repeated AE, and the outcome of "worsening"
- The AE verbatim term being the same for the first and repeated AE, so that the repeated AE can be easily identified as the worsening of the first one

### 9.1.8 **Pregnancy**

If an Investigator is notified that a subject has become pregnant after the first intake of any IMP, the Investigator must immediately notify UCB's PS department by providing the completed Pregnancy Report and Outcome Form (for contact details see SAE reporting information at the beginning of this protocol). The subject should be withdrawn from the study as soon as pregnancy is known (by positive pregnancy test), and the following should be completed:

- The subject should return for the ET Visit.
- The subject should immediately stop the intake of the IMP.
- An SFU Visit should be scheduled 20 weeks after the subject has discontinued her IMP.

The Investigator must inform the subject of information currently known about potential risks and about available treatment alternatives.

The pregnancy will be documented on the Pregnancy Report and Outcome Form provided to the Investigator. The progression of the pregnancy and the eventual birth (if applicable) must be followed up using the Pregnancy Report and Outcome Form in which the Investigator has to report on the health of the mother and of the child. Every reasonable attempt should be made to follow the health of the child for 30 days after birth for any significant medical issues. In certain circumstances, UCB may request that follow-up is continued for a period longer than 30 days. If the subject is lost to follow-up and/or refuses to give information, written documentation of attempts to contact the subject needs to be provided by the Investigator and filed at the site. UCB's PS department is the primary contact for any questions related to the data collection for the pregnancy, eventual birth, and follow-up.

In cases where the partner of a male subject enrolled in a clinical study becomes pregnant, the Investigator or designee is asked to contact the subject to request consent of the partner via the Partner Pregnancy Consent Form that has been approved by the responsible IRB/IEC and should be available in the Investigator site file. In case of questions about the consent process, the Investigator may contact the UCB/Contract Research Organization (CRO) contract monitor for the study. The Investigator will complete the Pregnancy Report and Outcome Form and send it to UCB's PS department (for contact details see SAE reporting information at the beginning of this protocol) only after the partner has agreed that additional information can be captured and has provided the signed Partner Pregnancy Consent Form. UCB's PS department is also the primary contact for any questions related to the data collection for the partner pregnancy, eventual birth, and follow-up.

A pregnancy becomes an SAE in the following circumstances: miscarriage, elective abortion when medically indicated (e.g. when pregnancy is endangering life or health of woman or when fetus will be born with severe abnormalities), unintended pregnancy after hormonal contraceptive failure (if the hormonal contraceptive was correctly used), ectopic pregnancy, fetal demise, or any congenital anomaly/birth defect of the baby. Those SAEs must be additionally reported using the Investigator SAE Report form.

# 9.1.9 Suspected transmission of an infectious agent via a medicinal product

For the purposes of reporting, any suspected transmission of an infectious agent via a medicinal product should be considered as an SAE; such cases must be reported immediately, recorded in the AE module of the eCRF, and followed as any other SAE. Any organism, virus, or infectious particle (eg, prion protein transmitting transmissible spongiform encephalopathy), pathogenic or nonpathogenic, is considered an infectious agent.

### 9.1.10 Overdose of investigational medicinal product

Excessive dosing (beyond that prescribed in the protocol and including overdose) should be recorded in the eCRF. Any SAE or nonserious AE associated with excessive dosing must be followed as any other SAE or nonserious AE. These events are only considered AEs or SAEs if there are associated clinical signs and symptoms or if the act of taking the excess medicine itself is an AE or SAE (eg, suicide attempt).

# 9.1.11 Safety signal detection

Selected data from this study will be reviewed periodically to detect as early as possible any safety concern(s) related to the IMP so that Investigators, clinical study subjects, regulatory authorities, and IRBs/IECs will be informed appropriately and as early as possible.

The Study Physician or medically qualified designee/equivalent will conduct an ongoing review of SAEs and perform ongoing SAE reconciliations in collaboration with the PS representative.

As appropriate for the stage of development and accumulated experience with the IMP, medically qualified personnel at UCB may identify additional safety measures (eg, AEs, vital signs, laboratory or ECG results) for which data will be periodically reviewed during the course of the study.

In addition, Cardiovascular and Neuropsychiatric Adjudication Committees will also periodically review and monitor the safety data from this study and advise UCB. Details are provided in the sions or variations thereof. Adjudication Committee Charters.

#### 9.2 **Serious AEs**

#### 9.2.1 **Definition of SAEs**

Once it is determined that a subject experienced an AE, the seriousness of the AE must be determined. An SAE must meet 1 or more of the following criteria:

- Death
- Life-threatening
- (Life-threatening does not include a reaction that might have caused death had it occurred in a more severe form.)
- Significant or persistent disability/incapacity
- Congenital anomaly/birth defect (including that occurring in a fetus)
- Important medical event that, based upon appropriate medical judgment, may jeopardize the patient or subject and may require medical or surgical intervention to prevent 1 of the other outcomes listed in the definition of serious.

(Important medical events may include, but are not limited to, potential Hy's Law [see Section 9.1.2], allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.)

Initial inpatient hospitalization or prolongation of hospitalization

A patient admitted to a hospital, even if he/she is released on the same day, meets the criteria for the initial inpatient hospitalization. An emergency room visit that results in admission to the hospital would also qualify for the initial inpatient hospitalization criteria. However, emergency room visits that do not result in admission to the hospital would not qualify for this criteria and, instead, should be evaluated for 1 of the other criteria in the definition of serious (eg, life-threatening adverse experience, important medical event).

Hospitalizations for reasons not associated with the occurrence of an AE (eg. preplanned surgery or elective surgery for a pre-existing condition that has not worsened or manifested in an unusual or uncharacteristic manner) do not qualify for reporting. For example, if a subject has a condition recorded on his/her medical history and later has a preplanned surgery for this condition, it is not appropriate to record the surgery or hospitalization as an SAE, since there is no AE upon which to assess the serious criteria. Please note that, if the pre-existing condition has worsened or manifested in an unusual or uncharacteristic manner, this would then qualify as an AE and, if necessary, the seriousness of the event would need to be determined.

Note: Confirmed active TB is always to be considered as an SAE and must be captured on an SAE Report Form and provided to the Sponsor in accordance with SAE reporting requirements. If an SAE is reported, UCB must be informed within 24 hours of receipt of this information by the site (see contact information for SAE reporting listed in the SAE Reporting section at the front of the protocol). The Investigator must forward to UCB (or its representative) a duly completed "Investigator SAE Report Form for Development Drug" (SAE report Form) provided by UCB, even if the data are incomplete, or if it is obvious that more data will be needed in order to draw any conclusions. Information recorded on this form will be entered into the global PS database.

An Investigator SAE report Form will be provided to the Investigator. The Investigator SAE Report Form must be completed in English.

It is important for the Investigator, when completing the SAE report Form, to include the assessment as to a causal relationship between the SAE and the IMP administration. This insight from the Investigator is very important for UCB to consider in assessing the safety of the IMP and in determining whether the SAE requires reporting to the regulatory authorities in an expedited manner.

Additional information (eg, autopsy or laboratory reports) received by the Investigator must be provided within 24 hours. All documents in the local language must be accompanied by a translation in English, or the relevant information included in the same document must be summarized in the Investigator SAE report Form.

The Investigator is specifically requested to collect and report to UCB (or its representative) any SAEs (even if the Investigator is certain that they are in no way associated with the IMP), up to 30 days from the end of the study for each subject, and to also inform participating subjects of the need to inform the Investigator of any SAE within this period. Serious AEs that the Investigator thinks may be associated with the IMP must be reported to UCB regardless of the time between the event and the end of the study.

Upon receipt of the SAE report Form, UCB will perform an assessment of expectedness of the reported SAE. The assessment of the expectedness of the SAE is based on the IB.

# 9.2.3 Follow-up of SAEs

An SAE should be followed until it has resolved, has a stable sequelae, the Investigator determines that it is no longer clinically significant, or the subject is lost to follow-up. This follow-up requirement applies to AEs, SAEs, AESIs, and other safety topics of interest; further details regarding follow-up of PDILI events are provided in Section 9.5.1.5. Information on SAEs obtained after clinical database lock will be captured through the PS database without limitation of time.

### 

The following AEs must be reported immediately:

- SAE: AE that the Investigator classifies as serious by the above definitions regardless of causality
- Suspected transmission of an infectious agent via a medicinal product
- AEs of special interest as defined in Section 9.1.2



### 9.4 **Anticipated SAEs**

The following list of Anticipated SAEs (Table 9–1) has been identified, as these events are Table 9-1: Anticipated SAEs for the next satisfactor of the study subject.

This list does not change the Investigator's obligation to report all SAEs (including Anticipated SAEs) as detailed in Section 9.2.2. anticipated to occur in the population studied in this protocol at some frequency that is

| MedDRA system organ class | MedDRA preferred term |
|---|---|
| Eye disorders | Uveitis |
| Cardiac disorders | Myocardial infarction Atrial fibrillation |
| Gastrointestinal disorders | Crohn's disease |
| Hepatobiliary disorders | Non-alcoholic steatohepatitis |
| Metabolism and Nutrition disorders | Metabolic syndrome<br>Diabetes mellitus |
| Musculoskeletal and connective tissue disorders | Psoriatic arthropathy |
| Neoplasms benign, malignant and unspecified (incl cysts and polyps) | Basal cell carcinoma Squamous cell carcinoma |
| Nervous system disorders | Embolic Stroke<br>Ischaemic Stroke |
| Psychiatric disorders | Anxiety<br>Depression |
| Skin and subcutaneous tissue disorders | Psoriasis |

MedDRA=Medical Dictionary for Regulatory Activities

Note: Exception: Eisted events will not be regarded as anticipated SAEs if they are life threatening or if they result in the death of the study subject.

### Laboratory measurements 9.5

Clinical laboratory assessments consist of serum chemistry, and hematology (Table 9-2). A centralized laboratory will be used to supply all laboratory test supplies and analyze all blood samples for hematology, and biochemistry measurements. Any unscheduled laboratory testing should also be collected using the central laboratory.

Specific details regarding the handling and processing of serum chemistry, hematology, and urinalysis samples are provided in the study laboratory manuals.

Clinical Study Protocol

**Table 9-2: Laboratory measurements** 

| Hematology | Chemistry | Urinalysis |
|---|---|---|
| Basophils | Calcium | Urine dipstick for pregnancy testing <sup>a</sup> |
| Eosinophils | Chloride | Urinalysis <sup>b</sup> |
| Lymphocytes | Magnesium | ii |
| Atypical lymphocytes | Potassium | Valid |
| Monocytes | Sodium | وما |
| Neutrophils | Glucose (random) | Elons |
| Hematocrit | BUN | tens |
| Hemoglobin | Creatinine | o and any or |
| MCH | AST | 20 |
| MCHC | ALT | |
| MCV | ALP | c alilo |
| Platelet count | GGT | Q. |
| RBC count | Total bilirubin | |
| WBC count | LDH KD Jahr | |
| | Total cholesterol | |
| | Uric acid | |
| | CRP Cill | |

ALP=alkaline phosphatase; ALT=alanine aminotransferase; AST=aspartate aminotransferase; BUN=blood urea nitrogen; CRP=C-reactive protein; GGT=gamma glutamyltransferase; LDH=lactate dehydrogenase; MCH=mean corpuscular hemoglobin, MCHC=mean corpuscular hemoglobin concentration; MCV=mean corpuscular volume

### 9.5.1 Evaluation of PDILI

The PDILI IMP discontinuation criteria for this study are provided in Section 6.3.1, with the accompanying required follow-up investigation and monitoring detailed below. All PDILI events must be reported as an AE and reported to the study site and sponsor within 24 hours of learning of their occurrence. Any PDILI event that meets the criterion for potential Hy's Law must be reported as an AE of special interest (see Section 9.1.2), and, if applicable, also reported as an SAE (see Section 9.2.2).

Evaluation of PDILI consists of the diagnostic testing and continued monitoring included in Table 9-3 (specific tests dependent on laboratory results and corresponding symptoms) and consultation with a local hepatologist (if applicable; discussed in Section 9.5.1.1). The local hepatologist is the expert usually consulted by the treating physician for assessment and

<sup>&</sup>lt;sup>a</sup> A urine pregnancy test will be performed for women of childbearing potential if there is a suspicion of pregnancy or a delay in menses. A positive urine pregnancy test should always be confirmed with a serum

<sup>&</sup>lt;sup>b</sup> These measurements will be performed only if a urinalysis is required for safety reasons.

management of potential hepatic disease. This would usually be a hepatologist but may be a gastroenterologist. Additional investigation and monitoring may be required and adapted based Variations thereof. on the diagnosis after the cause of the liver injury/abnormality is confirmed (details in Section 9.5.1.5).

The results of all monitoring, including laboratory testing and other testing, should be made available to the study site and sponsor.

All initial tests resulting in abnormal hepatic laboratory values need to be repeated, but appropriate medical action must not be delayed waiting for the repeat result.

If tests are done locally for more rapid results, a concurrent sample should also be sent to the central laboratory whenever possible. Medical care decisions are to be made initially using the most rapidly available results and a conservative approach must be taken if the results from the 2 laboratory tests are significantly different. Data from the local and central laboratory are to be recorded on the applicable eCRF pages.

When IMP is discontinued, all concomitant medications and herbal supplements that are not medically necessary should also be discontinued. In these cases, the Investigator should also consider dose reduction for medically necessary concomitant medication and consider changing any medically required concomitant medication known to be hepatotoxic to a suitable alternative.

Rechallenge with a substance potentially causing drug-induced liver injury is dangerous, may be o investiga arting arti fatal, and must not occur.

Table 9-3 summarizes the approach to investigate PDILI.

**Table 9-3:** Required investigations and follow-up for PDILI

| | | red investigatio | ns and follow-up fo | | T | Jajidji |
|---|---|---|---|---|---|---|
| | atory value | | Immediate | | | Follow-up |
| ALT or<br>AST | Total<br>bilirubin | Symptoms <sup>a</sup> of<br>hepatitis or<br>hypersensitivity | Consultation requirements | Actions | Testing | Evaluation |
| ≥3xULN | ≥2xULN <sup>b</sup> | NA | Hepatology consult. <sup>c</sup> Medical Monitor must be notified within 24 hours | Immediate IMP discontinuation. | Essential: Must have<br>repeat liver chemistry<br>values and additional<br>testing completed | Monitoring of liver chemistry values at least twice per week until values normalize, stabilize, or return to within Baseline values. <sup>d</sup> |
| ≥3xULN | NA | Yes | and subject discussed with Medical Monitor ASAP. | and subject discussed with | ASAP (see<br>Section 9.5.1.4);<br>Precommended to | |
| ≥5xULN | NA | NA | Need for hepatology consult to be discussed. (required if ALT or AST ≥8xULN) Medical Monitor must be notified within 24hours (eg, by laboratory alert) and subject discussed with Medical Monitor ASAP. | Immediate IMP discontinuation | occur at the site with HCP. | |
| Confidential This document cannot be used to support any marketing. | | | | | | |
| | | anot be used | | | | |

Table 9-3: Required investigations and follow-up for PDILI

| Laborate | ory value | | Immediate | | | Follow-up |
|---|---|---|---|---|---|---|
| ALT or<br>AST | Total<br>bilirubin | Symptoms <sup>a</sup> of<br>hepatitis or<br>hypersensitivity | Consultation requirements | Actions | Testing | Evaluation |
| ≥3xULN<br>(and ≥2x<br>baseline) and<br><5xULN<br>(and ≥2x<br>baseline) | <2xULN | No | Discussion with Medical Monitor required. Consider need for hepatology consult if there is no evidence of resolution (see Follow-up requirements) c | Further investigation – immediate IMP discontinuation not required (see Section 9.5.1.2). IMP discontinuation required if any of the following occur: Subject eannot comply with monitoring schedule. Liver chemistry values continue to increase Liver chemistry values remain ≥3xULN (and ≥2xbaseline) after 2 weeks of monitoring without evidence of resolution | Essential: Every attempt must be made to have repeat liver chemistry values and additional testing completed within 48hours at the site with HCP (see Section 9.5.1.4). | <ul> <li>Monitoring of liver chemistry values at least twice per week for 2 weeks.<sup>d</sup></li> <li>Immediate IMP discontinuation required if liver chemistry values continue to increase.</li> <li>After 2 weeks of monitoring liver chemistry values:</li> <li>Discontinue IMP if levels remain ≥3xULN (and ≥2x baseline) without evidence of resolution<sup>d</sup></li> <li>Continue to monitor until values normalize, stabilize, or return to within Baseline values<sup>d</sup>.</li> </ul> |

ALP=alkaline phosphatase; ALT=alanine aminotransferase; ASAP=as soon as possible; AST=aspartate aminotransferase; HCP=healthcare practitioner; IMP=investigational medicinal product; NA=not applicable; PDILI=potential drug induced liver injury; ULN=upper limit of normal

<sup>&</sup>lt;sup>a</sup> Hepatitis symptoms include fatigue, nausea, vomiting, and right upper quadrant pain or tenderness; hypersensitivity symptoms include eosinophilia (>5%), rash, and fever (without clear alternative cause).

<sup>&</sup>lt;sup>b</sup> If the subject also has  $\ge 2xULN$  ALP, the possibility of an indication of biliary obstruction should be discussed with the Medical Monitor.

<sup>&</sup>lt;sup>c</sup> Details provided in Section 9.5.1.1. The local hepatologist is the expert usually consulted by the treating physician for assessment and management of potential hepatic disease. This would usually be a hepatologist but may be a gastroenterologist.

<sup>&</sup>lt;sup>d</sup> Unless an alternative monitoring schedule is agreed by the investigator and UCB responsible physician. Determination of stabilization is at the discretion of the investigator in consultation with the hepatologist (as applicable) and UCB responsible physician, as needed.

### 9.5.1.1 Consultation with Medical Monitor and local hepatologist

Potential drug-induced liver injury events require notification of the Medical Monitor within sions of variations thereof. 24 hours (eg, by laboratory alert), and the subject must be discussed with the Medical Monitor as soon as possible. If required, the subject must also be discussed with the local hepatologist. The local hepatologist is the expert usually consulted by the treating physician for assessment and management of potential hepatic disease. This would usually be a hepatologist but may be a gastroenterologist. If determined necessary, this discussion should be followed by a full hepatology assessment (see Section 9.5.1.4) and SAE report (if applicable).

#### 9.5.1.2 Immediate action: determination of IMP discontinuation

All PDILI events require immediate action, testing, and monitoring.

The immediate action is dependent on the laboratory values and symptoms of hepatitis or hypersensitivity and ranges from continuation of IMP (followed by immediate investigation) to immediate discontinuation (see Section 6.3.1 and Table 9-3 for details).

When IMP is discontinued, all concomitant medications and herbal supplements that are not medically necessary should also be discontinued. The Investigator should also consider dose reduction for medically necessary concomitant medication and consider changing any medically required concomitant medication known to be hepatotoxic to a suitable alternative.

### 9.5.1.3 IMP restart/rechallenge

Rechallenge with a substance potentially causing drug-induced liver injury is dangerous, may be fatal, and must not occur.

### Testing: identification/exclusion of alternative etiology 9.5.1.4

The measurements and additional information required for the assessment of PDILI events when there is a reasonable possibility that they may have been caused by the IMP are included, but not limited to those listed in Table 9–4 (laboratory measurements) and Table 9–5 (additional information). Results of the laboratory measurements and information collected are to be submitted to the sponsor on the corresponding eCRF. If the medical history of the subject indicates a requirement for other assessments not included below, these additional assessments should be completed and submitted, as applicable.

All blood samples should be stored, if possible. If tests are done locally for more rapid results, a concurrent sample must also be sent to the central laboratory.

The measurements to be assessed are detailed in Table 9-4.

### Table 9-4: PDILI laboratory measurements

| Virology- | Hepatitis A IgM antibody |
|---|---|
| related | HBsAg |
| | Hepatitis E IgM antibody |
| | HBcAb-IgM |
| | Hepatitis C RNA |
| | Cytomegalovirus IgM antibody |
| | Epstein-Barr viral capsid antigen IgM antibody (if unavailable, obtain heterophil antibody or monospot testing) |
| Immunology | Anti-nuclear antibody (qualitative and quantitative) |
| | Anti-smooth muscle antibody (qualitative and quantitative) |
| | Type 1 anti-liver kidney microsomal antibodies (qualitative and quantitative) |
| Hematology | Eosinophil count |
| Urinalysis | Toxicology screen <sup>a</sup> |
| Chemistry | Amylase |
| | ALT, AST |
| | If total bilirubin ≥1.5xULN, obtain fractionated bilirubin to obtain % direct bilirubin |
| | Serum CPK and LDH to evaluate possible muscle injury causing transaminase elevation |
| Additional | Prothrombin time/INR |
| | Serum pregnancy test |
| | PK sample |

ALT=alanine aminotransferase; AST=aspartate aminotransferase; CPK=creatine phosphokinase; HBcAb-IgM=hepatitis B core antibody.IgM; HBsAg=hepatitis B surface antigen; IgM=immunoglobulin M; INR=international normalized ratio; LDH=lactate dehydrogenase; PDILI=potential drug-induced liver injury; PK=pharmacokinetic; RNA=ribonucleic acid; ULN=upper limit of normal

<sup>&</sup>lt;sup>a</sup> For detecting substances (ie, amphetamines, benzodiazepines, opioids, marijuana, cocaine, phencyclidine, and tricyclic antidepressants), additional tests may be performed based on the Investigator's medical judgment and patient's history.

patient's history.

b Measured only for subjects with ALT >8xULN, elevations in total bilirubin, and symptoms of hepatitis or hypersensitivity. Hepatitis symptoms include fatigue, nausea, vomiting, and right upper quadrant pain or tenderness; hypersensitivity symptoms include eosinophilia (>5%), rash, and fever (without clear alternative cause).

11 Dec 2019 PA0009

The following additional PDILI information is to be collected (Table 9–5):

#### Table 9–5: PDILI information to be collected

New or updated information

Concomitant prescription and over-the-counter medications (eg., acetaminophen, herbal remedies, vitamins); dosages and dates should be included.

Pertinent medical history, including the following:

- History of liver disease (eg, autoimmune hepatitis, nonalcoholic steatohepatitis or other "fatty liver disease")

  Adverse reactions to drugs

  Allergies

  Relevant familie 1.

- Relevant family history or inheritable disorders (eg, Gilbert's syndrome, alpha-1 antitrypsin deficiency)
- Recent travel
- Progression of malignancy involving the liver (Note: Metastatic disease to the liver, by itself, should not be used as an explanation for significant AST and/or ALT elevations.)

The appearance or worsening of clinical symptoms of hepatitis or hypersensitivity (eg., fatigue, nausea, vomiting, right upper quadrant pain or tenderness, decreased appetite, abdominal pain, jaundice, fever, or rash)

Recent clinically significant hypotension of hypoxemia with compromised cardiopulmonary function

Alcohol and illicit drug use

Results of liver imaging or liver biopsy, if done

Results of any specialist or hepatology consult, if done

Any postmortem/pathology reports

ALT=alanine aminotransferase AST=aspartate aminotransferase; PDILI=potential drug-induced liver injury

#### 9.5.1.5 Follow-up evaluation

Potential drug-induced liver injury events require follow-up monitoring as described in Table 9-3. Monitoring should continue until liver chemistry values normalize, stabilize, or return to baseline. Determination of stabilization is at the discretion of the Investigator in consultation with the hepatologist (as applicable) and UCB responsible physician, as needed.

# Other safety measurements

### Vital signs

The Investigator or designee should measure all vital signs (systolic and diastolic BP, temperature [oral, axillary, or otic], pulse rate) after the subject has been sitting for at least 5 minutes, and the subject should remain seated during the measurements. Body temperature should be obtained prior to dosing with IMP at study visits when IMP is administered. At PA0009 study entry, collect pulse and BP prior to drug administration and then at 30 minutes

and 1 hour after dosing. At all other visits collect pulse and BP prior to drug administration and once after dosing (any time).

#### 9.6.2 **Body weight**

The Investigator or designee will measure the weight of the subject in kilograms at the time points listed in Table 5–1. The same scale should be utilized throughout the study where possible.

#### 9.6.3 Physical examination

Valiations thereof. The physical examination should be conducted by the Investigator or designee at the time points listed in Table 5–1 and will include general appearance; ear, nose, and throat; eyes, hair, and skin; respiratory; cardiovascular; gastrointestinal; musculoskeletal; hepatic; neurological (including limb reflexes); and mental status. Findings considered clinically significant changes since the physical examination at the Baseline of PA0008 will be recorded as AEs.

#### 12-lead ECG 9.6.4

The Investigator or designee will perform the ECG at the time points listed in Table 5–1. The ECGs will be read locally.

### Tuberculosis and TB risk factor assessment and management 9.6.5

All subjects will be assessed for TB at prior to administration of IMP in PA0009 and at the time points specified in the schedule of study assessments (Table 5–1) through physical examination for signs and symptoms of TB, laboratory testing (Section 9.6.5.1), and subject questionnaire (Section 9.6.5.2).

Prior to administration of IMP, subjects will have an IGRA test (QuantiFERON TB Test is recommended) and examination for signs and symptoms of TB unless an IGRA negative result is available less than 6 weeks prior to the first dose of open-label bimekizumab. In addition, each subject will complete a TB questionnaire with questions directed at symptoms of TB and potential exposure to TB.

### **Test Conversion**

Tuberculosis test conversion is defined as a positive IGRA result for the current test, when previous IGRA test results were negative. All subjects with TB test conversion must immediately stop IMP administration. In case of a TB test conversion, the subject must be considered as having either a suspected new latent or an active TB infection and be promptly referred to an appropriate specialist (eg. pulmonologist, infectious disease specialist) for further evaluation. If test conversion indicates LTB infection, active TB, or nontuberculous mycobacteria (NTMB) then, per UCB TB working instructions, TB test conversion (confirmed) should be classified adequately, either as due to LTB infection, active TB infection, or NTMB, respectively. Additional assessments (eg, blood tests or IGRA, chest x-rays, or other imaging) should be performed where medically relevant and documented. Such conversions should be reported to the UCB PS function.

### Latent TB

In case the evaluation by the appropriate specialist indicates a new LTB infection during the study, a prophylactic TB treatment should be initiated, and the IMP can be continued no sooner **UCB** 11 Dec 2019 Bimekizumab PA0009

than 4 weeks after start of prophylactic TB treatment, if it is deemed likely by the Investigator that prophylactic TB treatment is continued to completion.

If prophylaxis is not initiated, the subject must be withdrawn.

Every related action should be discussed in advance with the Medical Monitor.

Once withdrawn from study treatment, subjects should return for the ET Visit, complete all ET Visit assessments, and complete a SFU Visit (20 weeks after the last dose of IMP).

### Active TB or NTMB infection

Subjects who develop active TB or NTMB infection during the study must be withdrawn from the study. The subject must be immediately discontinued from IMP and an ET Visit must be scheduled as soon as possible, but no later than the next scheduled visit. The subject should be encouraged to keep the SFU Visit as specified by the protocol. Treatment should be started immediately.

Note that subjects with history of NTMB or active NTMB infection are excluded from the study regardless of prior or current therapy for this condition.

### 9.6.5.1 **Tuberculosis assessment by IGRA**

During conduct of the study, the TB assessment by IGRA (QuantiFERON TB Test is recommended) will be performed at study entry (unless an IGRA negative result is available less than 4 weeks prior to the first dose of open-label bimekizumab) and should be repeated at Week 48, Week 96, and SFU Visits for all subjects. The test results will be reported as positive, negative, or indeterminate. UCB also recommends that a TB specialist be consulted where TB (latent or active) is suspected or if there are doubts regarding test results. If latent or active TB is identified, subject must undergo appropriate study-specified withdrawal procedures.

### **Tuberculosis questionnaire** 9.6.5.2

The questionnaire "Evaluation of signs and symptoms of tuberculosis" should be used as a source document. The questionnaire will be completed at PA0009 entry, every 12 weeks throughout the study, at Week 104, and at the SFU Visit (Table 5-1). The questionnaire will assist with the identification of subjects who may require therapy for TB. A "Yes" response to any of the questions during the study should trigger further assessments to determine if the subject has either LTB or active TB infection.

Subjects with a confirmed latent TB (where no prophylactic treatment is initiated) or active TB infection must be withdrawn from the study (as further detailed in Section 9.6.5).

# **Tuberculosis management**

# LTB infection and active TB identified during study

During the study, subjects who develop evidence of LTB infection or active TB must immediately stop further administration of IMP and will be referred to an appropriate TB specialist (pulmonologist or infectious disease specialist) for further evaluation. Evidence of LTB infection is defined as subject's IGRA test converts to positive or indeterminate (and confirmed indeterminate on repeat), or the subject's questionnaire or history and physical indicates that TB infection or exposure may have occurred. Evidence of active TB includes, in addition to the aforementioned tests, signs, and symptoms of organ involvement. In either



situation, the subject should be carefully assessed by a TB specialist for active TB. Subjects diagnosed with active TB or LTB infection should be withdrawn from the study and receive appropriate TB or prophylaxis therapy.

Any presumptive diagnosis or diagnosis of a TB infection is a reportable event. Confirmed active TB must be reported as an SAE. The Investigator is to complete and submit the TB follow we form provided.

The subject of the subject

The subject should be transferred to the care of his/her physician and managed according to the best available standard of care. Subjects identified as having converted to active TB during the study must be withdrawn and scheduled to return for the ET Visit as soon as possible, but no later than the next scheduled study visit and complete all ET Visit assessments.

The subject should be encouraged to complete a SFU Visit (20 weeks after the last dose of IMP).

If infection with NTMB is identified during the study, the same procedure as for active TB acquired during the study must be followed.

#### 9.6.6 Pregnancy testing

A urine pregnancy test will be performed at any scheduled or unscheduled visit if there is suspicion of pregnancy and will be confirmed with a serum pregnancy test if the urine test is positive.

Pregnancy test results must be negative prior to administering IMP.

### Assessment of suicidal ideation and behavior 9.6.7

Suicidal ideation and behavior will be assessed by trained study personnel using the eC-SSRS. This scale will be used to assess suicidal ideation and behavior that may occur during the study. The visits at which the eC-SSRS assessments will be performed are specified in the schedule of study assessments (Table 5-1).

The eC-SSRS is a standardized and validated instrument developed for the assessment of the severity and frequency of suicidal ideation and behavior (Posner et al, 2011; Mundt et al, 2010). Subjects respond to standardized clinical questions that are presented in a uniform fashion. The eC-SSRS defines 5 subtypes of suicidal ideation and behavior in addition to self-injurious behavior with no suicidal intent. The eC-SSRS takes approximately 3 to 10 minutes to complete.

### ASSESSMENT OF EFFICACY 10

Several assessments must be completed in order to determine the ACR response. These include the TJC and SJC based on 78 and 76 joints, respectively, PGADA, PhGADA, PtAAP, HAQ-DI, and CRP. The methods for the component measures will be described first, followed by ACR response and assessments used in secondary and other efficacy variables.

The timing for all assessments is specified in the schedule of study assessments (Table 5–1).

### 10.1 78/76 joint evaluation for ACR response

The Principal Investigator, another delegated physician, or an appropriately qualified medical professional (based on local requirements) who has had documented training on how to perform

these assessments correctly assesses the following joints for tenderness: the distal interphalangeal, proximal interphalangeal and metacarpophalangeal joints of the hands, and metatarsophalangeal joints of the feet, the carpometacarpal and wrist joints (counted separately), Artificial and ankylosed joints, as well as missing joints (ie, amputated joints), are excluded from both tenderness and swelling assessments.

One dactylitic digit is to be counted as 1 swollen joint (instead of counting as 3 in the finger or 2 in the toe).

Table 10–1 summarizes the swall:

Table 10–1: Swelling and tenderness grading

| Grade | Swelling response (76) | Tenderness response (78) |
|-------|--------------------------------|--------------------------|
| 0 | None | Not tender |
| 1 | Detectable synovial thickening | Tenderness present |

# 28 joint evaluation for determination of DAS28(CRP) 10.2

The following 28 joints will be used for calculation of the DAS28(CRP).

- Upper extremity (26)-bilateral shoulders, elbows, wrists (includes radiocarpal, and carpal and carpometacarpal bones considered as a single unit), metacarpophalangeal (MCP) I, II, III, IV, and V, thumb interphalangeals (IP), proximal interphalangeal (PIP) II, III, IV, and V
- Lower extremity (2)-knees

### Patient's Global Assessment of Disease Activity 10.3

Subjects will score their Global Assessment of Disease Activity using a visual analog scale (VAS) where 0 is "very good, no symptoms" and 100 is "very poor, severe symptoms".

The subject should be asked to consider both joint and skin components in their response to this question.

### Physician's Global Assessment of Disease Activity 10.4

The Investigator will assess the overall status of the subject with respect to their PsA signs and symptoms and functional capacity (considering both joint and skin components) using a VAS where 0 is "very good, asymptomatic and no limitation of normal activities" and 100 is "very poor, very severe symptoms which are intolerable and inability to carry out all normal activities".

This assessment by the Investigator should be made blind to the PGADA.

#### 10.5 Patient's Assessment of Arthritis Pain

The Patient's Assessment of Arthritis Pain VAS or 'Pain VAS' is part of the ACR core set of measures in arthritis (Felson et al, 1993). Subjects will assess their arthritis pain using a VAS where 0 is "no pain" and 100 is "most severe pain".

# 10.6 Health Assessment Questionnaire-Disability Index score

The HAQ-DI contains 20 items divided into 8 domains that measure: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. Subjects are required to indicate the degree of difficulty they have experienced in each domain in the past week on a 4-point scale that ranges from 0 (without difficulty) to 3 (unable to do). Any individual score of less than 2 is adjusted to 2 if the activity requires assistance from another individual or the use of an assistive device. The highest score in each category is then summed (0 to 24) and divided by the number of categories scored to give a score that ranges from 0 to 3.

### 10.7 CRP levels

C-reactive protein levels will be analyzed by the central laboratory.

# 10.8 ACR20, ACR50, and ACR70 response

The ACR20, ACR50, and ACR70 response rates are based on a 20%, 50%, and 70% or greater improvement relative to Baseline of PA0008 in the following measures:

- TJC based on 78 joints
- SJC based on 76 joints
- 3 of the 5 remaining core set measures:
  - PGADA
  - PhGADA
  - PtAAP
  - HAQ-DI
  - CRP

### 10.9 BSA-PSO

The BSA palm method will be used for the evaluation of BSA affected by PSO as follows:

The subject's hand, including the palm, fingers and thumb, is used as the reference point for measuring how much of their skin is affected by PSO, representing roughly 1% of the body's surface.

- Subject's palm=1%
- Head and neck=10% (10 palms)
- Upper extremities=20 % (20 palms)
- Trunk=30% (30 palms)
- Lower extremities=40 % (40 palms)

Total BSA=100%

### 10.10 Psoriasis Area and Severity Index (PASI)

Psoriasis Area and Severity Index will be assessed in all subjects with study entry BSA affected by PSO  $\geq$ 3% at Baseline of PA0008 determined by the method described in Section 10.9 (ie, the BSA palm method).

The PASI is the most commonly used and validated assessment for grading the severity of PSO in clinical studies (Feldman, 2004). The PASI quantifies the severity and extent of the disease and weighs these with the percentage of BSA involvement.

The percent area of involvement (BSA%) is estimated across 4 body areas; head, upper limbs, trunk, and lower limbs and then transferred into a grade (Table 10–2).

The Investigator assesses the average redness, thickness, and scaliness of lesions in each body area (each on a 5-point scale); 0=none, 1=slight, 2=moderate, 3=marked, and 4=very marked.

The PASI score ranges from 0 to 72 with a higher score indicating increased disease severity.

Table 10-2: Body areas for calculation of percent BSA for PASI

| Body area | Details of area | BSACation | Degree of involvement of body area <sup>a</sup> |
|---|---|---|---|
| Head | Face, back of head | 10% | 0 to 6 |
| Upper limbs | Left, right, upper lower, flexor surface, extensor surface | 20% | 0 to 6 |
| Trunk | Front, back, groin | 30% | 0 to 6 |
| Lower limbs Left, right, upper lower, flexor surface, extensor surface, including buttocks | | 40% | 0 to 6 |
| Total | M | 100% | |

BSA=body surface area; PASI=Psoriasis Area and Severity Index

The PASI75, PASI90, and PASI100 responses are based on at least 75%, 90%, and 100% improvement in the PASI score compared to Baseline in PA0008. Thereafter PASI will be analyzed for the purposes of determining response only in subjects with PSO involving at least 3% of BSA at Baseline of PA0008.

### 10.11 MDA

Minimal Disease Activity is a state of disease activity deemed a useful derived target of treatment by both the patient and physician, given current treatment possibilities and limitations. Criteria shown in Table 10–3 covering all of the domains of the disease have been developed to determine whether or not a patient has reached MDA based on key outcome measures in PsA.

 $<sup>^{\</sup>rm a}$  Where 0=none; 1=1% to <10% affected, 2=10% to <30% affected, 3=30% to <50% affected, 4=50% to <70% affected, 5=70% to <90% affected, 6=90% to 100% affected

A subject is considered as having MDA if 5 or more of the following 7 criteria in Table 10–3 are fulfilled:

### Table 10–3: MDA criteria in PsA

| A subject is classified as in MDA when they meet 5 of 7 of the following criteria: | |
|---|---|
| • Tender joint count ≤1 | Patient global activity VAS ≤20 |
| • Swollen joint count ≤1 | HAQ ≤0.5 Valida |
| • PASI ≤1 or BSA ≤3 | Tender enthesial points ≤1 |
| • Patient pain VAS ≤15 | sions |

BSA=body surface area; HAO=Health Assessment Questionnaire; MDA=minimal disease activity; PASI=Psoriasis Area and Severity Index; VAS=visual analog scale

Data sources: Mease, 2011; Coates et al, 2010

In addition, a modified MDA will be determined using the criteria in Table 10-3 by fulfilling the criterion PASI ≤1 or BSA ≤3 and 4 out of the 6 remaining criteria.

### 10.12 DAS28(CRP)

The components for DAS28(CRP) include the TJC and SJC based on 28 joints (Section 10.2), CRP (Section 10.7) and the PGADA (Section 10.3). DAS28(CRP) is calculated as follows:

$$DAS28(CRP) = 0.56 \cdot \sqrt{TJC} + 0.28 \cdot \sqrt{SJC} + 0.01A \cdot PGADA + 0.36 \cdot \ln(CRP + 1) + 0.96$$
13 MASES

### 10.13

The MASES is an index that measures the severity (ie, intensity and extent) of enthesitis through the assessment of 13 entheses (bilateral costochondral 1, costochondral 7, anterior superior iliac spine, posterior iliac spine, iliac crest and proximal insertion of the Achilles tendon sites, and the fifth lumbar vertebral body spinous process) (Heuft-Dorenbosch et al, 2003) each scored as 0 or 1 and then summed for a possible score of 0 to 13.

#### 10.14 LDI

Dactylitis, the swelling of an entire digit related to articular and peri-articular inflammation, is a characteristic of inflammatory spondyloarthropathies, including PsA. Presence of dactylitis will be assessed using the LDI basic which evaluates for a ≥10% difference in the circumference of the digit compared to the opposite digit (Healy and Helliwell, 2007; Helliwell et al, 2005). This is then multiplied by the tenderness score, using a simple grading system (0=absent, 1=present). The digits involved and the matching contralateral digit will also be recorded at the same visits.

### 10:15 **Hospital Anxiety and Depression Scale**

The HADS was chosen for its well-established psychometric properties and its use in clinical research on biological therapy in subjects with chronic plaque PSO (Langley et al, 2010; Dauden et al, 2009). The HADS scores for anxiety and for depression range from 0 to 21 with higher scores indicating worse state. A score below 8 is considered to be normal whereas a score of 15 and above is considered severe (Snaith and Zigmond, 1994).

#### 10.16 PsAID-9

The PsAID-9 is a patient-reported outcome measure for assessing the impact of PsA in 9 physical and psychological domains, including pain, fatigue, skin problems, work and/or leisure activities, functional capacity, discomfort, sleep disturbance, coping, and anxiety/fear/uncertainty. Each domain is assessed with a single question using a 0 to 10 numerical rating scale. Each domain score is multiplied by a weighting factor and the results are then summed to provide the total score. The total score ranges from 0 to 10, with higher scores indicating a worse status. The PsAID-9 demonstrated satisfactory psychometric properties in an international validation study; however, further validation is needed (Gossec et al, 2014). A score below 4 out of 10 is considered a patient-acceptable status. A change of 3 or more points is considered relevant absolute change.

#### 10.17 **SF-36**

The SF-36 (Version 2, standard recall) is a 36-item generic Health-Related Quality of Life (HRQoL) instrument that uses a recall period of 4 weeks. Items are grouped into 8 domains as follows: Physical Functioning (10 items), Role Physical (4 items), Bodily Pain (2 items), General Health (5 items), Vitality (4 items), Social Functioning (2 items), Role Emotional (3 items), Mental Health (5 items), and 1 item for perceived stability or change in health (Health Transition) during the last year. The concepts represented by these domains contribute to physical, mental, and social aspects of HRQoL.

In addition to domain scores, the Physical Component Summary and Mental Component Summary scores are calculated from the 8 domains (excluding the Health Transition item). Component scores appreciate the impact of each domain on physical and mental health status (Maruish, 2011). Each of the 8 domain scores and the component summary scores range from 0 to 100, with a higher score indicating a better health status. The 2 component summary scores are standardized with a mean of 50 and a standard deviation of 10 in the general US population.

### ASSESSMENT OF IMMUNOGENICITY 11

The Investigator or designee will obtain blood samples for measurement of bimekizumab plasma concentrations and antibodies to bimekizumab at the time points specified in Table 5–1. When these samples are required at a visit during which the subject is dosed with IMP, the blood samples will be drawn prior to dosing. Samples should be drawn at the same time of the sampling for clinical laboratory tests. The time and date of collection will be recorded in the eCRF. Instructions pertaining to sample collection, processing, storage, labeling, and shipping are provided in the laboratory manual for this study. Any characterization of the anti-bimekizumab antibody response will be done using validated assays. Detailed information on sample analysis will be provided in a bioanalytical report.

### 12 STUDY MANAGEMENT AND ADMINISTRATION

# Adherence to protocol

This document The investigator should not deviate from the protocol. However, the investigator should take any measure necessary in deviation from or not defined by the protocol in order to protect clinical study subjects from any immediate hazard to their health and safety. In this case, this action

11 Dec 2019 PA0009

should be taken immediately, without prior notification of the regulatory authority, IRB/IEC, or sponsor.

After implementation of such measure, the investigator must notify the Clinical Project Manager

UCB (or designee) will monitor the study to meet the sponsor's monitoring Standard Operating Procedures (SOPs), ICH-GCP guideline, and applicable regulatory requirements, and to ensure that study initiation, conduct, and closure are adequate. Monitoring Standard Operating that study initiation, conduct, and closure are adequate.

The investigator and his/her staff are expected to cooperate with UCB (or designee) and to be available during the monitoring visits to answer questions sufficiently and to provide any missing information. The investigator(s)/institution(s) will permit direct access to source data/documents for study-related monitoring, audits, IRB/IEC review, and regulatory inspection(s).

The investigator will allow UCB (or designee) to periodically review all eCRFs and corresponding source documents (eg, hospital and laboratory records for each study participant). Monitoring visits will provide UCB (or designee) with the opportunity to evaluate the progress of the study, verify the accuracy and completeness of eCRFs, ensure that all protocol requirements, applicable authorities' regulations, and investigator's obligations are being fulfilled, and resolve any inconsistencies in the study records.

### Definition of source data 12.2.1

All source documents must be accurate, clear, unambiguous, permanent, and capable of being audited. They should be made using some permanent form of recording (ink, typing, printing, optical disc). They should not be obscured by correction fluid or have temporary attachments (such as removable self-stick notes). Photocopies and/or printouts of eCRFs are not considered acceptable source documents.

Source documents are original records in which raw data are first recorded. These may include hospital/clinic/general practitioner records, charts, diaries, x-rays, laboratory results, printouts, pharmacy records, care records, ECG or other printouts, completed scales, or quality of life questionnaires, for example. Source documents should be kept in a secure, limited access area.

Sponsor or designee will review to ensure that computerized source documents produced by the site are compliant with Food and Drug Administration (FDA) Part 11 requirements and document appropriately. Source documents that are computer generated and stored electronically must be printed for review by the monitor (eg, ECG reports). Once printed, these copies should be signed and dated by the Investigator and become a permanent part of the subject's source documents. The Investigator will facilitate the process for enabling the monitor to compare the content of the printout and the data stored in the computer to ensure all data are consistent.

Electronic data records must be saved and stored as instructed by UCB (or designee).

#### 12.2.2 Source data verification

Source data verification ensures accuracy and credibility of the data obtained. During monitoring visits, reported data are reviewed with regard to being accurate, complete, and verifiable from

source documents (eg, subject files, recordings from automated instruments, tracings [ECG], x-ray films, laboratory notes). All data reported on the eCRF should be supported by source documents, unless otherwise specified in Section 12.2.1.

### 12.3 Data handling

### 12.3.1 Case Report form completion

This study will use electronic data capture (EDC); the Investigator is responsible for prompt reporting of accurate, complete, and legible data in the eCRF and in all required reports.

This study will also use an electronic device (Site Tablet) to capture patient reported outcomes.

Serious AE reporting will be done using the SAE Report Form (see Section 9.2.2) while also entering the event in the appropriate eCRF section. The safety database and the clinical database will be reconciled during the study and discrepancies will be corrected as needed.

The Investigator should maintain a list of personnel authorized to enter data into the eCRF. Access to the EDC will be given after training has been received. A training certificate will be provided and filed.

Detailed instructions on the use of the EDC will be provided in the eCRF Completion Guidelines.

Corrections made after the Investigator's review and approval (by means of a password/electronic signature) will be re-approved by the Investigator. Any change or correction to the eCRF after saving must be accompanied by a reason for the change.

### 12.3.2 Database entry and reconciliation

Case Report forms/external electronic data will be entered/loaded into a validated electronic database using a clinical data management system (CDMS). Computerized data cleaning checks will be used in addition to manual review to check for discrepancies and to ensure consistency of the data. This study is performed using EDC: the data are entered into the eCRFs once and are subsequently verified.

An electronic audit trail system will be maintained within the CDMS to track all data changes in the database once the data have been saved initially into the system or electronically loaded. Regular backups of the electronic data will be performed.

# 12.3.3 Subject Screening and Enrollment log/Subject Identification Code list

The subject's screening and enrollment will be recorded in the Subject Screening and Enrollment Log.

The investigator will keep a Subject Identification Code list. This list remains with the investigator and is used for unambiguous identification of each subject.

The subject's consent and enrollment in the study must be recorded in the subject's medical record. These data should identify the study and document the dates of the subject's participation.

### 12.4 Termination of the study

UCB reserves the right to temporarily suspend or prematurely discontinue this study either at a single site, multiple sites, or at all sites at any time for reasons including, but not limited to,

If the study is prematurely terminated or suspended, UCB (or its representative) will inform the investigators/institutions and the regulatory authority(ies) of the termination or suspension and the reason(s) for the termination or suspension, in accordance will requirement(s). The IRP/IEC 1 termination or suspension by the sponsor or by the investigator/institution, as specified by the applicable regulatory requirement(s). In addition, arrangements will be made for the return of all unused IMP and other material in accordance with UCB procedures for the study?

### 12.5 **Archiving and data retention**

The investigator will maintain adequate records for the study, including eCRFs, medical records, laboratory results, Informed Consent documents, drug dispensing and disposition records, safety reports, information regarding participants who discontinued, and other pertinent data.

All essential documents are to be retained by the investigator until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region, or at least 2 years have elapsed since the formal discontinuation of clinical development of the IMP. These documents should be retained for a longer period, however, if required by the applicable regulatory requirement(s) or by an agreement with UCB (CPMP/ICH/135/95, 2002 [Section 4.9.5]). The investigator will contact UCB for authorization prior to the destruction of any study records or in the event of accidental loss or destruction of any study records. The investigator will also notify UCB should he/she relocate or move the study-related files to a location other than that specified in the sponsor's trial master file.

### 12.6 Audit and inspection

The investigator will permit study-related audits mandated by UCB, after reasonable notice, and inspections by domestic or foreign regulatory authorities.

The main purposes of an audit or inspection are to confirm that the rights and well-being of the subjects enrolled have been protected, that enrolled subjects (ie, signing consent and undergoing study procedures) are appropriate for the study, and that all data relevant for the evaluation of the IMP have been processed and reported in compliance with the planned arrangements, the protocol, investigational site, and IRB/IEC SOPs, ICH GCP, and applicable regulatory requirements.

The investigator will provide direct access to all study documents, source records, and source data. If an inspection by a regulatory authority is announced, the investigator will immediately inform UCB (or designee).

Noncompliance with the protocol, ICH-GCP, or local regulatory requirements by the STATISTICS

A description of statistical methods follows and will be described in more detail in the Statistical Analysis Plan.

13.1 Definition of analysis sets

The Enrolled Set (ES) will compare the statistical analysis sets investigator, institution, institution staff, or designees of the sponsor will lead to prompt action

The Safety Set (SS) will consist of all subjects who receive at least 1 dose of the IMP in PA0009.

The Full Analysis Set (FAS) will consist of all enrolled subjects who receive at least 1 dose of the IMP and have a valid measurement for at least 1 efficacy variable after PA0009 entry visit.

#### 13.2 General statistical considerations

Summary statistics will consist of frequency tables for categorical variables. For continuous variables, summary statistics will consist of number of available observations, arithmetic mean, standard deviation, median, minimum, and maximum unless stated otherwise.

In general, summary statistics will be done by randomized treatment group and by treatment group at completion of PA0008 (ie, bimekizumab 160mg Q4W or bimekizumab 320mg Q4W).

Two subpopulations will be defined for this study. Subpopulation 1 will consist of all subjects who do not receive rescue therapy according to the criteria outlined in Section 5.1.1. Subpopulation 2 will consist of all subjects who receive rescue therapy according to the criteria outlined in Section 5.1.1. Analyses of the primary and secondary variables will also be done on both subpopulations.

Changes from Baseline will be calculated relative to the Baseline of PA0008. Variables measured at the start of PA0009 will be referred to as PA0009 entry values.

### Planned safety analyses 13.3

### Safety analyses 13.3.1

Safety variables will be analyzed for all subjects in the SS.

Adverse events will be coded according to the Medical Dictionary for Regulatory Activities.

Adverse events will be summarized descriptively by treatment group at completion of PA0008, primary system organ class, high level term, and preferred term. This summary will include raw incidence rates, exposure-adjusted incidence rates (EAIRs) with associated 95% CIs, and exposure-adjusted event rates (EAERs) where the EAIR and EAER are expressed per 100 patient-years of exposure.

Patient exposure at risk will be defined as date of last administration of study medication – date of first administration of bimekizumab +20 weeks. If a subject has an adverse event with fatal outcome, patient exposure at risk is censored at the date of death.

The extent of exposure to study medication in PA0009 will be summarized using descriptive statistics by treatment group at completion of PA0008.

Dasenne values in clinical laboratory variables (hematology and biochemistry, excepting high-sensitivity CRP) will be summarized descriptively by visit and by treatment group at completion of PA0008.

Due to a change in laboratory vendor between PA0008 and PA0009, laboratory values (excepting CRP) will use the PA0009 Laboratory Baseline, defined as the earliest post value recorded in PA0009. Change from PA0008 to the control of PA0009 to the Change from PA0008 Baseline values in vital signs variables will be summarized descriptively

these parameters. (The CRP values from the 2 analyzing laboratories have been calibrated, so change from PA0008 Baseline will be calculated for that parameter.)

All safety analyses will be conducted for both subpopulations.

### 13.4 Planned efficacy analyses

Secondary and other efficacy variables will be summarized for all subjects in the FAS; efficacy analyses will be performed over 104 weeks (2 years).

Responder variables (eg. ACR20 response) will be derived relative to the Baseline of PA0008 and summarized descriptively. Percentages will be summarized descriptively by visit, by randomized treatment group, and by treatment group at PA0009 entry.

Change from Baseline of PA0008 of all continuous variables will be summarized descriptively by visit, by randomized treatment group, and by treatment group at completion of PA0008.

### Subgroup analysis 13.4.1

Subgroup analyses will be performed on the efficacy variables. The following variables for subgroup analyses will be defined:

- Region
- Disease duration
- Previous tumor necrosis factor (TNF) inhibitor agent exposure
- Concomitant DMARD status at Baseline of PA0008

### Planned immunogenicity analyses 13.5

Immunogenicity variables will be analyzed for all subjects in the SS.

Bimekizumab plasma concentration and anti-bimekizumab antibody appearance will be summarized by visit, by randomized treatment group, and by treatment group at completion of PA0008. The first occurrence of anti-bimekizumab antibody positivity as well as persistent and transient anti-bimekizumab antibody positivity will be summarized by visit, by randomized treatment group, and by treatment group at completion of PA0008. Figures on persistent and transient anti-bimekizumab antibody positivity over time and on the relationship between ACR20 response and anti-bimekizumab antibody positivity over time will be produced.

### 13.6 Other analyses

Other variables will be summarized using descriptive statistics using the treatment group at completion of PA0008.

### 13.7 Handling of protocol deviations

Important protocol deviations are deviations from the protocol which potentially could have a meaningful impact on study conduct, or on the safety or efficacy outcomes for an individual subject. The criteria for identifying important protocol deviations will be defined within the appropriate protocol-specific document. Important protocol deviations will be reviewed as part of the ongoing data cleaning process.

# 13.8 Handling of dropouts or missing data

Missing binary efficacy variables will be imputed using nonresponder imputation (NRI). In NRI, each subject with missing data or who has prematurely finished the study will be counted as a nonresponder.

For missing continuous efficacy variables, a multiple imputation (MI) approach will be used. In MI, the missing value is replaced by a set of plausible values, where each value is a Bayesian draw from the conditional distribution of the missing data given the observed data. Non-monotone missing data (ie, intermittent missing data) will be imputed several times with the Markov Chain Monte Carlo (MCMC) method and monotone missing data will be imputed using a monotone regression model. Each set of imputed data will then be summarized and the summaries will be combined into a single inference (Carpenter and Kenward, 2013).

Safety data will not be imputed.

As a sensitivity analysis, the ACR, PASI, LDI, MASES, and MDA efficacy variables will be analyzed based on observed data in addition to a sensitivity analysis based on multiple imputation of ACR component scores and PASI scores for the ACR and PASI response variables, respectively. Subjects with missing data or who have prematurely finished the study will be treated as missing.

# 13.9 Planned interim analysis and data monitoring

No formal interim analysis is planned for this study. Additional data cuts may be prepared following regulatory requests or for publication purposes.

# 13.10 Determination of sample size

There is no formal sample size for this study. The sample size is determined by the number of subjects eligible for PA0009 and rolling over from PA0008. Up to 200 subjects from PA0008 could be enrolled into this study.

# 14 ETHICS AND REGULATORY REQUIREMENTS

### 14.1 Informed consent

Subject's informed consent must be obtained and documented in accordance with local regulations, ICH-GCP requirements, and the ethical principles that have their origin in the principles of the Declaration of Helsinki.


**UCB** 11 Dec 2019 Bimekizumab PA0009

Prior to obtaining informed consent, information should be given in a language and at a level of complexity understandable to the subject in both oral and written form by the investigator (or designee). Each subject will have the opportunity to discuss the study and its alternatives with the investigator.

Prior to participation in the study, the Informed Consent form should be signed and personally dated by the subject and by the person who conducted the informed consent discussion (investigator or designee). The subject must receive a copy of the signed and dated Informed Consent form. As part of the consent process, each subject must consent to direct access to his/her medical records for study-related monitoring, auditing, IRB/IEC review, and regulatory inspection.

If the Informed Consent form is amended during the study, the investigator (or the sponsor, if applicable) must follow all applicable regulatory requirements pertaining to the approval of the amended Informed Consent form by the IRB/IEC and use of the amended form.

All studies conducted at centers in the United States must include the use of a Health Insurance Portability and Accountability Act Authorization form.

The subject may withdraw his/her consent to participate in the study at any time. A subject is considered as enrolled in the study when he/she has signed the informed Consent form. An eCRF must not be started, nor may any study specific procedure be performed for a given subject, without having obtained his/her written consent to participate in the study.

### Subject identification cards 14.2

Upon signing the Informed Consent and Assent form (as applicable), the subject will be provided with a subject identification card in the language of the subject. The investigator will fill in the subject identifying information and medical emergency contact information. The investigator will instruct the subject to keep the card with him/her at all times.

### 14.3 Institutional Review Boards and Independent Ethics Committees <

The study will be conducted under the auspices of an IRB/IEC, as defined in local regulations, ICH-GCP, and in accordance with the ethical principles that have their origin in the Declaration of Helsinki.

The investigator/UCB will ensure that an appropriately constituted IRB/IEC that complies with the requirements of the current ICH-GCP version or applicable country-specific regulations will be responsible for the initial and continuing review and approval of the clinical study. Prior to initiation of the study, the investigator/UCB will forward copies of the protocol, Informed Consent form, Investigator's Brochure, investigator's curriculum vitae (if applicable), advertisement (if applicable), and all other subject-related documents to be used for the study to the IRB/IEC for its review and approval.

Before initiating a study, the investigator will have written and dated full approval from the responsible IRB/IEC for the protocol.

The investigator will also promptly report to the IRB/IEC all changes in the study, all unanticipated problems involving risks to human subjects or others, and any protocol deviations, to eliminate immediate hazards to subjects.

The investigator will not make any changes in the study or study conduct without IRB/IEC approval, except where necessary to eliminate apparent immediate hazards to the subjects. For minor changes to a previously approved protocol during the period covered by the original approval, it may be possible for the investigator to obtain an expedited review by the IRB/IEC as allowed.

As part of the IRB/IEC requirements for continuing review of approved studies, the investigator will be responsible for submitting periodic progress reports to the IRB/IEC (based on IRB/IEC) requirements), at intervals appropriate to the degree of subject risk involved, but no less than once per year. The investigator should provide a final report to the IRB/IEC following study completion.

UCB (or its representative) will communicate safety information to the appropriate regulatory authorities and all active investigators in accordance with applicable regulatory requirements. The appropriate IRB/IEC will also be informed by the investigator or the sponsor, as specified by the applicable regulatory requirements in each concerned country. Where applicable, investigators are to provide the sponsor (or its representative) with evidence of such IRB/IEC notification.

### 14.4 Subject privacy

UCB staff (or designee) will affirm and uphold the subject's confidentiality. Throughout this study, all data forwarded to UCB (or designee) will be identified only by the subject number assigned at Screening.

The investigator agrees that representatives of UCB, its designee, representatives of the relevant IRB/IEC, or representatives of regulatory authorities will be allowed to review that portion of the subject's primary medical records that directly concerns this study (including, but not limited to, laboratory test result reports, ECG reports, admission/discharge summaries for hospital admissions occurring during a subject's study participation, and autopsy reports for deaths occurring during the study).

#### 14.5 Protocol amendments

Protocol changes may affect the legal and ethical status of the study and may also affect the statistical evaluations of sample size and the likelihood of the study fulfilling its primary objective.

Significant changes to the protocol will only be made as an amendment to the protocol and must be approved by UCB, the IRB/IEC, and the regulatory authorities (if required), prior to being implemented.

# FINANCE, INSURANCE, AND PUBLICATION

Insurance coverage will be handled according to local requirements.

Finance, insurance, and publication rights are addressed in the investigator and/or CRO agreements, as applicable.

#### REFERENCES 16

Antoni CE, Kavanaugh A, Kirkham B, Tutuncu Z, Burmester GR, Schneider U, et al. Sustained Antoni C, Krueger GG, de Vlam K, Birbara C, Beutler A, Guzzo C, et al. Infliximab improves signs and symptoms of psoriatic arthritis: results of the IMPACT 2 trial. Ann Rheum Dis. 2005b;64:1150–57.

Baeten D, Sieper J, Braun J, Baraliakos X, Dougados M, Emery P et al. San Linding interleukin-17a inhibitor, in ankyloging and inhibitor, in ankyloging and inh benefits of infliximab therapy for dermatologic and articular manifestations of psoriatic arthritis:

Carpenter JR, Kenward MG. Multiple imputation and its application. West Sussex, United Kingdom: John Wiley & Sons; 2013.

Coates LC, Fransen J, Helliwell PS. Defining minimal disease activity in psoriatic arthritis: a proposed objective target for treatment. Ann Rheum Dis 2010;69:48–53.

CPMP/ICH/135/95. Note for guidance on good clinical practice. July 2002.

Dauden E, Griffiths CE, Ortonne JP, Kragballe K, Molta CT, Robertson D, et al. Improvements in patient-reported outcomes in moderate-to-severe psoriasis patients receiving continuous or paused etanercept treatment over 54 weeks: the CRYSTEL study. J Eur Acad Dermatol Venereol. 2009;23(12):1374-82.

Feldman SR. A quantitative definition of severe psoriasis for use in clinical trials. J Dermatolog Treat. 2004;15(1):27-9.

Felson DT, Anderson JJ, Boers M, Bombardier C, Chernoff M, Fried B, et al. The American College of Rheumatology preliminary core set of disease activity measures for rheumatoid arthritis clinical trials. The Committee on Outcome Measures in Rheumatoid Arthritis Clinical Trials. Arthritis Rheum. 1993;36(6):729-40.

Fujishima S, Watanabe H, Kawaguchi M, Suzuki T, Matsukura S, Homma T, et al. Involvement of IL-17F via the induction of IL-6 in psoriasis. Arch Derm Res. 2010;302:499-505.

Genovese MC, Mease PJ, Thomson GT, Kivitz AJ, Perdok RJ, Weinberg MA, et al. Safety and efficacy of adalimumab in treatment of subjects with psoriatic arthritis who had failed disease modifying antirheumatic drug therapy. J Rheumatol. 2007;34:1040–50.

Genovese MC, Van den Bosch F, Roberson SA, Bojin S, Biagini IM, Ryan P, et al. LY2439821, a humanized anti-interleukin-17 monoclonal antibody, in the treatment of patients with rheumatoid arthritis: a phase I randomized, double blind, placebo-controlled, proof-of-concept study. Arthritis Rheum. 2010;62:929-39.

Gladman DD, Mease PJ, Cifaldi MA, Perdok RJ, Sasso E, Medich J. Adalimumab improves joint-related and skin-related functional impairment in patients with psoriatic arthritis: patient-reported outcomes of the Adalimumab Effectiveness in Psoriatic Arthritis Trial. Ann Rheum Dis. 2007;66:163-68.

Gossec L, de Wit M, Klitz U, Braun J, Kalyoncu U, Scrivo R, et al. A patient-derived and patient-reported outcome measure for assessing psoriatic arthritis: elaboration and preliminary

validation of the Psoriatic Arthritis Impact of Disease (PsAID) questionnaire, a 13-country EULAR initiative. Ann Rheum Dis. 2014;73:1012-19.

Gottlieb A, Menter A, Mendelsohn A, Shen YK, Li S, Guzzo C, et al. Ustekinumab, a human

Transper EG, Guo C, Rizzo H, Lillis JV, Kurtz SE, Skorcheva I, et al. Th17 cytokines stimulate CCL20 expression in keratinocytes in vitro and in vivo: implications for psoriasis pathogenesis J Invest Dermatol. 2009;129:2175-83.

Healy PJ, Helliwell PS. Measuring dactylitis in clinical to the control of th

Helliwell PS, Firth J, Ibrahim GH, Melsom RD, Shah I, Turner DE. Development of an assessment tool for dactylitis in patients with psoriatic arthritis. J Rheumatol. 2005;32:1745-50.

Heuft-Dorenbosch L, Spoorenberg A, van Tubergen A, Landewé R, van der Tempel H, Mielants H, et al. Assessment of enthesitis in ankylosing spondylitis. Ann Rheum Dis. 2003;62:127-32.

Hueber W, Patel DD, Dryja T, Wright AM, Koroleva I, Bruin G, et al. Effects of AIN457, a fully human antibody to interleukin-17A on psoriasis, rheumatoid arthritis, and uveitis. Sci Transl Med. 2010;2:52ra72.

Ivanov II, Frutos Rde L, Manel N, Yoshinaga K, Rifkin DB, Sartor RB, et al. Specific microbiota direct the differentiation of IL-17-producing T-helper cells in the mucosa of the small intestine. Cell Host Microbe. 2008;4:337-49.

Johansen C, Usher PA, Kjellerup RB, Lundsgaard D, Iversen L, Kragballe K. Characterization of the interleukin-17 isoforms and receptors in lesional psoriatic skin. Br J Dermatol. 2009;160:319-24.

Kavanaugh A, Antoni C, Krueger GG, Yan S, Bala M, Dooley LT, et al. Infliximab improves health related quality of life and physical function in subjects with psoriatic arthritis. Ann Rheum Dis. 2006;65:471–77.

Kavanaugh A, McInnes J, Mease P, Krueger GG, Gladman D, Gomez-Reino J, et al. Golimumab, a new human tumor necrosis factor  $\alpha$  antibody, administered every four weeks as a subcutaneous injection in psoriatic arthritis: twenty-four-week efficacy and safety results of a randomized, placebo-controlled study. Arthritis Rheum. 2009;60:976-86.

Kavanaugh A, van der Heijde D, McInnes IB, Mease P, Krueger GG, Gladman DD, et al. Golimumab in psoriatic arthritis: one-year clinical efficacy, radiographic, and safety results from a phase III, randomized, placebo-controlled trial. Arthritis Rheum. 2012;64:2504-17.

Langley RG, Feldman SR, Han C, Schenkel B, Szapary P, Hsu MC, et al. Ustekinumab significantly improves symptoms of anxiety, depression, and skin-related quality of life in patients with moderate-to-severe psoriasis: Results from a randomized, doubleblind, placebo-controlled phase III trial. J Am Acad Dermatol. 2010;63(3):457-65.
11 Dec 2019 PA0009

Leonardi C, Matheson R, Zachariae C, Cameron G, Li L, Edson-Heredia E, et al. Anti-interleukin-17 monoclonal antibody ixekizumab in chronic plaque psoriasis. N Engl J Med. 2012;366:1190-9.

Maruish ME, editor. User's manual for the SF-36v2 Health Survey. 3rd ed. Lincoln, RI: QualityMetric Incorporated; 2011.

McHugh NJ, Balachrishnan C, Jones SM. Progression of peripheral joint disease in psoriatic arthritis: a 5-year prospective study. Rheumatology. 2003;42:778–83.

McInnes IB, Mease PJ, Kirkham B, Kavanaugh A, Ritchlin CT, Rahman P, et al. Secukinumab, a human anti-interleukin-17A monoclonal antibody, in patients with psoriatic arthritis (FUTURE 2): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2015;386:1137-46.

McInnes IB, Sieper J, Braun J, Emery P, van der Heijde D, Isaacs JD, et al. Efficacy and safety of secukinumab, a fully human anti-interleukin-IL17A monoclonal antibody, in patients with moderate-to-severe psoriatic arthritis: a 24-week, randomised, double-blind, placebo-controlled, phase II proof-of-concept trial. Ann Rheum Dis. 2014;73:349-56.

Mease PJ. Measures of psoriatic arthritis. Arthritis Care & Research 2011;63(S11):S64-85.

Mease PJ, Gladman DD, Ritchlin CT, Ruderman EM, Steinfeld SD, Choy EH, et al. Adalimumab for the treatment of subjects with moderately to severely active psoriatic arthritis: results of a double-blind, randomized, placebo-controlled trial. Arthritis Rheum. 2005;52:3279-89.

Mease PJ, Kivitz AJ, Burch FX, Siegel EL, Cohen SB, Ory P, et al. Etanercept treatment of psoriatic arthritis: safety, efficacy, and effect on disease progression. Arthritis Rheum. 2004;50:2264–72.

Mease PJ, McInnes IB, Kirkham B, Kavanaugh, A, Rahman, P, van der Heijde D, et al. Secukinumab inhibition of Interleukin-17A in patients with psoriatic arthritis. N Engl J Med. 2015;373:1329-39.

Mundt JC, Greist JH, Gelenberg AJ, Katzelnick DJ, Jefferson JW, Modell JG. Feasibility and Validation of a Computer-Automated Columbia-Suicide Severity Rating Scale Using Interactive Voice Response Technology. J Psychiatr Res. 2010;44(16):1224-8.

Ogdie A, Weiss P. The epidemiology of psoriatic arthritis. Rheum Dis Clin North Am. 2015;41(4):545-68.

Osterhaus J, Purcaru O, Richard L. Discriminant validity, responsiveness and reliability of the rheumatoid arthritis specific Work Productivity Survey (WPS-RA). Arthritis Res Ther. 2009;11(3):R:73.

Papp KA, Leonardi C, Menter A, Ortonne JP, Krueger JG, Kricorian G, et al. Brodalumab, an anti–interleukin-17–receptor antibody for psoriasis. N Engl J Med. 2012;366:1181-9.

Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, et al. The Columbia-Suicide Severity Rating Scale: Initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011;168(12):1266-77.

11 Dec 2019 PA0009

Raychaudhuri SP, Raychaudhuri SK, Genovese MC. IL-17 receptor and its functional significance in psoriatic arthritis. Mol Cell Biochem. 2012;359:419–29.

Watanabe H, Kawaguchi M, Fujishima S, Ogura M, Matsukura S, Takeuchi H, et al. Functional characterization of IL-17F as a selective neutrophil attractant in psoriasis. J Invest Dermatol 2009;129:650-6.

Woodworth T, Furst DE, Alten R Rimal assessment and

et al. Stand. cal trials II: the 14.

Let al. Stand. cal trials II: the 14.

Let al. Stand. cal assessment and reporting of adverse effects in rheumatology clinical trials II: the Rheumatology


### 17 APPENDICES

# 17.1 Markedly abnormal laboratory values

Table 17-1: Definitions of markedly abnormal hematology values

| | Markedly Abno | ormal Definition |
|---|---|---|
| Parameter (RCTC units) | Low | High |
| Hemoglobin (g/dL) | <lln< td=""><td>N/A</td></lln<> | N/A |
| | AND | |
| | >2.0 decrease from Baseline | ions |
| Hemoglobin (g/dL) | <8.0 | NA |
| Leukocytes (total x 1000) | <2.0 | © N/A |
| Lymphocytes (x 1000) | <0.5 | N/A |
| Neutrophils (x 1000) | <1.0a | N/A |
| Platelets (x 1000) | <50 | N/A |

LLN=lower limit of normal; N/A = Not Applicable; RCTC= Rheumatology Common Toxicity Criteria Data source: modified from Appendix Rheumatology Common Toxicity Criteria v.2.0 presented in Woodworth et al, 2007

Table 17-2: Definitions of markedly abnormal biochemistry values

| | Markedly Abn | ormal Definition |
|------------------------|--------------|------------------|
| Parameter (RCTC units) | Low | High |
| Alkaline Phosphatase | N/A | >3 x ULN |
| ALT | N/A | >3 x ULN |
| AST | N/A | >3 x ULN |
| Calcium (mg/dL) | <7.0 | >12.5 |
| Creatinine (mg/dl) | N/A | >1.8 x ULN |
| Glucose (mg/dL) | <40 | >250 |
| Potassium (mmol/L) | <3.0 | >6.4 |
| Sodium (mmol/L) | <125 | N/A |
| Total bilirubin | N/A | ≥2 x ULN |
| Uric acid | N/A | ≥3 x ULN |

ALT=alanine aminotransferase; AST=aspartate aminotransferase; N/A=Not applicable; RCTC= Rheumatology Common Toxicity Criteria; ULN=upper limit of normal

Data source: modified from Appendix Rheumatology Common Toxicity Criteria v.2.0 presented in Woodworth et al, 2007


<sup>&</sup>lt;sup>a</sup> Withdrawal criteria for neutrophils is <0.5 (Section 6.3)

11 Dec 2019 PA0009

### **Protocol Amendment 1** 17.2

### Rationale for the amendment

Ascline of accinations.

Ascline of accinations.

Ascline of accinations.

Ascline of accinations.

Ascline of accinations.

Ascline of accinations.

Ascline of Accinations.

Ascline of Accinatio

PA0009 entry value in the Maastricht Ankylosing Spondylitis Enthesitis Index (MASES) at Week 48, change from Baseline and PA0009 entry value in the Leeds Dactylitis Index (LDI) at


11 Dec 2019 PA0009

Week 48, the Psoriasis Area and Severity Index 75 (PASI75) response, and the Psoriasis Area and Severity Index 90 (PASI90) response at Week 48.

## Change #3

Section 7.8.1 item 3

### Has been changed to:

Up to 1 injection per joint for up to 3 discrete joints is permitted per 12-month period. Injected joints are censored for the joint examination.

as been changed to:

Up to 1 injection per joint for up to 3 discrete joints is permitted per 12-month period. Investigators should follow the guidance in the CRF instruction.

## Change #4

Prohibited concomitant treatments (medications and therapies), Vaccines, Section 7.8.2 paragraph 1

Administration of live, attenuated vaccines is not allowed during the conduct of the study or for 20 weeks after the last dose of study drug. Administration of non-live, attenuated vaccines is allowed during the study at the discretion of the Investigator.

## Has been changed to:

Administration of live, attenuated vaccines is not allowed during the conduct of the study or for 20 weeks after the last dose of study drug. Administration of non-live, **inactivated** vaccines is allowed during the study at the discretion of the Investigator.

## Change #5

Safety signal detection, paragraph 3 Section 9.1.11

In addition, an independent Data Monitoring Committee (DMC) will periodically review and monitor the safety data from this study and advise UCB. Details are provided in the DMC Charter. Cardiovascular and Neuropsychiatric Adjudication Committees will also periodically review and monitor the safety data from this study and advise UCB. Details are provided in the Adjudication Committee Charters.

## Has been changed to:

In addition, Cardiovascular and Neuropsychiatric Adjudication Committees will also periodically review and monitor the safety data from this study and advise UCB. Details are provided in the Adjudication Committee Charters.

**UCB** 11 Dec 2019 PA0009

### Change #6

Section 10.8 ACR20, ACR50, and ACR70 response, paragraph 1

The ACR20, ACR50, and ACR70 response rates are based on a 20%, 50%, and 70% or greater improvement relative to Baseline of PA0008 and PA0009 entry values in the following measures:

### Change #7

Section 10.10 Psoriasis Area and Severity Index (PASI), paragraph 6

The PASI75, PASI90, and PASI100 responses are based on at least 75%, 90%, and 100% improvement in the PASI score compared to Baseline in PA0008. Thereafter PASI will be assessed for the purposes of determining response only in subjects with PSO involving at least 3% of BSA at study entry.

### Has been changed to:

The PASI75, PASI90, and PASI100 responses are based on at least 75%, 90%, and 100% improvement in the PASI score compared to Baseline in PA0008 and PA0009 entry values. Thereafter PASI will be assessed for the purposes of determining response only in subjects with PSO involving at least 3% of BSA at study entry.

## Change #8

**MDA** Section 10.11

The following text was added beneath Table 10-3:

In addition, a modified MDA will be determined using the criteria in Table 10-3 by fulfilling the criterion PASI  $\leq 1$  or BSA  $\leq 3$  and 4 out of the 6 remaining criteria.

### 17.3 **Protocol Amendment 2**

### Rationale for the amendment

The purpose of this substantial amendment is as follows:

- Amend the open-label treatment period for clarification, as per request from the regulatory agency.

  Amend the study procedures and assessments to be a fine Efficacy assessments were assessments were assessments were assessments.
- Amend the study procedures and assessments to be performed at the Safety Follow-up visit.
- Include additional wording to the inclusion criteria (criterion #5) listing acceptable methods of contraception for female subjects.
- Amend the exclusion criteria (criterion #2) to include further clarification on when to consult the medical monitor.
- To revise the withdrawal criteria section to provide instructions for the management of subjects with newly diagnosed IBD or with IBD flares during the study.
- To revise and clarify the SAE criteria for pregnancy for consistency.
- Amend the table for identification/exclusion of alternative etiology to include ALT and AST.
- Amend and remove wording from the criteria determined for handling of dropouts or missing data.

### **Modifications and changes**

## Global change

The following global change was made for the duration of the open-label treatment period and period for administration of bimekizumab:

104 weeks (2 weeks)

## Has been changed to

100104 weeks (~2 weeks)

## Specific changes

## Change #1

List of Abbreviations

The following abbreviations have been added:

**IBD Inflammatory Bowel Disease** 

**IUD** intrauterine device

**IUS** intrauterine hormone-releasing system


UCB 11 Dec 2019 Bimekizumab PA0009

**Markov Chain Monte Carlo MCMC** 

**Rheumatology Common Toxicity Criteria RCTC** 

## Change #2

## **Sponsor Study Physician**

| Name: | , MD | 3 |
|----------|---------------------------|------------|
| Address: | UCB BIOSCIENCES Inc. | |
| | 8010 Arco Corporate Drive | sio |
| | Raleigh, NC 27617 | extension. |
| | UNITED STATES | et |
| Phone: | (office) | Y SU., |
| | (mobile) | alle |

# Has been changed to:

| Name: | MD, MSc, PhD |
|----------|-------------------------------------------------|
| Address: | UCB Pharma Ltd. <del>UCB BIOSCIENCES Inc.</del> |
| | 208 Bath Road 8010 Arco Corporate Drive |
| | Slough, SL1 3WE Raleigh, NC 27617 |
| | UNITED KINGDOM UNITED STATES |
| Phone: | (office) |
| | (mobile) |

## Change #3

Change #3
Study contact information

# Clinical Trial Biostatistician

| Name: | Dr. , Senior Biostatistician |
|----------|------------------------------------------|
| Address: | UCB BIOSCIENCES GmbH Alfred-Nobel-Str.10 |
| | 40789 Monheim am Rhein<br>GERMANY |
| Phone: | |

### Has been changed to:

### **Clinical Trial Biostatistician**

| Name: | <del>Biostatistician</del> <del>, Senior</del> | |
|---|---|---|
| Address: | UCB BIOSCIENCES GmbH Alfred-Nobel-Str.10 0789 Monheim am Rhein GERMANY | SÓ |
| Phone: | | Office |

## Change #4

Section 5.1 Study design, paragraph 3

Additionally, as described in (Section 5.1.1), other treatments may be used in addition to bimekizumab per Investigator discretion. Subjects not responding to treatment may be withdrawn from the study at the discretion of the Investigator.

### Has been changed to:

Additionally, as described in (Section 5.1.1), other treatments may be used in addition to bimekizumab per Investigator discretion. Subjects not responding to treatment may be withdrawn from the **treatment and** study at the discretion of the Investigator.

## Change #5

Section 5.1.2 Study duration per subject

The study duration for each subject is estimated to be up to a maximum of 120 weeks:

- Open Label Treatment Period: up to 104 weeks (2 years)
- SFU Visit: 20 weeks after the final dose of bimekizumab

The subject may remain in the study until the study ends after 2 years (104 weeks of treatment), until the Sponsor decides to close the study, or until bimekizumab development is stopped by the Sponsor, whichever comes first. The Sponsor may consider transitioning the subject into another bimekizumab study or program.

The end of the study is defined as the date of the last visit of the last subject in the study.

## Has been changed to:

The study duration for each subject is estimated to be up to a maximum of 120 weeks:

• Open-Label Treatment Period: up to 104100 weeks (~2 years)

e study.

...e study.

...e stu


| JCB<br>Clinical Study Protocol | | | | | | | | | | Bim | nekiz | umab | | | | | | | | variation |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| hange #6 | | | | | | | | | | | | | | | | | | | | · atio |
| ection 5.2 Schedule of | study | y ass | essn | nent | ts, T | able | 5-1 | | | | | | | | | | | | O. | Asilio |
| Protocol activity | | | | | | | | T | reatr | nent l | Perio | d | | | | | | | 01501 | SFU |
| Weeksa | EVb | 4 | 12 | 16 | 24 | 28 | 36 | 40 | 48 | 52 | 60 | 64 | 72 | 76 | 84 | 88 | 96 | | W104/ | - |
| | | 8 | | 20 | | 32 | | 44 | | 56 | 1 | 68 | 1 | 80 | 1 | 92 | 1 , | tier | ET | 1 |
| Visita | 1 | 2/3 | 4 | Hc | 5 | Hc | 6 | Hc | 7 | Hc | 8 | Hc | 9 | Hc | 10 | Hc | $\mathcal{H}$ | 12 | 13 | |
| Informed consent | Xd | | | | | | | | | | | | | | | 6. | | | | |
| Inclusion/exclusion | Xe | | | | | | | | | | | | | | | SIL | | | | |
| Concomitant medications | Xf | X | X | | X | | X | | X | | X | | X | | 8 | | X | X | X | X |
| Adverse events | Xf | X | X | | X | | X | | X | | X | | X | 110 | X | | X | X | X | X |
| C-SSRS | $X^{e,f}$ | X | X | | X | | X | | X | | X | 2 | X | 66, | X | | X | X | X | X |
| HADS | Xe,f | | X | | X | | X | | X | | X( | ) .:( | SX. | | X | | X | X | X | X |
| HAQ-DI | X <sup>e,f</sup> | | X | | X | | X | | X | _< | X | 130 | X | | X | | X | X | X | X |
| SF-36 | X <sup>e,f</sup> | | X | | X | | X | | X | C) | XC | 1 | X | | X | | X | X | X | X |
| PGADA | Xe,f | | X | | X | | X | | X | n' | X | | X | | X | | X | X | X | X |
| PtAAP | X <sup>e,f</sup> | | X | | X | | X | 8 | X | 10 | X | | X | | X | | X | X | X | X |
| PsAID-9 | X <sup>e,f</sup> | | X | | X | | X | | ĹØŽ | | X | | X | | X | | X | X | X | X |
| ΓB questionnaire | X <sup>e,f</sup> | | X | | X | | X | 40 | X | | X | | X | | X | | X | X | X | X |
| Vital signs (pulse,<br>temperature, BP) <sup>g</sup> | Xe | X | X | | Х | × | O.A. | | X | | X | | X | | X | | X | X | X | X |
| Body weight | X <sup>e,f</sup> | | X | | X | 0 | X | | X | | X | | X | | X | | X | X | X | X |
| Physical examination <sup>h</sup> | X <sup>e,f</sup> | | | | 2716 | | | | X | | | | | | | | X | | X | X |
| JC (78) and SJC (76) | X <sup>e,f</sup> | | X, | ×O | X | | X | | X | | X | | X | | X | | X | X | X | X |
| BSA affected by PSO (BSA palm method) | X <sup>e,f</sup> | | J.S. | Ď | Х | | Х | | X | | Х | | X | | X | | X | X | X | X |
| PASIi | Xe,f | 100 | X | | X | | X | | X | | X | | X | | X | | X | X | X | X |
| MASES | Xer | | X | | X | | X | | X | | | | X | | | | X | | X | X |

11 Dec 2019

| Protocol activity | | | | | | | | T | reatr | nent l | Perio | d | | | | | | | | SEU |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Weeks <sup>a</sup> | EVb | 4 | 12 | 16 | 24 | 28 | 36 | 40 | 48 | 52 | 60 | 64 | 72 | 76 | 84 | 88 | 96 | 100 | W104/ | 101- |
| | | 8 | | 20 | | 32 | | 44 | | 56 | | 68 | | 80 | | 92 | | | ETO | |
| Visita | 1 | 2/3 | 4 | Hc | 5 | Hc | 6 | Hc | 7 | Hc | 8 | Hc | 9 | Hc | 10 | Hc | 11 | 12 | . 13 | |
| LDI | Xe,f | | X | | X | | X | | X | | X | | X | | X | | X | X | X | X |
| PhGADA | Xe,f | | X | | X | | X | | X | | X | | X | | X | | X | X | X | X |
| ECG | Xe,f | | | | | | | | X | | | | | | | | (X) | | X | |
| Hematology/biochemistry/<br>urine pregnancy <sup>j,k</sup> | Xe,f | | X | | Х | | Х | | X | | X | | Х | | Х | and | X | X | X | X |
| Blood Sample for CRPk | Xe,f | | X | | X | | X | | X | | X | | X | | .X | | X | X | X | X |
| Blood sample for<br>bimekizumab plasma<br>concentrations <sup>k</sup> | Xe,f | | X | | X | | X | | X | | | 04 | X | Oblica | | | Х | | X | X |
| Blood sample for anti-<br>bimekizumab antibodies <sup>k</sup> | Xe,f | | X | | X | | X | | X | | | | X | | | | X | | X | X |
| IGRA TB test <sup>1</sup> | Xe | | | | | | | | X | | ( ) | KIL. | | | | | X | | | X |
| IXRS | X | X | X | | X | | X | | Χſ | ٢, | 13 | | X | | X | | X | X | X | X |
| Bimekizumab<br>administration | X | X | X | X | X | X | X | X | X | Q <sub>X</sub> | X | X | X | X | X | X | X | X | | |


# Has been changed to:

| Protocol activity | | | | | | | | Tı | reatn | nent 1 | Perio | d | | | | | | | 1 | SF |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Weeksa | EVb | 4 | 12 | 16 | 24 | 28 | 36 | 40 | 48 | 52 | 60 | 64 | 72 | 76 | 84 | 88 | 96 | 100 | W104/ | |
| | | 8 | 1 | 20 | | 32 | | 44 | | 56 | | 68 | | 80 | | 92 | | _< | ET | |
| Visit <sup>a</sup> | 1 | 2/3 | 4 | Hc | 5 | Hc | 6 | Hc | 7 | Hc | 8 | Hc | 9 | Hc | 10 | Hc | 11 | 12 | 13 | |
| Informed consent | Xd | | | | | | | | | | | | | | | | 7 | 87 | | |
| Inclusion/exclusion | Xe | | | | | | | | | | | | | | | 20 | Z, | | | |
| Concomitant medications | Xf | X | X | | X | | X | | X | | X | | X | | X | SILO. | X | X | X | 2 |
| Adverse events | Xf | X | X | | X | | X | | X | | X | | X | | <i>K</i> | | X | X | X | 2 |
| eC-SSRS | X <sup>e,f</sup> | X | X | | X | | X | | X | | X | | X | ,'C | X | | X | X | X | 2 |
| HADS | X <sup>e,f</sup> | | X | | X | | X | | X | | X | 07 | X | 26,, | X | | X | X | X | 3 |
| HAQ-DI | X <sup>e,f</sup> | | X | | X | | X | | X | | X <sub>(</sub> | O, | /X | | X | | X | X | X | 2 |
| SF-36 | X <sup>e,f</sup> | | X | | X | | X | | X | | N) | 1311 | X | | X | | X | X | X | 3 |
| PGADA | X <sup>e,f</sup> | | X | | X | | X | | X | 3 | X | | X | | X | | X | X | X | 3 |
| PtAAP | X <sup>e,f</sup> | | X | | X | | X | | X | | X | | X | | X | | X | X | X | 3 |
| PsAID-9 | X <sup>e,f</sup> | | X | | X | | X | 0 | X | 0 | X | | X | | X | | X | X | X | 3 |
| TB questionnaire | X <sup>e,f</sup> | | X | | X | | X | | St. | | X | | X | | X | | X | X | X | 2 |
| Vital signs (pulse,<br>temperature, BP) <sup>g</sup> | Xe | Х | Х | | X | | X | USI | X | | X | | X | | X | | X | X | X | 3 |
| Body weight | X <sup>e,f</sup> | | X | | X | . ( | S.S. | | X | | X | | X | | X | | X | X | X | 2 |
| Physical examination <sup>h</sup> | X <sup>e,f</sup> | | | | , | Oir | | | X | | | | | | | | X | | X | 2 |
| TJC (78) and SJC (76) | X <sup>e,f</sup> | | X | | 30 | K | X | | X | | X | | X | | X | | X | X | X | 3 |
| BSA affected by PSO (BSA palm method) | X <sup>e,f</sup> | | X | 10 | X | | X | | X | | X | | X | | X | | X | X | X | 3 |
| PASIi | X <sup>e,f</sup> | | 7.38° | | X | | X | | X | | X | | X | | X | | X | X | X | 3 |
| onfidential | Xe,f | 00 | X | | X | | X | | X | | | | X | | | | X | | X | 3 |

11 Dec 2019

| Protocol activity | | | | | | | | T | reatr | nent l | Perio | d | | | | | | | | SFN |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Weeksa | EVb | 4 | 12 | 16 | 24 | 28 | 36 | 40 | 48 | 52 | 60 | 64 | 72 | 76 | 84 | 88 | 96 | 100 | W104/ | 101- |
| | | 8 | | 20 | | 32 | | 44 | | 56 | | 68 | | 80 | | 92 | | | ETO | |
| Visita | 1 | 2/3 | 4 | Hc | 5 | Hc | 6 | Hc | 7 | Hc | 8 | Hc | 9 | Hc | 10 | Hc | 11 | 12 | . 13 | |
| LDI | Xe,f | | X | | X | | X | | X | | X | | X | | X | | X | X | Э X | X |
| PhGADA | X <sup>e,f</sup> | | X | | X | | X | | X | | X | | X | | X | | X | X | X | X |
| ECG | Xe,f | | | | | | | | X | | | | | | | | (X) | | X | |
| Hematology/biochemistry/<br>urine pregnancy <sup>j,k</sup> | Xe,f | | Х | | Х | | Х | | X | | X | | Х | | X | and | O'X | X | X | X |
| Blood Sample for CRPk | Xe,f | | X | | X | | X | | X | | X | | X | | %, | | X | X | X | X |
| Blood sample for<br>bimekizumab plasma<br>concentrations <sup>k</sup> | Xe,f | | X | | X | | X | | X | | | 04 | X | Oblics | | | X | | X | X |
| Blood sample for anti-<br>bimekizumab antibodies <sup>k</sup> | X <sup>e,f</sup> | | X | | X | | X | | X | | | | Ö.X. | | | | X | | X | X |
| IGRA TB test <sup>1</sup> | Xe | | | | | | | | X | | ( ) | KI. | | | | | X | | | X |
| IXRS | X | X | X | | X | | X | | Χſ | ν, | 1/X | | X | | X | | X | X | X | X |
| Bimekizumab<br>administration | X | X | X | X | X | X | X | X | X | Q <sub>X</sub> O | X | X | X | X | X | X | X | X | | |


**UCB** 

Section 5.2 Schedule of study assessments, Table 5-1, Footnote '1'

Valiations thereof. It is recommended that the QuantiFERON TB GOLD test be performed. This assessment will be performed at study entry, unless an IGRA negative result is available less than 4 weeks prior to the first dose of open-label bimekizumab.

### Has been changed to:

It is recommended that the QuantiFERON TB GOLD test Test be performed. This assessment will be performed at study entry, unless an IGRA negative result is available less and any extension than 64 weeks prior to the first dose of open-label bimekizumab.

### Change #8

Section 6.1 Inclusion criteria (criterion #5)

5. Female subjects must be postmenopausal (at least 1 year), permanently sterilized (eg, tubal occlusion, hysterectomy, bilateral salpingectomy) or, if of childbearing potential (and engaged in sexual activity that could result in procreation), must be willing to use a highly effective method of contraception until 20 weeks after last administration of study medication, and have a negative pregnancy test at the last visit of PA0008.

Male subjects with a partner of childbearing potential must be willing to use a condom when sexually active, up until 20 weeks after the last administration of study medication (anticipated 5 half-lives).

## Has been changed to:

- 5. Female subjects must be postmenopausal (at least 1 year), permanently sterilized (eg, tubal occlusion, hysterectomy, bilateral salpingectomy) or, if of childbearing potential (and engaged in sexual activity that could result in procreation), must be willing to use a highly effective method of contraception until 20 weeks after last administration of study medication, and have a negative pregnancy test at the last visit of PA0008. The following methods are considered highly effective when used consistently and correctly:
  - combined (estrogen and progestogen) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal)
  - progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
    - intrauterine device (IUD)
  - intrauterine hormone-releasing system (IUS)
  - bilateral tubal occlusion
  - vasectomized partner

sexual abstinence if it is in accordance with a subject's preferred and common lifestyle. Subjects who use abstinence as a form of birth control must agree to abstain from heterosexual intercourse until 20 weeks after the last dose of IMP.

Male subjects with a partner of childbearing potential must be willing to use a condom when sexually active, up until 20 weeks after the last administration of study medication (anticipated 5 half-lives).

ange #9

tion 6.2 Exclusion criteria (criterion #2)

ubjects with any current sign or symptom that may indicate a medically significant infection (except for the common cold) and indicate a medically significant.

### Change #9

Section 6.2 Exclusion criteria (criterion #2)

2. Subjects with any current sign or symptom that may indicate a medically significant active infection (except for the common cold) or has had an infection requiring systemic antibiotics within 2 weeks of study entry.

### Has been changed to:

2. Subjects with any current sign or symptom that may indicate a medically significant active infection (except for the common cold) or has had an infection requiring systemic antibiotics within 2 weeks of study entry. The medical monitor must be consulted prior to subject's entry into PA0009 in such cases.

### Change #10

Section 6.3 Withdrawal criteria

The following was added to the withdrawal criteria:

- 12. Subjects with newly diagnosed inflammatory bowel disease (IBD) or with IBD flares during the study must:
  - Be referred, as appropriate, to a health care professional treating IBD, such as a gastroenterologist
  - Discontinue IMP and be followed-up until resolution of active IBD symptoms

If IBD flares increase in severity or frequency during the study, the Investigator should use clinical judgment in deciding whether the subject should continue in the study and contact the Medical Monitor and UCB study physician to confirm the subject's suitability for continued participation in the study.

## Change #11

Section 8.9 SFU Visit (20 weeks after the final dose of IMP)

The following procedures or assessments will be completed:

Record concomitant medications

- Record AEs
- eC-SSRS

- Description of active and BP)

  Measure body weight

  Perform a physical examination, including an evaluation for signs and symptoms of active TB and risk for exposure to TB

  Perform TJC/SJC

  Determine BSA affected by PSO using the BSA palm method the BSA affected by PSO is ≥3%, determine the PASI termine the MASES ermine the LDI

  Dorm the PhGADA

  ct samples for '

  e¹-

- If there has been a delay in menses, perform a urine pregnancy test
- Collect blood sample for CRP
- Collect blood sample for bimekizumab plasma concentrations and anti bimekizumab antibody detection
- Perform an IGRA TB test
- Record visit in the IXRS

### Has been changed to:

The following procedures or assessments will be completed:

- Record concomitant medications
- Record AEs
- eC-SSRS
- HADS

- Administer the HAQ-DI
- Administer the SF-36
- Administer the PGADA
- Administer the PtAAP
- Administer the PsAID-9
- Administer the TB questionnaire
- Measure vital signs (temperature, pulse, and BP)
- Measure body weight
- Perform a physical examination, including an evaluation for signs and symptoms of active
- Perform TJC/SJC
- Determine BSA affected by PSO using the BSA palm method
- If the BSA affected by PSO is >3%, determine the PASI
- Determine the MASES
- Determine the LDI

- Collect blood sample for bimekizumab plasma concentrations and anti bimekizumab
- Perform an IGRA TB test
- Record visit in the XRS

Section 9.1.1 Definition of AE

The following was added to the definition of AEs:

Adverse events that occurred during the PA0008 lead-in study and are still deemed ongoing at the time of enrolment (signed ICF) will be captured in the database and followed up, as described in Section 9.1.6.

Section 9.1.8 Pregnancy, paragraph 5

unintended pregnancy after hormonal contraceptive failure on mormonal contraceptive was correctly used), ectopic pregnancy, fetal demise, or any congenital anomaly/birth defect of the baby. Those SAEs must be additionally reported using the Investigator SAE Report Form.

Has been changed to:

A pregnancy becomes an SAE in the following circumstances: miscarriage, elective abortion when medically indicated (e.g. when pregnancy is endangering life or health of woman or when fetus will be born with severe abnormalities), unintended pregnancy after hormonal contraceptive failure (if the hormonal contraceptive was correctly used), ectopic pregnancy, fetal demise, or any congenital anomaly/birth defect of the baby. Those SAEs must be additionally reported using the Investigator SAE Report form.

Change #14
Section 9.5.1.4 Testing: identification/exclusion of alternative etiology, Table 9-4 (PDILI laboratory measurements)

| Virology- | Hepatitis A IgM antibody HBsAg |
|---|---|
| related | HBsAg OF JHO |
| | Hepatitis E IgM antibody |
| | HBcAb-IgM |
| | Hepatitis C RNA |
| | Cytomegalovirus IgM antibody |
| | Epstein-Barr viral capsid antigen IgM antibody (if unavailable, obtain heterophile antibody or monospot testing) |
| Immunology | Anti-nuclear antibody (qualitative and quantitative) |
| -0) | Anti-smooth muscle antibody (qualitative and quantitative) |
| othe | Type 1 anti-liver kidney microsomal antibodies (qualitative and quantitative) |
| Hematology | Eosinophil count |
| Orinalysis | Toxicology screen <sup>a</sup> |
| Chemistry | Amylase |
| | If total bilirubin ≥1.5xULN, obtain fractionated bilirubin to obtain % direct bilirubin |

| | Serum CPK and LDH to evaluate possible muscle injury causing transaminase elevation |
|---|---|
| Additional | Prothrombin time/INR <sup>b</sup> |
| | Serum pregnancy test |
| | PK sample |

- ALT=alanine aminotransferase; CPK=creatine phosphokinase; HBcAb-IgM=hepatitis B core antibody-IgM; HBsAg=hepatitis B surface antigen; IgM=immunoglobulin M; INR=international normalized ratio; LDH=lactate dehydrogenase; PDILI=potential drug-induced liver injury; PK=pharmacokinetic; RNA=ribonucleic acid; ULN=upper limit of normal
- <sup>a</sup> For detecting substances (ie, amphetamines, benzodiazepines, opioids, marijuana, cocaine, phencyclidine, and tricyclic antidepressants), additional tests may be performed based on the Investigator's medical judgment and patient's history.
- b Measured only for subjects with ALT >8xULN, elevations in total bilirubin, and symptoms of hepatitis or hypersensitivity. Hepatitis symptoms include fatigue, nausea, vomiting, and right upper quadrant pain or tenderness; hypersensitivity symptoms include eosinophilia (>5%), rash, and fever (without clear alternative cause).

## Has been changed to:

| 1 | ,,0 |
|---|---|
| Virology- | Hepatitis A IgM antibody |
| related | HBsAg |
| | Hepatitis E IgM antibody |
| | Hepatitis A IgM antibody HBsAg Hepatitis E IgM antibody HBcAb-IgM Hepatitis C RNA |
| | Hepatitis C RNA |
| | Cytomegalovirus IgM antibody |
| | Epstein-Barr viral capsid antigen IgM antibody (if unavailable, obtain heterophile antibody or monospot testing) |
| Immunology | Anti-nuclear antibody (qualitative and quantitative) |
| | Anti-smooth muscle antibody (qualitative and quantitative) |
| | Type 1 anti-liver kidney microsomal antibodies (qualitative and quantitative) |
| Hematology | Eosinophil count |
| Urinalysis | Toxicology screen <sup>a</sup> |
| Chemistry | Amylase |
| nent | ALT, AST |
| | If total bilirubin ≥1.5xULN, obtain fractionated bilirubin to obtain % direct bilirubin |
| | Serum CPK and LDH to evaluate possible muscle injury causing transaminase elevation |

| Additional | Prothrombin time/INR <sup>b</sup> |
|------------|-----------------------------------|
| | Serum pregnancy test |
| | PK sample |

- ALT=alanine aminotransferase; AST=aspartate aminotransferase; CPK=creatine phosphokinase; HBcAb-IgM=hepatitis B core antibody-IgM; HBsAg=hepatitis B surface antigen; IgM=immunoglobulin M; INR=international normalized ratio; LDH=lactate dehydrogenase; PDILI=potential drug-induced liver injury; PK=pharmacokinetic; RNA=ribonucleic acid; ULN=upper limit of normal
- <sup>a</sup> For detecting substances (ie, amphetamines, benzodiazepines, opioids, marijuana, cocaine, phencyclidine, and tricyclic antidepressants), additional tests may be performed based on the Investigator's medical judgment and patient's history.
- <sup>b</sup> Measured only for subjects with ALT >8xULN, elevations in total bilirubin, and symptoms of hepatitis or hypersensitivity. Hepatitis symptoms include fatigue, nausea, vomiting, and right upper quadrant pain or tenderness; hypersensitivity symptoms include eosinophilia (>5%), rash, and fever (without clear alternative cause).

Tuberculosis and TB risk factor assessment and management, 2nd paragraph Section 9.6.5

Prior to administration of IMP, subjects will have an IGRA test (QuantiFERON TB GOLD is recommended) and examination for signs and symptoms of TB unless an IGRA negative result is available less than 4 weeks prior to the first dose of open label bimekizumab. In addition, each subject will complete a TB questionnaire with questions directed at symptoms of TB and potential exposure to TB.

## Has been changed to:

Prior to administration of IMP, subjects will have an IGRA test (QuantiFERON TB TestGOLD is recommended) and examination for signs and symptoms of TB unless an IGRA negative result is available less than 64 weeks prior to the first dose of open label bimekizumab. In addition, each subject will complete a TB questionnaire with questions directed at symptoms of TB and potential exposure to TB.

## Change #16

Section 9.6.5.1 Tuberculosis assessment by IGRA

During conduct of the study, the TB assessment by IGRA (QuantiFERON TB Test is recommended) will be performed at study entry (unless an IGRA negative result is available less than 4 weeks prior to the first dose of open-label bimekizumab) and should be repeated at (latent or active) is suspected or if there are doubts regarding test results. If latent or active TB is identified, subject must undergo appropriate study-specified withdrawal procedures.

### Has been changed to:

During conduct of the study, the TB assessment by IGRA (QuantiFERON TB GOLDTest is negative, or indeterminate. UCB also recommends that a TB specialist be consulted where TB (latent or active) is suspected or if there are doubts regarding test results. If latent or active TB is identified, subject must undergo appropriate study-specified withdrawal procedures.

Change #47 recommended) will be performed at study entry (unless an IGRA negative result is available less tensions of varif

### Change #17

**UCB** 

Section 13.8 Handling of dropouts or missing data, paragraph 3

Missing binary efficacy variables will be imputed using nonresponder imputation (NRI). In NRI, each subject with missing data or who has prematurely finished the study will be counted as a nonresponder.

For missing continuous efficacy variables, a multiple imputation (MI) approach will be used. In MI, the missing value is replaced by a set of plausible values, where each value is a Bayesian draw from the conditional distribution of the missing data given the observed data. Non-monotone missing data (ie, intermittent missing data) will be imputed several times with the Markov Chain Monte Carlo (MCMC) method and monotone missing data will be imputed using a monotone regression model. Each set of imputed data will then be summarized and the summaries will be combined into a single inference (Carpenter and Kenward, 2013).

Imputation of efficacy data will be performed for only those assessments that the patient had in PA0008. Safety data will not be imputed.

As a sensitivity analysis, all efficacy variables will be analyzed based on observed data. Subjects with missing data or who have prematurely finished the study will be treated as missing.

## Has been changed to:

Missing binary efficacy variables will be imputed using nonresponder imputation (NRI). In NRI, each subject with missing data or who has prematurely finished the study will be counted as a nonresponder.

For missing continuous efficacy variables, a multiple imputation (MI) approach will be used. In MI, the missing value is replaced by a set of plausible values, where each value is a Bayesian draw from the conditional distribution of the missing data given the observed data. Non monotone missing data (ie, intermittent missing data) will be imputed several times with the Imputation of efficacy data will be performed for only those as PA0008. Safety data will not 1 Markov Chain Monte Carlo (MCMC) method and monotone missing data will be imputed using a monotone regression model. Each set of imputed data will then be summarized and the

Imputation of efficacy data will be performed for only those assessments that the patient had in

As a sensitivity analysis, all efficacy variables will be analyzed based on observed data. Subjects with missing data or who have prematurely finished the study will be treated as missing.


Markedly abnormal laboratory values, Tables 17-1 (Definitions of markedly Section 17.1 abnormal hematology values) and 17-2 (Definitions of markedly abnormal biochemistry values)

Amended units in both table headers:

| | Markedly Abno | y Abnormal Definition |
|----------------------|---------------|-----------------------|
| Parameter (SI units) | Low | High |
| | | 100 |

### Has been changed to:

| | Markedly Abnormal Definition | |
|--------------------------|------------------------------|------|
| Parameter (SIRCTC units) | Low | High |

### Change #19

Markedly abnormal laboratory values, Table 17-1 (Definitions of markedly Section 17.1 abnormal hematology values), abbreviations in table footer:

LLN=lower limit of normal; N/A = Not Applicable; SI = standard international

### Has been changed to:

LLN=lower limit of normal; N/A = Not Applicable; SI = standard international RCTC= Rheumatology Common Toxicity Criteria

## Change #20

Markedly abnormal laboratory values, Table 17-2 (Definitions of markedly Section 17.1 abnormal biochemistry values), abbreviations in table footer:

ALT=alanine aminotransferase; AST=aspartate aminotransferase; N/A=Not applicable; SI=standard international; ULN=upper limit of normal

## Has been changed to:

LLN=lower limit of normal; N/A = Not Applicable; SI=standard international RCTC= Rheumatology Common Toxicity Criteria

### **Protocol Amendment 3** 17.4

### Rationale for the amendment

The purpose of this nonsubstantial amendment is as follows:

- with PSO involving at least 3% of BSA at

  output estudy contact information

  To make minor spelling, editorial, and formatting changes throughout the document odifications and changes

  bal change

  following global changes were made.

  The compact

### **Modifications and changes**

### Global change

The following global changes were made:

- The company name was changed from UCB Biopharma SPRL to UCB Biopharma SRL
- The term "legal representative" was deleted from protocol, as it is not applicable to PA0009
- Throughout the protocol "Baseline" was changed to "Baseline of PA0008" or similar wording

  Throughout the protocol "Baseline" was changed to "Baseline of PA0008" or similar wording

  Throughout the protocol "Baseline of PA0008" or similar wording

  Throughout the protocol "Baseline of PA0008" or similar

## Specific changes

### Change #1

**Study Contact Information** 

## Sponsor

UCB BIOPHARMA SPRL

Allée de la Recherche 60

1070 Brussels

**BELGIUM** 

## Sponsor Study Physician

| Name: | , MD, MSc, PhD |
|----------|-----------------|
| Address: | UCB Pharma Ltd. |
| MINO | 208 Bath Road |
| 0 | Slough, SL1 3WE |
| | UNITED KINGDOM |
| Phone: | |

## **Clinical Project Manager**

| Name: | , Clinical Project Manager |
|----------|----------------------------|
| Address: | UCB BIOSCIENCES Inc. |
| | 8010 Arco Corporate Drive |
| | Raleigh, NC 27617 |
| | UNITED STATES |
| Phone: | |

## **Clinical Trial Biostatistician**

| Name: | et et |
|---|---|
| Address: | UCB BIOSCIENCES GmbH Alfred-Nobel-Strasse 10 40789 Monheim am Rhein GERMANY |
| Phone: | ot oplie |

## Has been changed to:

## **Sponsor**

UCB BIOPHARMA SPRLSRL

Allée de la Recherche 60

1070 Brussels

**BELGIUM** 

# Sponsor Study Physician

| Name: | , MD, MSc, PhD |
|---------|----------------------------|
| Address | UCB <del>Pharma Ltd.</del> |
| ne s | 208 Bath Road |
| not b | Slough, SL1 3WE |
| 300 | UNITED KINGDOM |
| Phone: | |

### **Clinical Project Manager**

| Name: | , Clinical Project Manager |
|----------|-----------------------------------------|
| Address: | UCB BIOSCIENCES Inc. |
| | 8010 Arco Corporate Drive-208 Bath Road |
| | Raleigh, NC 27617 Sough, SL1 3WE |
| | UNITED STATES-UNITED KINGDOM |
| Phone: | |

### **Clinical Trial Biostatistician**

| Name: | CAT COL |
|----------|---------------------------------------|
| Address: | UCB BIOSCIENCES GmbH |
| | Alfred-Nobel-Strasse 10-208 Bath Road |
| | 40789 Monheim am Rhein-Slough SL1 3WE |
| | GERMANY UNITED KINGDOM |
| Phone: | |

The following abbreviations were added:

PFS prefilled syring and authorization

TEAE treatment-emergent adverse event

### Change #3

Section 1 Summary, paragraphs 5 and 6

The primary objective of PA0009 is to assess the long-term safety and tolerability of bimekizumab administered over a period of up to 100 weeks (~2 years). The primary safety variables are the incidences of adverse events (AEs) and serious adverse events (SAEs).

The secondary objective is to assess the long-term efficacy of bimekizumab over a period of up to 104 weeks (~2 years). The secondary efficacy variables include the American College of Rheumatology 20% (ACR20) response at Week 48 (with a responder defined as a subject with an improvement from PA0008 Baseline and PA0009 entry value of ≥20% in the swollen and tender joint counts and at least 3 of the other 5 components of the core set of American College of Rheumatology [ACR] response measures), American College of Rheumatology 50% (ACR50) response at Week 48; American College of Rheumatology 70% (ACR70) response at Week 48, change from Baseline and PA0009 entry value in the Maastricht Ankylosing Spondylitis Enthesitis Index (MASES) at Week 48, change from Baseline and PA0009 entry value in the Leeds Dactylitis Index (LDI) at Week 48, the Psoriasis Area and Severity Index 75

(PASI75) response, and the Psoriasis Area and Severity Index 90 (PASI90) response at Week 48. The secondary safety variable is the withdrawal due to AEs.

### Has been changed to:

The primary objective of PA0009 is to assess the long-term safety and tolerability of bimekizumab administered over a period of up to 100 weeks (~2 years). The primary safety variables are the incidences of treatment-emergent adverse events (TEAEs) and treatment-emergent serious adverse events (SAEs).

The secondary objective is to assess the long-term efficacy of bimekizumab over a period of up to 104 weeks (~2 years). The secondary efficacy variables include the American College of Rheumatology 20% (ACR20) response at Week 48 (with a responder defined as a subject with an improvement from PA0008 Baseline and PA0009 entry value of >20% in the swollen and tender joint counts and at least 3 of the other 5 components of the core set of American College of Rheumatology [ACR] response measures), American College of Rheumatology 50% (ACR50) response at Week 48; American College of Rheumatology 70% (ACR70) response at Week 48, change from **PA0008** Baseline and PA0009 entry value in the Maastricht Ankylosing Spondylitis Enthesitis Index (MASES) at Week 48, change from PA0008 Baseline and PA0009 entry value in the Leeds Dactylitis Index (LDI) at Week 48, the Psoriasis Area and Severity Index 75 (PASI75) response, and the Psoriasis Area and Severity Index 90 (PASI90) response at Week 48. The secondary safety variable is the withdrawal due to AEs-TEAEs.

### Change #4

Section 4 Study Variables

Changes from Baseline will be analyzed relative to the Baseline Visit of PA0008. Variables measured at the start of PA0009 will be referred to as PA0009 entry values.

## Has been changed to:

All efficacy variables Change from Baseline will be analyzed relative to the Baseline Visit of PA0008. Safety v-variables measured at the start of PA0009 will be referred to as PA0009 entry values.

## Change #5

Section 4.1.1 Primary safety variables

The primary safety variables are the incidences of AEs and SAEs.

## Has been changed to:

The primary safety variables are the incidences of TEAEs and treatment-emergent SAEs.

## Change #6

Section 4.2.1 Secondary safety variable

The secondary safety variable is the withdrawal due to AEs.

### Has been changed to:

The secondary safety variable is the withdrawal due to AEsTEAEs.

### Change #7

Section 4.2.2 Secondary efficacy variables

The secondary efficacy variables are:

- ACR20, ACR50, and ACR70 response at Week 48
- Change from Baseline and PA0009 entry value in MASES at Week 48
- Change from Baseline and PA0009 entry value in the LDI at Week 48
- PASI75 and PASI90 response at Week 48

### Has been changed to:

The secondary efficacy variables are:

- ACR20, ACR50, and ACR70 response at Week 48
- which and any extensions or variations thereof. Change from Baseline of PA0008 and PA0009 entry value in MASES at Week 48
- Change from Baseline of PA0008 and PA0009 entry value in the LDI at Week 48
  PASI75 and PASI90 response at Week 48

  nange #8
  ction 4.3.1 Safety variables

  her safety variables are listed below.

### Change #8

Section 4.3.1 Safety variables

Other safety variables are listed below

- Change from Baseline and PA0009 entry value in clinical laboratory variables (hematology and biochemistry)
- Change from Baseline and PA0009 entry value in vital signs (pulse, temperature, and blood pressure) and body weight

## Has been changed to:

Other safety variables are listed below.

- Change from Baseline and PA0009 entry value in Laboratory Baseline (defined as the earliest date in PA0009 at or prior to PA0009 Week 12) for clinical laboratory variables (hematology and biochemistry, excepting high-sensitivity C-reactive protein [CRP]) at each visit)
- Change from Baseline of PA0008 and PA0009 entry value in vital signs (pulse, temperature, and blood pressure) and body weight

Section 4.3.2 Efficacy variables

, sions or variations thereof. Other efficacy variables are listed below and will be evaluated at scheduled visits in accordance with the schedule of study assessments in Table 5-1.

- ACR20, ACR50, and ACR70 response
- PASI100 response
- PASI75 and PASI90 response
- Minimal Disease Activity (MDA) as defined in Table 10-3
- Change from Baseline and PA0009 entry value in the Disease Activity Score-28 based on C-reactive protein (DAS28 [CRP]) by visit
- Change from Baseline and PA0009 entry value in MASES
- Change from Baseline and PA0009 entry value in the LDI
- Change from Baseline and PA0009 entry value in Psoriatic Arthritis Impact of Disease (PsAID)-9
- Change from Baseline and PA0009 entry value in Short Form 36-item Health Survey (SF-36)
- Change from Baseline and PA0009 entry value in the Hospital Anxiety and Depression Scale (HADS): HADS-Anxiety (HADS-A) and HADS-Depression (HADS-D) scores
- Depression and anxiety status "normal" as defined by HADS-D and HADS-A <8

### Has been changed to:

Other efficacy variables are listed below and will be evaluated at scheduled visits in accordance with the schedule of study assessments in Table 5-1.

- ACR20, ACR50, and ACR70 response
- PASI75, PASI90, and PASI100 response
- PASI75 and PASI90 response
- Minimal Disease Activity (MDA) as defined in Table 10-3
- Change from Baseline of PA0008 and PA0009 entry value in the Disease Activity Score-28 based on C-reactive protein (DAS28 [CRP]) by visit
- Change from Baseline of PA0008 and PA0009 entry value in MASES
- Change from Baseline of PA0008 and PA0009 entry value in the LDI
- Change from Baseline of PA0008 and PA0009 entry value in Psoriatic Arthritis Impact of Disease (PsAID)-9
- Change from Baseline of PA0008 and PA0009 entry value in Short Form 36-item Health Survey (SF-36)

- Change from Baseline of PA0008 and PA0009 entry value in the Hospital Anxiety and Depression Scale (HADS): HADS-Anxiety (HADS-A) and HADS-Depression (HADS-D) scores
- Depression and anxiety status "normal" as defined by HADS-D and HADS-A <8

Table 5-1: Schedule of study assessments (footnote a)

<sup>a</sup> Visit windows are ±7 days from the scheduled visit day (relative to the first dose) with a minimum of 21 days and a maximum of 35 days in between doses at all visits except the SFU Visit. The SFU Visit window is -3 to +7 days from last dose.

### Has been changed to:

a Visit windows are ±7 days from the scheduled visit day (relative to the first dose) with a minimum of 21 days and a maximum of 35 days in between doses at all visits except the SFU Visit. For the SFU Visit, the visit should occur no more than window is 3 days prior to the scheduled visit date and within days after the scheduled visit date (-3 days/-to +7 days) from last dose.

### Change #11

Table 5-1: Schedule of study assessments (footnote it

<sup>1</sup> If the BSA affected by PSO was ≥3% at this visit, determine the PASI.

### Has been changed to:

i If the BSA affected by PSO was ≥3% at this visit Baseline of PA0008, determine the PASI.

## Change #12

Section 6.1 Inclusion criteria, #1 and #

- 1. An Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written Informed Consent form is signed and dated by the subject or legal representative.
- 2. Subject or legal representative is considered reliable and capable of adhering to the protocol (eg, able to understand and complete questionnaires), visit schedule, or medication intake according to the judgment of the Investigator.

### Has been changed to:

- 1a. An Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written
- 2a. Subject or legal representative is considered reliable and capable of adhering to the protocol

11 Dec 2019

PA0009

### Change #13

Section 6.3.1 Potential drug-induced liver injury investigational medicinal product discontinuation criteria, paragraph 2

The PDILI criteria below require immediate and permanent discontinuation of IMP:

### Has been changed to:

The PDILI criteria below require immediate and permanent discontinuation of IMP:

### Change #14

Section 7.1 Description of investigational medicinal product

The IMP will consist of the following:

Bimekizumab will be supplied as a clear to opalescent, colorless to slightly brown, sterile, preservative–free solution in a

### Has been changed to:

The IMP will consist of the following:

• Bimekizumab will be supplied as a clear to opalescent, colorless to slightly brown, sterile, preservative—free solution in a 1mL prefilled syringe (PFS).

for sc injection.

## Change #15

Section 8.1 Visit 1

• If the BSA affected by PSO is ≥3%, determine the Psoriasis Area and Severity Index (PASI)\*

## Has been changed to:

• If the BSA affected by PSO is ≥3% at Baseline of PA0008, determine the Psoriasis Area and Severity Index (PASI)\*

## Change #16

Section 8.3 Week 12 (Visit 4), Week 24 (Visit 5), Week 36 (Visit 6), and Week 72 (Visit 9)

If the BSA affected by PSO is  $\geq 3\%$ , determine the PASI

## Has been changed to:

• If the BSA affected by PSO is  $\geq 3\%$  at Baseline of PA0008, determine the PASI

**UCB** 

Section 8.5 Week 48 (Visit 7) and Week 96 (Visit 11)

If the BSA affected by PSO is  $\geq 3\%$ , determine the PASI

### Has been changed to:

any extensions of variations thereof. If the BSA affected by PSO is  $\geq 3\%$  at Baseline of PA0008, determine the PASI

### Change #18

Section 8.6 Week 60 (Visit 8) and Week 84 (Visit 10)

If the BSA affected by PSO is  $\geq 3\%$ , determine the PASI

### Has been changed to:

If the BSA affected by PSO is  $\geq 3\%$  at Baseline of PA0008, determine the PASI

### Change #19

Section 8.7 Week 100 (Visit 12)

If the BSA affected by PSO is  $\geq 3\%$ , determine the PASI

### Has been changed to:

If the BSA affected by PSO is ≥3% at Baseline of PA0008, determine the PASI

### Change #20

Section 8.8 Week 104 (Visit 13) or Early Termination Visit

If the BSA affected by PSQ is ≥3%, determine the PASI

## Has been changed to:

If the BSA affected by PSO is ≥3% at Baseline of PA0008, determine the PASI

# Change #21

Section 9.1.3 AEs for special monitoring

UCB has identified AEs for special monitoring (AESM). An AESM is an AE or safety topic for which special monitoring, additional data collection activities, and/or enhanced signal detection activities (within UCB), are considered appropriate. Identified AESM can be of particular concern based on findings from the IMP clinical program to date, potential risks generally associated with biologic immunomodulators, or comorbidities and risk factors prevalent in the study population.

Adverse events for special monitoring for this study include: serious infections (including opportunistic infections and TB, see Section 9.6.5), cytopenias, hypersensitivities, suicide ideation or behavior (assessed using the eC-SSRS), depression and anxiety (assessed using the HADS, see Section 10.15), major cardiovascular events and liver function test changes/enzyme elevations (ALT, AST, and bilirubin; see Section 9.1.5), malignancies, and inflammatory bowel diseases.

UCB has identified AEs for special monitoring (AESM). An AESM is an AE or Pre-specified safety topics of interest for which special monitoring, additional data collection activities enhanced signal detection activities (within UCB), are considered. neutropenia, hypersensitivity, suicidal ideation and behavior, depression, major cardiovascular events, liver function test changes/enzyme elevations, malignancies, and inflammatory bowel diseases (with gastroenterology referral, as appropriate). This is based on findings from the IMP clinical program to date, potential risks generally associated with biologic immunomodulators, or comorbidities and risk factors prevalent in the study population findings from other medicines with a related mechanism of action. There are no specific AE reporting requirements for these topics, however special monitoring, additional data collection activities, and/or enhanced signal detection activities (within UCB) are in place.

Adverse events for special monitoring for this study include; serious infections (including opportunistic infections and TB, see Section 9.6.5), cytopenias, hypersensitivities, suicide ideation or behavior (assessed using the eC-SSRS), depression and anxiety (assessed using the HADS, see Section 10.15), major cardiovascular events and liver function test changes/enzyme elevations (ALT, AST, and bilirubin; see Section 9.1.5), malignancies, and inflammatory bowel diseases.

### Change #22

Section 9.1.6 Follow-up of AEs, first paragraph

An AE should be followed until it has resolved, has a stable sequelae, the Investigator determines that it is no longer clinically significant, or the subject is lost to follow-up. This follow-up requirement applies to AEs, SAEs, AESIs, and AESMs; further details regarding follow-up of PDILI events are provided in Section 9.5.1.5. Information on SAEs obtained after clinical database lock will be captured through the Patient Safety (PS) database without limitation of time.

## Has been changed to:

An AE should be followed until it has resolved, has a stable sequelae, the Investigator determines that it is no longer clinically significant, or the subject is lost to follow-up. This follow-up requirement applies to AEs, SAEs, AESIs, and other safety topics of interestAESMs; further details regarding follow-up of PDILI events are provided in Section 9.5.1.5. Information on SAEs obtained after clinical database lock will be captured through the Patient Safety (PS) database without limitation of time.

Section 9.2.3 Follow-up of SAEs

tollow-up requirement applies to AEs, SAEs, AESIs, and AESMs; further details regarding follow-up of PDILI events are provided in Section 9.5.1.5. Information on SAEs obtained after clinical database lock will be captured through the PS database without limitation of time.

Has been changed to:

An SAE should be followed until it has resolved, has a stable sequelae, the Investigator determines that it is no longer clinically significant, or the subject is lost to follow-up. This follow-up requirement applies to AEs, SAEs, AESIs and AESIs are also at the AESIs and AESIs and AESIs and AESIs are also at the AESIs and AESIs are also at the AESIs and AESIs and AESIs are also at the AESIs and AESIs are also at the AE

where ad in Section and the used to support any marketing authorization and the used to support any marketing authorization and the used to support any marketing authorization and the used to support any marketing authorization. further details regarding follow-up of PDILI events are provided in Section 9.5.1.5. Information on SAEs obtained after clinical database lock will be captured through the PS database without

### Required investigations and follow-up for PDILI **Table 9-3:**

| Change | | | Bimekizumab | | | PA0009 |
|---|---|---|---|---|---|---|
| Table 9-3: Required investigatio | | ns and follow-up for PDILI Immediate | | Follow-up | | |
| ALT or Total bilirubin | | | | Actions | Testing Evaluation | |
| ≥3xULN | ≥2xULN <sup>b</sup> | NA | Hepatology consult. <sup>c</sup> Medical Monitor must be notified within 24 hours | Immediate, permanent IMP discontinuation. | repeat liver chemistry values and additional | Monitoring of liver chemistry values at least twice per week until values normalize, stabilize, or return to within Baseline values. <sup>d</sup> |
| ≥3xULN | NA | Yes | (eg, by laboratory alert)<br>and subject discussed with<br>Medical Monitor ASAP. | , cari | | |
| ≥5xULN | NA | NA | Need for hepatology consult to be discussed. (required if ALT or AST ≥8xULN) Medical Monitor must be notified within 24hours (eg, by laboratory alert) and subject discussed with Medical Monitor ASAP | Immediate, permanent IMP discontinuation | | |
| | | it cannot be used to | Medical Monitor ASAP | | | |

**Table 9-3:** Required investigations and follow-up for PDILI

| Table 9-3 | | red investigatio | ns and follow-up fo | | <u> </u> | - Jajia |
|---|---|---|---|---|---|---|
| Laborate ALT or AST | Total<br>bilirubin | Symptoms <sup>a</sup> of hepatitis or hypersensitivity | atitis or requirements | I | Testing Evaluation | |
| ≥3xULN<br>(and ≥2x<br>baseline) and<br><5xULN<br>(and ≥2x<br>baseline) | <2xULN | No | Discussion with Medical Monitor required. Consider need for hepatology consult if there is no evidence of resolution (see Follow-up requirements) c | Further investigation – immediate IMP discontinuation not required (see Section 9.5.1.2). IMP discontinuation required if any of the following occur: Subject eannot comply with monitoring schedule. Liver chemistry values continue to increase Liver chemistry values remain ≥3xULN (and ≥2xbaseline) after 2 weeks of monitoring without evidence of resolution | Essential: Every attempt must be made to have repeat liver chemistry values and additional testing completed within 48hours at the site with HCP (see Section 9.5.1.4). | <ul> <li>Monitoring of liver chemistry values least twice per week for 2 weeks.<sup>d</sup></li> <li>Immediate IMP discontinuation required if liver chemistry values continue to increase.</li> <li>After 2 weeks of monitoring liver chemistry values:</li> <li>Discontinue IMP if levels remain ≥3xULN (and ≥2x baseline) without evidence of resolution<sup>d</sup></li> <li>Continue to monitor until values normalize, stabilize, or return to within baseline values<sup>d</sup>.</li> </ul> |
| | cuner | i cannot be used to | SUPPORT ANY MIC | | | |

## Has been changed to:

**Table 9-3:** Required investigations and follow-up for PDILI

| Has bee | n changed | l to: | Bimekizumab | | | PA0009 |
|---|---|---|---|---|---|---|
| Table 9- | | red investigatio | ons and follow-up fo | | I | or de |
| ALT or<br>AST | Total bilirubin | Symptoms <sup>a</sup> of hepatitis or hypersensitivity | Consultation requirements | Actions | Testing extensi | Follow-up Evaluation |
| ≥3xULN | ≥2xULN <sup>b</sup> | NA | Hepatology consult. <sup>c</sup> Medical Monitor must be notified within 24 hours (eg, by laboratory alert) | Immediate <del>, permanent</del> IMP discontinuation. | Essential Must have<br>repeat liver chemistry<br>values and additional<br>testing completed | Monitoring of liver chemistry values at least twice per week until values normalize, stabilize, or return to within Baseline values. <sup>d</sup> |
| ≥3xULN | NA | Yes | and subject discussed with<br>Medical Monitor ASAP. | , jicati' | ASAP (see<br>Section 9.5.1.4);<br>recommended to | |
| ≥5xULN | NA | NA | Need for hepatology consult to be discussed. (required if ALT or AST ≥8xULN) Medical Monitor must be notified within 24hours (eg, by laboratory alert) and subject discussed with Medical Monitor ASAP. | Immediate, permanent IMP discontinuation | occur at the site with HCP. | |
| | | it cannot be used to | subject discussed with Medical Monitor ASAR | | | |
| | *OCALL | | Page 10 | | | |

**Table 9-3:** Required investigations and follow-up for PDILI

| UCB<br>Clinical Stud | y Protocol | | Ві | imekizumab | | PA0009 |
|---|---|---|---|---|---|---|
| Table 9-3 | | red investigatio | ons and follow-up fo | | I | ariatilo. |
| Laborat ALT or | ory value<br>Total | Symptoms <sup>a</sup> of | Immediate Follow-up of Consultation Actions Testing Evaluation | | Follow-up Evaluation | |
| AST | bilirubin | hepatitis or<br>hypersensitivity | requirements | Actions | resung | Evaluation |
| ≥3xULN (and ≥2x baseline) and <5xULN (and ≥2x baseline) | <2xULN | No | Discussion with Medical Monitor required. Consider need for hepatology consult if there is no evidence of resolution (see Follow-up requirements) c | Further investigation – immediate IMP discontinuation not required (see Section 9.5.1.2). IMP discontinuation required if any of the following occur: Subject cannot comply with monitoring schedule. Liver chemistry values continue to increase Liver chemistry values remain ≥3xULN (and ≥2xbaseline) after 2 weeks of monitoring without evidence of resolution | Essential: Every attempt must be made to have repeat liver chemistry values and additional testing completed within 48hours at the site with HCP (see Section 9.5.1.4). | <ul> <li>Monitoring of liver chemistry values at least twice per week for 2 weeks.<sup>d</sup></li> <li>Immediate IMP discontinuation required if liver chemistry values continue to increase.</li> <li>After 2 weeks of monitoring liver chemistry values:</li> <li>Discontinue IMP if levels remain ≥3xULN (and ≥2x baseline) without evidence of resolution<sup>d</sup></li> <li>Continue to monitor until values normalize, stabilize, or return to within Baseline values<sup>d</sup>.</li> </ul> |

Section 9.5.1.2 Immediate action: determination of IMP discontinuation, paragraph 2

The immediate action is dependent on the laboratory values and symptoms of hepatitis or hypersensitivity and ranges from continuation of IMP (followed by immediate investigation) to immediate and permanent discontinuation (see Section 6.3.1 and Table 9-3 for details).

### Has been changed to:

The immediate action is dependent on the laboratory values and symptoms of hepatitis or hypersensitivity and ranges from continuation of IMP (followed by immediate investigation) to immediate and permanent discontinuation (see Section 6.3.1 and Table 9-3 for details).

### Change #26

Section 10.8 ACR20, ACR50, and ACR70 response, paragraph 1

The ACR20, ACR50, and ACR70 response rates are based on a 20%, 50%, and 70% or greater improvement relative to Baseline of PA0008 and PA0009 entry values in the following measures:

### Has been changed to:

The ACR20, ACR50, and ACR70 response rates are based on a 20%, 50%, and 70% or greater improvement relative to Baseline of PA0008 and PA0009 entry values in the following measures:

Change #27
Section 10.10 Psoriasis Area and Severity Index (PASI), paragraph 1

Psoriasis Area and Severity Index will be assessed in all subjects with study entry BSA affected by PSO  $\geq$ 3% determined by the method described in Section 10.9 (ie, the BSA palm method).

## Has been changed to:

Psoriasis Area and Severity Index will be assessed in all subjects with study entry BSA affected by PSO  $\geq$ 3% at Baseline of PA0008 determined by the method described in Section 10.9 (ie, the BSA palm method).

## Change #28

Section 10.10 Psoriasis Area and Severity Index (PASI), last paragraph

The PASI75, PASI90, and PASI100 responses are based on at least 75%, 90%, and 100% improvement in the PASI score compared to Baseline in PA0008 and PA0009 entry values. Thereafter PASI will be assessed for the purposes of determining response only in subjects with PSO involving at least 3% of BSA at study entry.

### Has been changed to:

S Or Variations thereof. The PASI75, PASI90, and PASI100 responses are based on at least 75%, 90%, and 100% improvement in the PASI score compared to Baseline in PA0008 and PA0009 entry values. Thereafter PASI will be assessed analyzed for the purposes of determining response only in subjects with PSO involving at least 3% of BSA at study entry Baseline of PA0008.

### Change #29

Section 13.1 Definition of analysis sets, last paragraph

The Full Analysis Set (FAS) will consist of all enrolled subjects who receive at least I dose of the IMP and have a valid measurement for at least 1 efficacy variable at PA0009 study entry.

### Has been changed to:

The Full Analysis Set (FAS) will consist of all enrolled subjects who receive at least 1 dose of the IMP and have a valid measurement for at least 1 efficacy variable at after PA0009 study

change #30
Section 13.3.1 Safety analyses, last 2 paragraphs
Change from PA0009 entry values in laboratory and vital signs variables will be summarized descriptively by visit and by treatment group at completion of PA0008.

All safety analyses will be conducted for both subpopulations.

## Has been changed to:

Change from PA0009 entry PA0008 Baseline values in laboratory and vital signs variables will be summarized descriptively by visit and by treatment group at completion of PA0008. Change from PA0009 Laboratory Baseline values in clinical laboratory variables (hematology and biochemistry, excepting high-sensitivity CRP) will be summarized descriptively by visit and by treatment group at completion of PA0008.

Due to a change in laboratory vendor between PA0008 and PA0009, laboratory values (excepting CRP) will use the PA0009 Laboratory Baseline, defined as the earliest postentry visit value recorded in PA0009. Change from PA0009 Laboratory Baseline will be calculated for these parameters. (The CRP values from the 2 analyzing laboratories have been calibrated, so change from PA0008 Baseline will be calculated for that parameter.)

All safety analyses will be conducted for both subpopulations.

Section 13.4 Planned efficacy analyses, paragraphs 2 and 3

Change from Baseline or PA0009 entry values of all continuous variables will be summarized descriptively by visit, by randomized treatment group, and by treatment group at completion of PA0008.

Has been changed to:

Responder

Responder variables (eg, ACR20 response) will be derived relative to the Baseline of PA0008 and PA0009 entry values, and summarized descriptively. Percentages will be summarized descriptively by visit, by randomized treatment group, and by treatment group at PA0009 entry.

Change from Baseline of PA0008 or PA0009 entry values of all continuous variables will be summarized descriptively by visit, by randomized treatment group, and by treatment group at Concomitant DMARD status at PA0009 entry it and its speed to:

Concomitant DMARD status at PA0009 entry it is speed to: completion of PA0008.

### Change #32

Section 13.4.1 Subgroup analysis, last bullet

## Has been changed to:

• Concomitant DMARD status at Baseline of PA0008 PA0009 entry

## Change #33

Section 13.8 Handling of dropouts or missing data

The following paragraph was added to the end of this section:

As a sensitivity analysis, the ACR, PASI, LDI, MASES, and MDA efficacy variables will be analyzed based on observed data in addition to a sensitivity analysis based on multiple imputation of ACR component scores and PASI scores for the ACR and PASI response variables, respectively. Subjects with missing data or who have prematurely finished the study will be treated as missing.

## Change #34

Section 13.9 Planned interim analysis and data monitoring

No formal interim analysis is planned for this study.

The document control be used to support any materials as the control of the contr


## 18 DECLARATION AND SIGNATURE OF INVESTIGATOR

I confirm that I have carefully read and understood this protocol and agree to conduct this clinical study as outlined in this protocol, according to current Good Clinical Practice and local laws and requirements.

I will ensure that all subinvestigators and other staff members read and understand all aspects of this protocol.

I have received and read all study-related information provided to me.

The objectives and content of this protocol as well as the results deriving from it will be treated confidentially and will not be made available to third parties without prior authorization by UCB.

All rights of publication of the results reside with UCB, unless other agreements were made in a separate contract.

| separate contract. | et |
|---|---|
| Investigator: | dalla |
| | Dustin and any ext |
| | icatil |
| Printed name | Date/Signature |
| Printed name Religh Age in the support any marketing and be used to support any marketing and the support and the support any marketing and the support a | Contion |
| | it knows |
| DED Y | all |
| ike iii. | |
| " Ing" | |
| of all, | |
| <sub>e</sub> upp <sup>o</sup> | |
| 9403 | |
| J580 | |
| O, De | |

The document control be used to support any materials alterial and any state of the control of t


# **Approval Signatures**

| Version: | 1.0 | |
|---|---|---|
| Document Number: | CLIN-000143809 | in the second se |
| Title: | PA0009 Protocol Amendme | nt 3 |
| Approved Date: | 13 Dec 2019 | sionson |
| | | nt 3 Approvals |
| | Document | Approvals |
| Approval<br>Verdict: Approved | ACTED OF | Name: Capacity: Medical Date of Signature: 12-Dec-2019 15:54:05 GMT+0000 |
| Approval<br>Verdict: Approved | SUPPORT SITY MORKETING SUTTO | Name: Capacity: Subject Matter Expert Date of Signature: 12-Dec-2019 16:46:36 GMT+0000 |
| Approval<br>Verdict: Approved | ort any mis | Name: Capacity: Clinical Date of Signature: 13-Dec-2019 08:05:13 GMT+0000 |
| cument cannot be used to | 301 | |